# Janssen Research & Development Statistical Analysis Plan

A Randomized, Active-Controlled, Open-Label, Flexible-Dose Study to Assess the Safety and Tolerability of Topiramate as Monotherapy Compared With Levetiracetam as Monotherapy in Pediatric Subjects with New or Recent-Onset Epilepsy

Protocol TOPMATEPY4067; Phase 3

Amendment 3

**RWJ-17021-000** (topiramate)

Status: Approved

Date: June 8, 2020

**Prepared by:** Janssen Research and Development

**Document No.:** EDMS-ERI-199060224: 4.0

Compliance: The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

#### **Confidentiality Statement**

The information provided herein contains Company trade secrets, commercial or financial information that the Company customarily holds close and treats as confidential. The information is being provided under the assurance that the recipient will maintain the confidentiality of the information under applicable statutes, regulations, rules, protective orders or otherwise.

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

1

# **TABLE OF CONTENTS**

| TABL | E OF CONTENTS | 2 |
|-----------|-----------------------------------------------------------|----|
| LIST | OF IN-TEXT TABLES | 4 |
| AMEN | NDMENTHISTORY | 5 |
| ABBR | EVIATIONS | 6 |
| 1. | CHANGES IN CONDUCT OF THE STUDY | 7 |
| <b>2.</b> | INTRODUCTION | 7 |
| 2.1. | Trial Objectives | |
| 2.2. | Trial Design | |
| 2.3. | Statistical Hypotheses for Trial Objectives | |
| 2.4. | Sample Size Justification | |
| 2.5. | Randomization and Blinding | |
| 2.6. | Time and Events Schedule | |
| | GENERAL ANALYSIS DEFINITIONS | 15 |
| 3.1. | VisitWindows | |
| 3.2. | Pooling Algorithm for Analysis Centers | 18 |
| 3.3. | Analysis Sets | 18 |
| 3.3.1. | Efficacy Analysis Set(s) | 18 |
| 3.3.1. | 1. Primary Efficacy Analysis Set | 18 |
| 3.3.1.2 | 2. Secondary Efficacy Analysis Set | 18 |
| 3.3.2. | All Randomized Set | 18 |
| 3.3.3. | | |
| 3.3.4. | , | |
| 3.3.5. | Pharmacodynamics Analysis Set | 18 |
| 3.4. | Definition of Subgroups | 19 |
| <b>4.</b> | INTERIM ANALYSIS AND DATA MONITORING COMMITTEE REVIEW | 19 |
| 5. | SUBJECT INFORMATION | 20 |
| 5.1. | Demographics and Baseline Characteristics | |
| 5.2. | Disposition Information | |
| 5.3. | TreatmentCompliance | |
| 5.4. | Extent of Exposure | 21 |
| 5.5. | Protocol Deviations | 21 |
| 5.6. | Prior and Concomitant Medications | 22 |
| 5.7. | Medical History | 22 |
| <b>6.</b> | EFFICACY | |
| 6.1. | Analysis Specifications | 22 |
| 6.1.1. | | 22 |
| 6.1.2. | Data Handling Rules | 22 |
| 6.2. | PrimaryEfficacyEndpoint(s) | 22 |
| | SAFETY | |
| 7.1. | Kidney Stones | |
| 7.2. | Weight | |
| 7.3. | Height | |
| 7.4. | Bone Mineral Density (BMD) and Bone Mineral Content (BMC) | |
| 7.5. | Biochemical Markers of Bone Mineralization | |
| 7.6. | Bone Age | |
| 7.7. | Seizure Count | |
| 7.8. | Cognitive, Developmental, and Behavioral Assessments | 25 |

| 7.9.<br>7.10.<br>7.11.<br>7.12.<br>7.13. | Adverse Events Clinical Laboratory Tests Vital Signs and Physical Examination Findings Electrocardiogram Other Safety Parameters | 28<br>28<br>29 |
|---|---|---|
| | PHARMACOKINETICS/PHARMACODYNAMICS | |
| 8.1. | Pharmacokinetics | |
| 8.2. | Immune Response | |
| 8.3. | Pharmacodynamics | |
| 8.4. | Pharmacokinetic/Pharmacodynamic Relationships | 30 |
| 9. I | HEALTH ECONOMICS | 30 |
| 10. | APPENDICES | 30 |
| Ap | ppendix 1: Cogstate Pediatric Normative Data | 31 |
| Αŗ | ppendix 2: Markedly Abnormal Laboratory Parameter Values | 34 |
| 11. l | URINALYSIS | 43 |
| Ap | ppendix 3: AE of clinical interest | 44 |
| Αŗ | pendix 4: Vineland scores | 73 |
| 12. | VARIABLE DESCRIPTION | 75 |
| | opendix 5: CBCL scoring instruction | |
| | opendix 6: Method for computing height velocity values and z-scores for individual subjects | |
| | ppendix 7: List of generic and brand names of AED medications | |

# **LIST OF IN-TEXT TABLES**

| Table 1: | Time and Events Schedule | 11 |
|---|---|---|
| Table 2: | Definition of windows for height, weight, exposure, vital signs, laboratory tests, physical examination and neurological examinations: | 15 |
| Table 3: | Definition of windows for Renal Ultrasound, Cogstate, Tanner Staging and 24 hour urine | |
| | collection: | 15 |
| Table 4: | Definition of windows for C-SSRS: | 16 |
| Table 5: | Definition of windows for Vineland Scale and CBCL: | 16 |
| Table 6: | Definition of windows for Bone age: | 16 |
| Table 7: | Definition of windows for seizure count: | 16 |
| Table 8: | Definition of windows for DEXA: | 17 |
| Table 9: | Definition of windows for Pharmacokinetics | 17 |
| Table 10: | Clinically Important Vital Sign Values | 29 |

#### **AMENDMENT HISTORY**

SAP version issue date

\_\_\_\_\_

Original December 03, 2019

1<sup>st</sup> Amendment February 24, 2020

2<sup>nd</sup> Amendment May 13, 2020

3<sup>rd</sup> Amendment June 4, 2020

#### The overall reason for the amendment 1:

<u>Major:</u> 1. re-insertion of MMRM analysis in a pre-specified way of analysis & 2. additional sensitivity analysis for subjects who took concomitant AED after the first study medication intake.

#### MMRM analysis:

An MMRM analysis is included as sensitivity analysis to explore longitudinal safety data and will be analyzed in the following order.

- 1. The model includes treatment group, study center, age group (4 age groups), visit, treatment-by- visit interaction, baseline measure, and baseline-by-visit interaction with the unstructured covariance matrix.
- 2. If this model experiences convergence issues, then the same model with compound symmetric matrix followed by AR1 will be explored instead of unstructured.
- 3. If the above doesn't work, then a reduced model with treatment group, age group, visit, treatment-by-visit interaction, and baseline measure will be explored. Age will be collapsed to two categories: 2-9 years of age (pre-pubertal) and 10-15 years of age (pubertal). The unstructured covariance matrix will be explored first and if it doesn't work, then compound symmetric followed by AR1 will be applied.
- 4. If above doesn't work, then no additional MMRM analysis will be performed.

#### Sensitivity analyses:

Sensitivity analyses for height z-scores, weight-z-scores and BMD z-scores will be conducted for subset of safety analysis set: for subjects who started taking at least one concomitant AED, data collected after the start of taking AED medication will be excluded from the analysis.

<u>Minor</u>: 1. Insertion of correct schedule of events, 2. Addition of AED medication list in the Appendix, 3. Widening of screening window. 4. Age calculation at each visit for markedly abnormal labs and vital signs. 5. Update to SAS code for Vineland score calculation.

#### The overall reason for the amendment 2:

- 1. Widen the interval for DEXA scan to include 4 subject whose scans were done after baseline but within 1 month post-baseline
- 2. Calculate the exact age at each dosing visit
- 3. Total daily dose calculation for overlapping intervals: capped at their maximum allowed dose

# The overall reason for the amendment 3:

1. Baseline is defined as the last non-missing observation (including an unscheduled visit) prior to or equal to Day 1 (except for DEXA and Bone age, where baseline includes up to 30 days and 180 days post-baseline, respectively).

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

Status: Approved, Date: 08 June 2020

5

# **ABBREVIATIONS**

| AE | Adverse event |
|--------|----------------------------------------------|
| AED | anti-epileptic drug |
| ATC | Anatomical Therapeutic Chemical |
| BMC | bone mineral content |
| BMD | bone mineral density |
| BMDCS | Bone Mineral Density in Childhood Study |
| BMI | Body Mass Index |
| CBCL | Child Behavior Checklist |
| CDC | Centers for Disease Control |
| CI | confidence interval |
| CRF | case report form |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| DEXA | dual energy x-ray absorptiometry |
| DMC | data monitoring committee |
| IWRS | interactive web-based response system |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | Mixed Model Repeated Measures |
| PGTCS | primary generalized tonic-clonic seizures |
| POS | partial-onset seizures |
| PT | preferred term |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SAS | statistical analysis system |
| SD | standard deviation |
| SOC | system organ class |
| SSG | statistical support group |
| TEAE | treatment-emergent adverse event |
| TLF | table, listing, figure |
| WHO | World Health Organization |

#### 1. CHANGES IN CONDUCT OF THE STUDY

On 12 December 2018, the independent Data Monitoring Committee (DMC) recommended to stop the TOPMATEPY4067 study because of futility of study enrollment. On 12 August 2019, Janssen has received the US FDA decision as follows:

- Stop enrolling new subjects at all sites and discontinue the study at all the sites that do not have either subject under study treatment or subjects who require a repeat bone mineral density (BMD) measurement 6 months after discontinuing study treatment.
- All sites with any subject on treatment in the study should continue following the subject according to the protocol until treatment has been completed, the subject has discontinued prematurely, or a repeat DEXA scan (which is indicated 6 months after treatment discontinuation) has been completed.

The US FDA decision is based on the slow rate of study enrollment of subjects despite continuous efforts to improve recruitment in the study. The decision is not related to any safety issues.

Interim analyses on the key endpoints (change in BMD z-score at Month 12, change in height z- score at Month 12 and change in weight z-score at Month 12) were conducted on 13 December 2018. This SAP has been modified based on the early termination of the study.

#### 2. INTRODUCTION

Protocol TOPMATEPY4067 is a randomized (1:1), active-controlled, open-label, flexible-dose, multicenter, Phase 3 study of approximately 282 eligible subjects to evaluate the effects of topiramate monotherapy compared with levetiracetam, another standard antiepileptic drug (AED), as monotherapy for new-onset or recent-onset epilepsy on pediatric growth and maturation, bone mineralization, and kidney stone formation in children 2 to 15 years of age.

The purpose of the Statistical Analysis Plan is to lay out key elements including definition, statistical methods, and tables, listings, and graphs (TLFs).

# 2.1. Trial Objectives

# **Primary Objective:**

The primary objective is to evaluate the effects of topiramate monotherapy compared with levetiracetam, another standard AED, as monotherapy for new-onset or recent-onset epilepsy on pediatric growth and maturation and bone mineralization, in children 2 to 15 years of age.

#### Secondary Objective:

To evaluate the effects of topiramate monotherapy compared with levetiracetam, another standard AED, as monotherapy for new-onset or recent-onset epilepsy on kidney stone formation in children 2 to 15 years of age.

Overall safety will be assessed.

# 2.2. Trial Design

This is a 1-year, active-controlled, randomized, outpatient, multicenter, open-label, 2-arm flexible-dose monotherapy study of topiramate compared with 1 other AED (levetiracetam) in pediatric subjects with epilepsy. Subjects will be required to have newly or recently diagnosed epilepsy characterized by partial-onset seizures (POS) with or without secondary generalized tonic-clonic seizures or primary generalized tonic-clonic seizures (PGTCS).

The study will include the following 3 phases: a screening phase of up to 28 days, an open-label treatment phase of 1 year's duration, and a posttreatment phase of 30 days' duration. There may be an optional post-study follow-up phase to obtain dual energy x-ray absorptiometry (DEXA) measurements in a subgroup of subjects who experience a clinically important reduction in bone mineral density (BMD) (change in Z-score of -0.5 or greater) after 1 year of treatment with topiramate, to determine whether a decrease in BMD after or during 1 year of treatment with topiramate is reversible. These subjects will have a repeat DEXA scan 6 months after discontinuation of study drug.

To minimize any bias in measurement, after randomization 3 of the safety assessments will be obtained in a blinded fashion, including the DEXA scan, renal ultrasound, and height.

An external, independent Data Monitoring Committee (DMC) will be commissioned for this study and will evaluate safety data periodically throughout the study.

# 2.3. Statistical Hypotheses for Trial Objectives

The study will test the hypothesis that flexible dosages of topiramate monotherapy have the same effect as flexible dosages of levetiracetam monotherapy on pediatric growth and bone mineralization, in children 2 to 15 years of age with new-onset or recent-onset epilepsy, versus the alternative hypothesis that the effect of topiramate is different from that of levetiracetam.

### 2.4. Sample Size Justification

A total of 282 randomized subjects, 141 in each treatment group, will be enrolled in the study. The sample size takes into account a 1-year dropout rate of 29%, which is a conservative estimate based on the dropout rates was observed in a previous monotherapy study in the 6- to 15-year-old age group, Study TOPMAT-EPMN-106, including a dropout rate of 22% in the study overall (both double-blind and open-label phases) and a dropout rate of 35% for the double-blind phase. The sample size was estimated in order to achieve a sufficient precision for the estimates of the treatment effect on the key endpoints. The precision of the confidence interval (CI) estimates for the key safety parameters are shown below:

• Annual change in BMD (L1-L4) Z-score: In the Bone Mineral Density in Childhood Study (BMDCS), mean annual change in BMD (L1-L4) Z-score in 6- to 15-year-old healthy subjects was, as expected, minimal (0.01-0.07). The standard deviation (SD) varied from 0.3 to 0.48 across sex and age groups. Assuming an SD of 0.4, with 100 completed subjects per group, the 95% CI for the treatment difference will have a precision of 0.12.

- Annual change in height Z-score in the 2- to 9-year-old age group: In the monotherapy epilepsy study TOPMAT-EPMN-106, the observed change from baseline in mean height Z-score at 1 year among the 2- to 9-year-old subjects treated with topiramate 400 mg/day was -0.18, with an SD of 0.28. Assuming that 53% of the subjects will be recruited in the 2 to 9-year-old age group, i.e., 53 completed subjects per treatment group, the 95% CI for the treatment difference will have a precision of 0.11.
- Change in weight Z-score in the 2- to 15-year-old age group: In the monotherapy epilepsy study TOPMAT-EPMN-106, a -0.59 decrease from baseline in weight Z-score, with an SD of 0.43, was observed after 1 year of treatment with topiramate 400 mg/day. Assuming an SD of 0.43, a sample size of 100 completed subjects per treatment group will provide a 95% CI with a precision of 0.12.

### 2.5. Randomization and Blinding

### Procedures for Randomization and Stratification

Subjects will be randomly assigned to 1 of 2 treatment groups based on a computer-generated randomization schedule prepared before the study by or under the supervision of the sponsor. The randomization will be balanced using randomly permuted blocks and will be stratified by country and age group (2 to 5 years of age, 6 to 9 years of age, 10 to 12 years of age, and 13 to 15 years of age). The enrollment will be monitored throughout the study to ensure that subjects are enrolled for each integer year in each treatment group.

Based on this information, the interactive web-based response system (IWRS) will assign a unique treatment code, which will dictate the treatment assignment and matching study drug kit for the subject. As subjects are randomly assigned to treatment, the IWRS will assign a study drug kit to be dispensed at that visit. New study drug kits will be assigned each time the IWRS is accessed for dispensing additional study drug.

#### **Blinding**

As this is an open-label study, blinding procedures are not applicable for treatment assignment.

To minimize any bias in measurement, after randomization 3 of the safety assessments will be obtained in a blinded fashion, including the DEXA scan, renal ultrasound, and height.

Renal ultrasound will be read/interpreted centrally (local reading at the screening visit is acceptable to determine eligibility for study enrollment). Both the technicians administering the renal ultrasound scans and the local and central readers will be blinded to the study treatment group.

All DEXA scans will be centrally analyzed (the baseline scans will be read locally to determine eligibility for the study). Both the technicians administering the DEXA scans and the central reader will be blinded to the treatment group.

Height will be measured by a trained individual who is blinded (unaware of the treatment).

Nominal blinding or "non-disclosure" of study treatment (i.e., study assessor is not aware of the subject's study treatment assignment) will also be made for assessments related to bone age and cognitive studies (excluding CBCL and Vineland). Nominal blinding will also be applicable to Tanner Staging, in the event site has available a pediatric endocrinologist/trained physician obtaining assessments. The assessors' non-disclosure status at each visit of these assessments will be captured in the eCRF. A sensitivity analysis of these endpoints (bone age, cogstate batteries and Tanner staging) based on nominal blinding may be considered if deemed necessary.

# 2.6. Time and Events Schedule

The flow chart showing trial phases and timing of treatment and assessments is given in Table 1.

**Table 1:** Time and Events Schedule

| Phase | Screening | | Open-Label Treatment <sup>a</sup> | | | | | End-of-<br>Study/Early<br>Withdrawal | Follow-up<br>Telephone<br>Contact |
|---|---|---|---|---|---|---|---|---|---|
| Week(W)/Month(M) Study Day | ≤-28 | Baseline/<br>W1 | M1<br>30 | M2<br>60 | M3<br>90 | M6<br>180 | M9<br>270 | M12<br>360 | M13<br>390 <sup>d</sup> |
| StudyDayWindow | -7days | ±7days | ±7days | ±7days | ±7days | ±7days | ±7days | ±7days | ±7days |
| Visite | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | NA |
| Screening/Administrative | | | | | | | | | |
| Informed consent and assent | X | | | | | | | | |
| Inclusion/exclusion criteria | X | X | | | | | | | |
| Medical/seizurehistory | X | X | | | | | | | |
| Physicalactivityevaluation <sup>f</sup> | X | | | | | | | | |
| Prestudy AED and other therapy <sup>g</sup> | X | | | | | | | | |
| Randomization | | X | | | | | | | |
| StudyDrug | | | | | | | | | |
| Dispensestudydrug | | X | X | X | X | X | X | | |
| Studydrug accountability | | | X | X | X | X | X | X | |
| Pharmacokinetics | | | | | | | | | |
| Blood sample collection for quantitation of studydrug <sup>h</sup> | | | X | | X | X | | X | |
| Safety | | | | | | | | | |
| Physicalexamination | X | X | X | | X | X | X | X | |
| Neurologicexamination | X | X | X | | X | X | X | X | |
| 12-leadECG | X | | | | | | | | |
| Height/weight <sup>i</sup> | X | X | X | | X | X | X | X | |
| Vital signs (temperature, HR, RR, BP) <sup>j</sup> | X | X | X | | X | X | X | X | |
| Clinicallaboratorytests <sup>k</sup> | X | | X | | X | X | X | X | |
| Pregnancy test <sup>l</sup> | X | X | X | X | X | X | X | X | |
| 24-hour urinecollection <sup>m</sup> | X | | | | | X | | X | |
| Tannerstaging <sup>n</sup> | | X | | | | X | | X | |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

**Table 1:** Time and Events Schedule

| Phase | Screening | | Open-Label Treatment <sup>a</sup> | | | | | End-of-<br>Study/Early<br>Withdrawal | Follow-up<br>Telephone<br>Contact |
|---|---|---|---|---|---|---|---|---|---|
| Week(W)/Month(M) | | Baseline/<br>W1 | M1 | M2 | М3 | M6 | M9 | M12 | M13 |
| Study Day | ≤-28 | 1° | 30 | 60 | 90 | 180 | 270 | 360 | 390 <sup>d</sup> |
| StudyDayWindow | -7days | ±7days | ±7days | ±7days | ±7days | ±7days | ±7days | ±7days | ±7days |
| Visit <sup>e</sup> | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | NA |
| Renalultrasoundo | X | | | | | X | | X | |
| Biochemical bone markersp | X | | | | | X | | X | |
| DEXA scanb,q | | X | | | | X | | X | |
| Bone age x-rayr | | X | | | | | | X | |
| Dispense seizure diary and take- | | X | X | X | X | X | X | | |
| Review seizure diary and take- | | | X | X | X | X | X | X | |
| CogstateBatteryt | X | X | | | | X | | X | |
| Animal Fluency Test NEPSY-IIu | X | X | | | | X | | X | |
| Vineland Adaptive Behavior Scalev | | X | | | X | X | | X | |
| CBCL-Parent Versionw | | X | | | X | X | | X | |
| C-SSRSx | | X | X | X | X | X | X | X | |
| OngoingReview | | | | | | | | | |
| Concomitanttherapy | X | X | X | X | X | X | X | X | X |
| Adverse event monitoring | X | X | X | X | X | X | X | X | X |

Footnotes appear on the following page.

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

<sup>&</sup>lt;sup>a</sup> Includes a titration period of approximately 6 to 8 weeks, followed by a maintenance period.

b There may be an optional post-study follow-up phase to obtain DEXA measurements in a subgroup of subjects who experience a clinically important reduction (change in Z-score of -0.5 or greater) in BMD, based on local DEXA scan results, after 1 year of treatment with topiramate; these subjects will have a repeat DEXA scan 6 months after discontinuation of study drug.

<sup>&</sup>lt;sup>c</sup> The Day 1 visit will serve as the baseline visit. All procedures on Day 1 (except dispensing of study drug) should be completed before randomization.

<sup>&</sup>lt;sup>d</sup> The site will contact the subject via telephone at Month 13, to collect data on adverse events and concomitant medications.

<sup>&</sup>lt;sup>e</sup> Window for all visits will be  $\pm 7$  days.

 $<sup>^{\</sup>rm f}\ A dequacy\, of\, physical\, activity\, will\, be\, assessed\, with\, the\, Habitual\, Activity\, Estimation\, Scale.$ 

<sup>&</sup>lt;sup>g</sup> Investigator will document inadequacyof any epilepsy treatment that the subject is receiving at the time of screening. Information regarding AED use and other medications within 2 years prior to the study will also be collected.

- h If possible, blood samples for determination of plasma topiramate and levetiracetam concentrations should be trough samples (taken immediately before the morning dose) and should coincide with samples drawn for clinical laboratory tests.
- <sup>i</sup> Subjects will be weighed in examination gowns or in lightweight clothing and without shoes.
  - Height will be assessed using a wall-mounted stadiometer.
  - All study site personnel measuring height will be blinded to treatment to avoid/minimize bias.
- Orthostatic vital signs will be obtained for all subjects pending cooperation of subjects. A set of 3 measurements will be obtained at baseline only at intervals of 10 minutes. Thereafter, only 1 orthostatic vital sign measurement will be taken at all subsequent visits. The method for obtaining orthostatic vital signs will be as follows: subject will be supine for 5 minutes prior to measurement, and standing for 2 minutes prior to measurement.
- k Clinical laboratory tests (nonfasting) include serumchemistry, hematology, venous ammonia and urinalysis. Insulin-like growth factor 1, 1,25-dihydroxy-vitamin D, 25-hydroxy-vitamin D, and parathyroid hormone will be measured at screening and at Months 6 and 12/early withdrawal. The laboratory tests for 25-hydroxy-vitamin D, 1,25-dihydroxy-vitamin D, Parathyroid hormone (intact) and IGF-1 at screening will be evaluated centrally, but additional evaluation at a local laboratory is allowed in order to reduce the duration of the screening phase.
- Serum pregnancy test at screening; urine pregnancy test at all other visits.
- m A 24-hour urine collection will be analyzed for pH, calcium, citrate, phosphorus, and creatinine levels. Collection instructions and storage conditions will be specified in the laboratory manual. A 14-day window on either side of the scheduled Month 6 visit will be allowed for 24-hour urine collection. The collection at Month 12 should be completed before the Month–12 visit as this evaluation should be obtained while the subject is still receiving study–drug therapy.
- <sup>n</sup> Tanner staging of subjects of age 8 years and above will be conducted by a qualified pediatric endocrinologist or by a physician trained in the method.
- Renal ultrasound will be obtained under blinded conditions after randomization and will be read/interpreted centrally (local reading at the screening visit is
  acceptable to determine eligibility for randomization). Both the technicians administering the renal ultrasound scans and the local and central readers will be
  blinded to the study treatment group.
- P Biochemical bone markers will include serum calcium, phosphorus, parathyroid hormone [intact], 25-hydroxy-vitamin D, and 1,25-dihydroxy-vitamin D.
- <sup>q</sup> DEXA measurements will include posterior-anterior spine (lumbar) and total body less head areal BMD and BMC. Short-term precision testing will be performed for DEXA measurements according to standard protocols. The same DEXA machine will be used at each site for all subjects and all measurements; only clinical sites using recent-generation Hologic or General Electric Lunar systems will participate in the study; the GE/Lunar systems will only be used for subjects ≥5 years of age. If possible, the same technician should acquire all scans for any particular subject.
- Both the technicians administering the DEXA scans and the central reader will be blinded to the treatment group.
- For each time point, up to 3 scan attempts will be performed all on the same day (with repositioning between each scan), with the goal of obtaining 2 complete, movement-free scans of both the spine and whole bodyat screening.
- $^{\rm r}$  A hand/wrist x-ray (in the nondominant hand/wrist) will be used to determine bone age.
- s Subjects will be given a take-home record, to capture data on study drug administration, concomitant medications, and items of general health, and a seizure diary with instructions to record seizure counts and the date and description of each seizure.
- <sup>t</sup> The computerized Cogstate Battery will be administered by non-expert (non-psychologist) study site personnel trained in the Cogstate administration method, with 2 practice sessions, 1 at screening and 1 at baseline prior to the baseline assessment. For subjects 6 to 15 years of age, the Detection Test, Identification Test, One Card Learning Test, One Back Test, and Groton Maze Learning Test will be administered. For cooperative subjects 4 to 5 years of age, the Detection Test and Identification Test will be administered.
- <sup>u</sup> The Animal Fluency Test NEPSY-II will be administered for subjects 6 to 15 years of age, with 1 practice session at screening.
- <sup>v</sup> The Vineland Adaptive Behavior Checklist will be completed by a parent or guardian for subjects 2 to 5 years of age.
- w The CBCL-Parent version will be used for all subjects. For subjects 2 to 5 years of age, the preschool version will be administered. For subjects 6 to 15 years of age, the school-age version will be administered.
- <sup>x</sup> The C-SSRS will be administered for subjects 6 to 15 years of age and will not be administered for subjects 2 to 5 years of age.

AED=antiepilepticdrug;BMC=bone mineralcontent;BMD=bone mineraldensity;BP=bloodpressure;CBCL=ChildBehaviorChecklist;C-SSRS=Columbia Suicide Severity Rating Scale; DEXA=dual energy x-ray absorptiometry; ECG=electrocardiogram; HR=heartrate; IGF-1=insulin-like growth factor 1; NEPSY =A DevelopmentalNEuroPSYchologicalAssessment; RR=respiratory rate.

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

#### 3. GENERAL ANALYSIS DEFINITIONS

Unless otherwise specified, all continuous endpoints (e.g., height, weight, BMD [observed and change from baseline values], etc.) will be summarized using descriptive statistics, which will include the number of subjects with a valid measurement (n), mean, SD, median, minimum, and maximum. Pharmacokinetics will be summarized using descriptive statistics including geometric mean and coefficient of variation (CV in percent will be defined as CV(%) = 100\* SD / mean). All categorical endpoints (e.g., sex, adverse events, BMD Z-score decrease [>0.5, >1.0, >2.0], etc.) will be summarized using frequencies and percentages. In general, percentages will be calculated by dividing the number of subjects with the characteristic of interest by the number of subjects in the analysis population.

#### 3.1. Visit Windows

The statistical analysis for safety will be based on time intervals that are constructed according to the number of days in trial from day 1. (See table 2-8)

The analysis windows for height, weight, exposure, vital signs, laboratory tests, physical examination and neurological examinations is given in Table 2.

Table 2: Definition of windows for height, weight, exposure, vital signs, laboratory tests, physical examination and neurological examinations:

| Scheduled Visit<br>Number | TimeInterval (label on output) | TimeInterval (Day) <sup>a</sup> | Target Time Point |
|---|---|---|---|
| 1,2 | Baseline | -35 to1 | 1 |
| 3 | Month 1 | 2 to 60 | 30 |
| 5 | Month 3 | 61 to 135 | 90 |
| 6 | Month 6 | 136 to 225 | 180 |
| 7 | Month 9 | 226 to 315 | 270 |
| 8 | Month 12 | >=316 | 360 |

<sup>&</sup>lt;sup>a</sup> The randomization day is Day 1.

The analysis windows for Renal Ultrasound, Cogstate, Tanner Staging and 24 hour urine collection is given in Table 3.

Table 3: Definition of windows for Renal Ultrasound, Cogstate, Tanner Staging and 24 hour urine collection:

| Scheduled Visit<br>Number | TimeInterval (label on output) | TimeInterval<br>(Day) <sup>a</sup> | Target Time Point |
|---|---|---|---|
| 1, 2 | Baseline | -35 to1 | 1 |
| 6 | Month 6 | 2 to 270 | 180 |
| 8 | Month 12 | >=271 | 360 |

<sup>&</sup>lt;sup>a</sup> The randomization day is Day 1.

The analysis windows for C-SSRS is given in Table 4.

**Table 4:** Definition of windows for C-SSRS:

| Scheduled Visit<br>Number | TimeInterval<br>(label on output) | TimeInterval (Day) <sup>a</sup> | Target Time Point |
|---|---|---|---|
| 1, 2 | Baseline | -35 to1 | 1 |
| 3 | Month 1 | 2 to 45 | 30 |
| 4 | Month 2 | 46 to 75 | 60 |
| 5 | Month 3 | 76 to 135 | 90 |
| 6 | Month 6 | 136 to 225 | 180 |
| 7 | Month 9 | 226 to 315 | 270 |
| 8 | Month 12 | >=316 | 360 |

<sup>&</sup>lt;sup>a</sup> The randomization day is Day 1.

The analysis windows for Vineland Scale and CBCL is given in Table 5.

 Table 5:
 <u>Definition of windows for Vineland Scale and CBCL:</u>

| 1, 2 Baseline -35 to1 1 5 Month 3 2 to 135 90 | Scheduled Visit<br>Number | TimeInterval (label on output) | TimeInterval<br>(Day) <sup>a</sup> | Target Time Point |
|---|---|---|---|---|
| | 1, 2<br>5 | Month 3 | 2 to 135 | |
| 6 Month 6 136 to 270 180<br>8 Month 12 >=271 360 | 6<br>8 | | | |

<sup>&</sup>lt;sup>a</sup> The randomization day is Day 1.

The analysis windows for Bone Age is given in Table 6.

**Table 6:** Definition of windows for Bone age:

| Scheduled Visit Number | TimeInterval (label on output) | TimeInterval (Day) <sup>a</sup> | Target Time Point |
|---|---|---|---|
| 1 8 | Baseline | -35 to 180 | 1 |
| | Month 12 | >=181 | 360 |

The randomization day is Day 1.

The analysis windows for seizure count is given in Table 7.

**Table 7:** Definition of windows for seizure count:

| Scheduled Visit<br>Number | TimeInterval<br>(label on output) | TimeInterval (Day) <sup>a</sup> | Target Time Point |
|---|---|---|---|
| 3 | Month 1 | 2 to 45 | 30 |
| 4 | Month 2 | 46 to 75 | 60 |
| 5 | Month 3 | 76 to 135 | 90 |
| 6 | Month 6 | 136 to 225 | 180 |
| 7 | Month 9 | 226 to 315 | 270 |
| 8 | Month 12 | >=316 | 360 |

The randomization day is Day 1.

The analysis windows for DEXA is given in Table 8.

**Table 8: Definition of windows for DEXA:** 

| Scheduled Visit<br>Number | TimeInterval (label on output) | TimeInterval (Day) <sup>a</sup> | Target Time Point |
|---|---|---|---|
| 1, 2 | Baseline | -35 to 30 | 1 |
| 6 | Month 6 | 31 to 270 | 180 |
| 8 | Month 12 | >=271 | 360 |

<sup>&</sup>lt;sup>a</sup> The randomization day is Day 1.

The analysis windows for Pharmacokinetics is given in Table 9.

**Table 9: Definition of windows for Pharmacokinetics** 

| Scheduled Visit Number | Time Interval (label on | Time Interval | Target Time Point |
|---|---|---|---|
| | output) | (Day) <sup>a</sup> | |
| 3 | Month 1 | 2 to 45 | 30 |
| 5 | Month 3 | 46 to 135 | 90 |
| 6 | Month 6 | 136 to 270 | 180 |
| 8 | Month 12 | >=271 | 360 |

<sup>&</sup>lt;sup>a:</sup> The randomization day is Day 1

Baseline is defined as the last non-missing observation (including an unscheduled visit) prior to or equal to Day 1 (except for DEXA and Bone age, where baseline includes up to 30 days and 180 days post-baseline, respectively).

For post baseline observations, if more than one visit (including an unscheduled visit) occurs in the same time window, the visit nearest to the target day will be used in the analysis. In the case of an equal distance in time, the latest visit will be used.

Data that are not used in the analysis due to multiple observations or being excluded from the above defined time intervals will be displayed in the data listing.

## 3.2. Pooling Algorithm for Analysis Centers

NA

# 3.3. Analysis Sets

All analyses, except for subject disposition, will use data for the safety analysis set. Demographics will also be summarized based on all randomized set and subject disposition will be based on all subjects.

# 3.3.1. Efficacy Analysis Set(s)

There will be no efficacy analysis set.

# 3.3.1.1. Primary Efficacy Analysis Set

NA

### 3.3.1.2. Secondary Efficacy Analysis Set

NA

#### 3.3.2. All Randomized Set

This will include all randomized subjects.

#### 3.3.3. Safety Analysis Set

This will include all randomized subjects who received at least 1 dose of study medication. This population will be used for all analyses, including any DMC analyses. All subjects will be analyzed according to treatment they received by first study drug dispensation.

#### 3.3.4. Pharmacokinetics Analysis Set

The PK analysis set will consist of all subjects in the safety analysis set with available plasma concentrations.

#### 3.3.5. Pharmacodynamics Analysis Set

NA

# 3.4. Definition of Subgroups

Data will be summarized in addition by age group of 2 to 5 years of age, 6 to 9 years of age, 10 to 12 years of age, and 13 to 15 years of age, separately. For height, Z-scores for height, height velocity and height velocity Z-scores, data will also be summarized by 2 to 9 years of age.

#### 4. INTERIM ANALYSIS AND DATA MONITORING COMMITTEE REVIEW

There will be no interim analyses, but an external, independent DMC will be established to review safety data on a quarterly basis or less frequent basis (but not more than six months) when deemed necessary and ensure the continuing safety of the subjects enrolled in this study. Additional adhoc meetings can be requested by the DMC or the Sponsor. After the review, the DMC will make recommendations regarding the continuation of the study. The details will be provided in a separate DMC charter.

The DMC is comprised of four clinicians and one statistician. The Chairperson and one member are pediatric endocrinologists with expertise in bone, growth and maturation; the other two clinicians are a pediatric nephrologist and a pediatric neurologist. Mention one member is statistician. The DMC responsibilities, authorities, and procedures will be documented in its charter.

The safety analyses will be performed by Statistical Support Group (SSG) independent of the Sponsor. The output tables in the data package will be displayed by each age group (2-5, 6-9, 10-12, and 13-15) and overall. All data and output should be held in strict confidentiality with access to DMC and SSG only before they can be transferred to the Sponsor.

Separate outputs will be generated for the open- and closed-sessions of the DMC meetings. The outputs in the data package for the open-session will be unblinded, except for Ultra Sound, DEXA and height analyses. These will present summaries for all subjects combined (e.g., tables will only present a Total column). All outputs in the data package for the closed-session will be unblinded and will present the data by the subjects' true treatment group assignment.

Before each scheduled DMC meeting, data cut-off dates (6 to 8 weeks prior to the meeting) will be identified and the clinical database will be made as clean as possible, with particular focus on safety data. For the purpose of the DMC review of the results, all available data needed for the TLFs up to the time of data cut-off dates, unless otherwise specified will be included in the TLFs.

The Contract Research Organization, PAREXEL, will provide the SDTM datasets containing the electronic case report form (eCRF) data, the cognitive battery data (computerized cognitive battery as well as NEPSY testing), and the central laboratory data to the SSG statistician using the Janssen MBOX. The DEXA and US data will be provided directly to the SSG statistician by Bioclinica. Given that this is an open-label study, the treatment assignment will be included in the CRF data.

### 5. SUBJECT INFORMATION

# 5.1. Demographics and Baseline Characteristics

Subject demographics and baseline disease characteristics will be listed and summarized for the randomized analysis set by treatment group. Descriptive statistics (mean, standard deviation, median, minimum, and maximum) will be presented for age, height, weight, body mass index (BMI), and years since diagnosis of epilepsy. Frequency counts and percentages will be presented for categorical variables sex, age group (2-5 years, 6-9 years, 10-12 years, 13-15 years), ethnicity, race, geographic region, , seizure types present within the last 2 years, seizure occurred within the last 2 years beyond 3 or 5 month , seizure occurred in last 3 or 5 months and any AED drug/therapy at study entry and bicarbonate categories. Bicarbonate values are categorized as low (<20 mEq/L at screening) and non-low bicarbonate values (>=20 mEq/L at screening).

Age in years will be used from eCRF. In case of missing eCRF for age, 15th of the month will be used as day. Missing day and moth at date of birth will be imputed by June 30. Years since diagnosis of epilepsy will be calculated based on year of Day 1 minus year of diagnosis (if both in the same year it will be 0).

#### • Age calculation:

- For Height and Weight Z-Scores, it is given in CDC guidance document, age is in month with one decimal.
- For demographics, it is floor (ICF date minus birth date)/365.25), age is in full years.
- For Vineland it is floor ((intck ('month', birth date, visit date)-(day (visit date)<day(birth date)))), age is in full month.
- For CBCL it is floor (visit date minus birth date)/365.25), age is in full years.
- For Cogstate it is floor (visit date minus birth date)/365.25), age is in full years.
- For vital signs it is floor (visit date minus birth date)/365.25), age is in full years.
- For labs it is floor (visit date minus birth date)/365.25), age is in full years.
- Age for determination of max daily dose for Topiramate or Levetiracetam it is floor (date of dosing minus birth date)/365.25), age is in full years.
- BMI is calculated as weight (kg) / height  $(m)^2$ .

Geographic region will be summarized as North America, South America, Europe and Asia Pacific.

- North America: US, Canada
- South America: Argentina, Mexico
- Europe: Belgium, France, Germany, Hungary, Italy, Poland, Russian Federation, Austria, South Africa, UK
- Asia Pacific: Australia, Taiwan, Philippines

# 5.2. Disposition Information

Distribution of subjects will be provided for the all randomized analysis set. The number of subjects screened, screen failures, randomized, dosed, completed, and discontinued will be listed and summarized. Treatment discontinuation will be summarized according to reasons of discontinuation as documented in the CRF. The screen failures and the reasons will be listed.

### 5.3. Treatment Compliance

Treatment compliance will not be summarized.

### 5.4. Extent of Exposure

Treatment duration is defined as time between the first dose date and last dose date of topiramate or levetiracetam and will be presented as a continuous summary and classified into the following categories by the amount of time on study medication: 0 to <3 months, 3 to <6 months, 6 to <9 months, 9 to <12 months, and  $\ge 12$  months. The number and percentage of subjects in each category will be reported.

A summary of the average total daily dose and the weight-adjusted average daily dose (mg/kg) will also be presented. The weight will be used at start of the respective period (titration and maintenance). For exposure with overlapping records, if a 'total daily dose' exceeds the maximum dose allowed for the subject, a total daily dose of 350 mg or 400 mg for Topiramate will be used for the subject with age <10 years or >=10 years, respectively. For Levetiracetam, the total daily dose of 3,000 mg will be used if the exposure with overlapping records exceeds the maximum allowed dose of 3,000 mg. It will also be summarized by the treatment period (titration and maintenance). The start of maintenance period is defined as "date maintenance achieved" from titration CRF, and the end of titration period is defined as "start of maintenance period minus 1".

A listing of dispensed medication will also be provided.

#### 5.5. Protocol Deviations

The major protocol deviations will be listed and summarized by treatment group. A subject can be counted under multiple deviation categories.

The major Protocol Deviation categories

- Developed withdrawal criteria but not withdrawn
- Entered but did not satisfy criteria
- Received a disallowed concomitant treatment
- Received wrong treatment or dose deviation
- Selection criteria not met
- Informed consent not correctly signed
- Visit schedule is not followed according to protocol
- Safety assessments not performed according to protocol

• Safety assessments not documented properly

The minor protocol deviations will not be summarized.

#### 5.6. Prior and Concomitant Medications

Medications administered prior to the first dose of study medication will be considered prior medications. Concomitant medications include those taken on or after first dose date. Incidence of prior and concomitant medications will be summarized by Anatomical Therapeutic Chemical (ATC) code levels 2 and 4, and preferred term. Only prior anti-epileptic drugs (AEDs) will be summarized. Concomitant medications will be listed and summarized separately for AED and non-AED medications. Tables will be sorted by decreasing frequency in incidence (the highest to lowest incidence) first within ATC code level 2, followed by ATC code level 4, and then preferred term. Medications with partial onset date will be handled as follows: a missing day should be set to first of month. If month is missing the missing month should be set to January.

Please see Appendix 7 for the list of AED medications.

## 5.7. Medical History

Medical history will be listed only.

#### 6. EFFICACY

There are no efficacy data collected for the study.

# 6.1. Analysis Specifications

# 6.1.1. Level of Significance

NA

### 6.1.2. Data Handling Rules

NA

# 6.2. Primary Efficacy Endpoint(s)

NA

#### 7. SAFETY

The safety variables to be summarized include kidney stones, height, weight, BMD and bone mineral content (BMC), biochemical markers of bone mineralization, bone age XR, seizure counts, cognitive, developmental, and behavioral assessments, treatment-emergent AEs, Columbia-Suicide Severity Rating Scale (C-SSRS), cognitive, developmental and behavioral assessments (COGSTATE computerized battery and NEPSY Language scale; Vineland Adaptive Behavioral Scale, Child Behavior Checklist (CBCL)), clinical laboratory tests (hematology, chemistry, urinalysis, and 24-hour urine collection), vital signs and physical exam. Safety variables are to be tabulated by descriptive statistics (n, mean, median, SD, minimum, and maximum; or n and percent). No formal statistical testing is planned.

For markedly abnormal labs and vital signs, age will be calculated at each visit to determine the criteria. Similarly, Vineland, CBCL and Cogstate will be calculated by age at each visit.

Z-scores for weight and height will be calculated using the SAS programs provided by the Centers for Disease Control (CDC) for the calculation of the 2000 CDC growth charts. Z-scores for the BMD and BMC will be provided by the central DEXA reading center (Bioclinica).

Z-scores for the DEXA scans will be calculated locally at baseline only to determine eligibility for the study, and centrally for all statistical analyses. The Z-score calculation will take the DEXA machine and the subject's age, sex, height, and ethnicity into consideration. The reference databases for calculating the Z-scores are provided in the DEXA Manual for this study (please see the imaging charter of attachment 1 for more details).

Longitudinal endpoints will be analyzed using a mixed-model repeated measures (MMRM) analysis. An MMRM analysis is included as sensitivity analysis to explore longitudinal safety data and will be analyzed in the following order.

- 1. The model includes treatment group, study center, age group (4 age groups), visit, treatment-by-visit interaction, baseline measure, and baseline-by-visit interaction with the unstructured covariance matrix.
- 2. If this model experiences convergence issues, then the same model with compound symmetric matrix followed by AR1 will be explored instead of unstructured.
- 3. If the above doesn't work, then a reduced model with treatment group, age group, visit, treatment-by-visit interaction, and baseline measure will be explored. Age will be collapsed to two categories: 2-9 years of age (pre-pubertal) and 10-15 years of age (pubertal). The unstructured covariance matrix will be explored first and if it doesn't work, then compound symmetric followed dby AR1 will be applied.
- 4. If above doesn't work, then no additional MMRM analysis will be performed. 95% CI for the estimated treatment differences will be provided.

#### Example of MMRM is as follows:

```
ods output estimates=est;
PROC MIXED data=dat method=REML noclprint=10;
CLASS trt center usubjid age_group visit;
MODEL change=trt base visit center age_group trt*visit base*visit / solution; repeated visit / type=un subject=usubjid;
lsmeans trt/diff cl;
```

Sensitivity analyses for height z-scores, weight-z-scores and BMD z-scores will be conducted for subset of safety analysis set: for subjects who started taking at least one concomitant AED, data collected after the start of taking AED medication will be excluded from the analysis.

# 7.1. Kidney Stones

Percentage of subjects with kidney stones and other US findings suggestive of stones will be summarized by treatment group.

The renal ultrasound findings will also be presented in a listing.

# 7.2. Weight

Observed weight values, change from baseline, Z-scores for weight, and change from baseline in Z-scores for weight will be listed and summarized by visit using descriptive statistics. The change in weight z-scores will also be summarized by subject's serum bicarbonate categories.

MMRM analysis will also be performed for changes from baseline and changes in Z-Scores from baseline.

# 7.3. Height

Observed height values, change from baseline, Z-scores for height, change from baseline in Z-scores for height, height velocity at 1 year, and height velocity Z-score will be summarized by visit using descriptive statistics. Height, Z-scores for height, height velocity and height velocity Z-scores will be calculated as the mean of the three measurements. The number and percentage of subjects with a height Z-score decrease of >0.5, >1.0, and >2.0 will be listed and summarized by visit using descriptive statistics. MMRM analysis will also be performed for changes from baseline and changes in Z-Scores from baseline.

The change in height z-scores will also be summarized by subject's serum bicarbonate categories.

Height velocity values and associated Z-scores will be computed for each post-baseline year in the study, based on the methods described in Appendix 6.

# 7.4. Bone Mineral Density (BMD) and Bone Mineral Content (BMC)

DEXA measurements will include posterior-anterior spine and total body less head areal (TBLH) BMD and BMC. Observed BMD (spine and TBLH) and BMC (spine and TBLH) values change from baseline, Z-scores as well as height adjusted Z-scores for BMD and BMC, change from baseline in Z-scores and height adjusted Z-scores for BMD and BMC, and percent change from baseline in BMD and BMC will be summarized by visit using descriptive statistics. The number and percentage of subjects with a BMD Z-score and adjusted Z-score decrease of >0.5, >1.0, and >2.0 will be listed and summarized by visit using descriptive statistics. MMRM analysis will also be performed for changes from baseline, changes in Z-Scores from baseline, and changes in height adjusted Z-Scores from baseline.

Subjects with a clinically important reduction in BMD defined as change in Z-score and height adjusted Z-score of -0.5 or greater) at 6 months or 12 months, will have a repeat DEXA scan 6 months after discontinuation of study drug. These subjects will be summarized and listed in the DEXA table and listing.

The change in BMD z-scores will also be summarized by subject's serum bicarbonate categories.

#### 7.5. Biochemical Markers of Bone Mineralization

Observed and change from baseline in biochemical markers of bone mineralization (serum levels of alkaline phosphatase, calcium, phosphorus, parathyroid hormone (intact), 25-hydroxy vitamin D, 1,25-dihyroxy vitamin D, and IGF-1) will be listed and summarized by visit using descriptive statistics.

# 7.6. Bone Age

Observed and change from baseline in bone age will be listed and summarized by visit using descriptive statistics. Bone age will be summarized as "chronological age" and "bone age" as reported as XR report.

#### 7.7. Seizure Count

Observed seizure counts will be listed and summarized by visit using descriptive statistics, for both the overall seizure count and by seizure type (Partial, Partial Evolving into Secondary Generalized, Primary Generalized Tonic-Clonic, and Other).

# 7.8. Cognitive, Developmental, and Behavioral Assessments

#### **Cognitive Assessments**

For the cognitive assessments (Detection Test, Identification Test, One Card Learning Test, One Back Test, and Groton Maze Learning Test) the standardized observed scores and change from baseline in standardized scores will be listed and summarized by visit using descriptive statistics. The standardized scores will be calculated by setting the observed raw score in relation to the expected within-subject standard deviations for each Cogstate task (see table 1-5 of Appendix 1 for normative data). For the tasks which lower scores indicate improvement (e.g., Detection Test and Identification Test), the score will be multiplied by (-1), so that a negative change in standardized scores represent a decline in cognitive performance consistently across all tasks.

A meaningful decline in cognition has been defined as a change in standardized score of less than -1.65 from the baseline standardized score. These calculations will indicate meaningful decline at the subject level. Each individual change in standardized scores that meet the definition of a meaningful decline will be identified using a binary flag, where 1 represents a meaningful decline from baseline and 0 otherwise. The number and percentage of subjects with a meaningful decline in cognition will be listed and summarized by visit.

Cognitive assessments will be provided to subjects of 4 years and older. Cognitive data collected after a subject turn 16 will not be included in the analysis.

For example, if a 10-year-old female subject has an observed raw score at baseline of 1.2 for the detection test, then the standardized score will be 1.2/0.0882\*(-1)=-13.605. For a post baseline visit the subject had an observed raw score of 1.0, which is a standardized score of -11.338. The

change from baseline would be 2.267. The lower score at post baseline indicates an improvement in Detection Test which is reflected by the positive change (see table 1 of Appendix 1).

# **Developmental Assessments**

The Vineland Scales of Adaptive Behavior provide age-specific assessment of function in the domains of communication, daily living, socialization, and motor skills, as well as a composite scale. The subject's sub-domain raw scores are entered on the CRF. The derived domain scores (standardized scores) based on the national standardization sample must be obtained from these raw scores. The derived scores are used in the analyses. The Vineland standardized scores for domain scores have a mean of 100 and a standard deviation of 15.

The composite score will be the sum of 4 standardized domain scores. If a subject has only 3 domains, then the standardized score for the missing domain will be prorated and the composite score will be calculated as sum of 4 domains. If a subject has less than 3 domains, then the composite score will not be calculated.

The standardized scores and the changes in standardized scores from baseline will by listed and summarized by visit using descriptive statistics.

For manuals and SAS program calculating the standardized domain scores, please see Appendix 4.

The Vineland Adaptive Behavior Scale will be administered for subjects 2 to 5 years of age only.

#### **Behavioral Assessments**

For CBCL preschool (up to 5 years of age), a raw total score will be sum of 99 non-missing answers (range of 0-198).

For CBCL school age (6 to 18 years of age), a raw total score will be the sum of 112 non-missing answers (range of 0-224).

The domains will be:

| СВ | CL preschool | CBCL school age |
|---|---|---|
| 1. | Emotionally Reactive | 11. Anxious/depressed |
| 2. | Anxious/Depressed | 12. Withdrawn/depressed |
| 3. | Somatic Complaints | 13. Somatic complaints |
| 4. | Withdrawn | 14. Social problems |
| 5. | Sleep Problems | 15. Thought problems |
| 6. | Attention Problems | 16. Attention problems |
| 7. | Aggressive Behavior | 17. Rule breaking behavior |
| 8. | Internalizing Problems | 18. Aggressive behavior |
| 9. | Externalizing Problems | 19. Internalizing Problems |
| 10. | Total Problems | <ul><li>20. Externalizing Problems</li><li>21. Total Problems</li></ul> |

The standardized total scores (T score) for all domains will be derived using the charts based on the raw scores (Appendix 5).

The standardized scores and the changes in standardized scores from baseline will by listed and summarized by visit using descriptive statistics.

#### 7.9. Adverse Events

Adverse events are coded to System Organ Class (SOC) and preferred terms (PT) using the Medical Dictionary for Regulatory Activities (MedDRA) coding system, version 21.1 or higher. Treatment-emergent adverse events (TEAEs) are those AEs which start or worsen after receipt of the first study drug and before the end of the REACH. REACH is defined as follows: AEs with onset date within therapeutic reach (i.e. 3 days) or SAEs/deaths with onset date within 30 days, inclusive, after end of treatment. AE's with partial onset date will be handled as follows: a missing day should be set to first of month. If month is missing the missing month should be set to January.

Summaries of TEAEs will be provided as incidence tables (number of subjects experiencing an event) by treatment group within each age group and overall (age 2-15). For each TEAE, the percentage of subjects who experience at least 1 occurrence of the given event will be summarized. Tables will be sorted by decreasing frequency in incidence (the highest to lowest incidence) first within the SOC and then the PT. Treatment-emergent serious AEs (SAEs), TEAEs leading to discontinuation, TEAEs by severity, TEAEs by relationship and TEAEs of special interest will be summarized. Adverse events of special interest for topiramate include: effects on liver function; metabolic acidosis; effects on growth and maturation; vision abnormalities; oligohidrosis, hyperthermia and secondary rash; hyperammonemia and/or encephalopathy; kidney stones; neuropsychiatric and cognitive disorders; and suicidality. Adverse events of clinical interest for levetiracetam are as listed previously, notably somnolence, asthenia, and behavior disturbances

(especially hostility and nervousness). Please see Appendix 3 for the MedDRA codes for these AE of clinical interest.

A listing of AEs will also be provided.

### 7.10. Clinical Laboratory Tests

Figures of the mean change from screening (+/- Standard Error) values in continuous hematology, urinalysis and serum chemistry laboratory parameters will be presented by visit. The observed and change from baseline values of lab parameters will also be summarized by visit. For calculation, the signs "<" or ">" will be removed and resulting numerical value will be used. The reference ranges for labs from the SAP will be used, not the reference ranges provided from the Covance.

The shift table of pre- vs. post-treatment with classes for below, within, and above normal ranges will be presented.

The number and percentage of subjects with markedly abnormal (low, high) laboratory hematology, urinalysis/24-hour urine and serum chemistry parameters during the study (from treatment start to 30 days after last dose or the end of treatment visit date, whichever is later) that were not present at baseline will be provided. Appendix 2 presents the markedly abnormal criteria. The conversion factors for 25 Vitamin D, 1, 25 Vitamin D and PTH are also listed.

The laboratory data will be listed. The subjects with any laboratory results outside the reference ranges and the subjects with any markedly abnormal laboratory results will be listed.

# 7.11. Vital Signs and Physical Examination Findings

At baseline, 3 orthostatic vital signs will be measured 10 min apart and the baseline score will be calculated as the average of 3 scores.

Observed and change from baseline in vital sign parameters (temperature, pulse/heart rate, respiratory rate, and blood pressure [standing and supine]]) will be summarized by visit using descriptive statistics.

The number and percentage of subjects with any clinically important vital sign values during the study will also be summarized by visit. Table 10 presents the criteria for the clinically important values.

Table 10: Clinically Important Vital Sign Values

| Parameter | Age group (Years) | Low | High |
|---|---|---|---|
| Systolic Blood Pressure | 2-5 yrs | <75 | >110 |
| | 6-9 yrs | <80 | >120 |
| | ≥10 yrs | <90 | >130 |
| Diastolic Blood Pressure | 2-5 yrs | <35 | >65 |
| | 6-9 yrs | <45 | >75 |
| | ≥10 yrs | < 50 | >80 |
| Heart Rate | 1-2 yrs | <89 | >151 |
| | 3-4 yrs | <73 | >137 |
| | 5-7 yrs | <65 | >133 |
| | 8-11 yrs | <62 | >130 |
| | ≥12 yrs | <60 | >119 |
| Respiratory Rate | 1-3 yrs | <22 | >30 |
| • | 4-6 yrs | <20 | >24 |
| | 7-9 yrs | <18 | >24 |
| | 10-14 yrs | <16 | >22 |
| | 15-18 yrs | <14 | >20 |
| Temperature | Allages | <35° C (95° F) | ≥37.5° C (99.5° F) |

The vital signs data will be listed. The subjects with any clinically important vital signs data will be listed in addition.

The number and percentage of subjects with abnormal physical examination will be listed and summarized by body system and visit.

# 7.12. Electrocardiogram

ECG at screening will not be listed.

# 7.13. Other Safety Parameters

#### Columbia-Suicide Severity Rating Scale (C-SSRS):

From the C-SSRS, the number and percentage of subjects reporting (1) at least one occurrence of suicidal ideation or behavior, (2) any type of suicidal behavior, and (3) any type of suicidal ideation during the study (from treatment start to 30 days after last dose or the end of treatment visit date, whichever is later) will be summarized.

#### **Tanner Staging:**

Observed and change from baseline in Tanner Staging will be listed and summarized by visit using descriptive statistics. Frequency distribution of tanner staging (1 thru 5) will also be summarized by visit.

#### 8. PHARMACOKINETICS/PHARMACODYNAMICS

#### 8.1. Pharmacokinetics

All concentrations below the lowest quantifiable concentration or missing data will be labeled as such in the concentration data presentation. Concentrations below the lowest quantifiable concentration will be treated as zero in the summary statistics. All subjects and samples excluded from the analysis will be clearly documented in the study report.

For each treatment group, descriptive statistics, including arithmetic mean, SD, coefficient of variation, geometric mean, median, minimum, and maximum will be calculated for the Topiramate or Levetiracetam plasma concentrations at each sampling time.

Topiramate and Levetiracetam plasma concentrations will be provided as listings.

# 8.2. Immune Response

NA

# 8.3. Pharmacodynamics

NA

### 8.4. Pharmacokinetic/Pharmacodynamic Relationships

NA

#### 9. HEALTH ECONOMICS

NA

#### 10. APPENDICES

### Appendix 1: Cogstate Pediatric Normative Data

Table 1: CogState Pediatric Normative Data for the Detection Task.

| | | Males | | | Females | |
|-------------|------|--------|--------|------|---------|--------|
| Age (years) | N | М | SD | N | М | SD |
| 2 | _ | _ | _ | _ | _ | _ |
| 3 | _ | _ | _ | 1 | 2.9041 | _ |
| 4 | 2 | 2.8775 | 0.0534 | 3 | 2.8581 | 0.1732 |
| 5 | 4 | 2.7714 | 0.1001 | 10 | 2.7341 | 0.0871 |
| 6 | 5 | 2.6002 | 0.0717 | 11 | 2.8240 | 0.1660 |
| 7 | 6 | 2.6733 | 0.1357 | 9 | 2.7294 | 0.0622 |
| 8 | 4 | 2.6115 | 0.1769 | 6 | 2.8202 | 0.1598 |
| 9 | 4 | 2.5632 | 0.1146 | 3 | 2.5398 | 0.0714 |
| 10 | 1224 | 2.5631 | 0.0870 | 210 | 2.5882 | 0.0882 |
| 11 | 1499 | 2.5388 | 0.0826 | 506 | 2.5641 | 0.0899 |
| 12 | 1882 | 2.5290 | 0.0842 | 816 | 2.5447 | 0.0831 |
| 13 | 2322 | 2.5177 | 0.0851 | 1076 | 2.5255 | 0.0767 |
| 14 | 6551 | 2.5121 | 0.0853 | 3315 | 2.5252 | 0.0826 |
| 15 | 6399 | 2.5086 | 0.0810 | 3347 | 2.5213 | 0.0821 |

Note: The primary outcome variable for the Detection task is Reaction Time (Log10 transformation).

Table 2: CogState Pediatric Normative Data for the Identification Task.

| _ | | Males | | | Females | |
|-------------|------|--------|--------|----------------|---------|--------|
| Age (years) | N | M | SD | N | M | SD |
| 2 | _ | _ | _ | _ | _ | _ |
| 3 | _ | = | = | $\overline{1}$ | 3.1028 | _ |
| 4 | 2 | 3.0312 | 0.0142 | 3 | 3.1244 | 0.0795 |
| 5 | 4 | 2.9061 | 0.0266 | 10 | 2.9546 | 0.1075 |
| 6 | 5 | 2.9199 | 0.0931 | 11 | 2.9938 | 0.1276 |
| 7 | 6 | 2.9238 | 0.1067 | 9 | 2.9310 | 0.0849 |
| 8 | 4 | 2.8885 | 0.1575 | 6 | 2.9726 | 0.1053 |
| 9 | 4 | 2.7421 | 0.0453 | 3 | 2.7632 | 0.0634 |
| 10 | 1198 | 2.7637 | 0.0759 | 203 | 2.7796 | 0.0735 |
| 11 | 1456 | 2.7323 | 0.0739 | 499 | 2.7453 | 0.0727 |
| 12 | 1823 | 2.7163 | 0.0712 | 811 | 2.7186 | 0.0726 |
| 13 | 2279 | 2.7007 | 0.0725 | 1073 | 2.6973 | 0.0711 |
| 14 | 6470 | 2.6889 | 0.0731 | 3300 | 2.6903 | 0.0719 |
| 15 | 6324 | 2.6809 | 0.0700 | 3335 | 2.6800 | 0.0717 |

Note: The primary outcome variable for the Identification task is Reaction Time (Log10 transformation).

Table 3: CogState Pediatric Normative Data for the One Card Learning Task.

| | Males | | | Females | | |
|-------------|-------|--------|--------|---------|--------|--------|
| Age (years) | N | M | SD | N | M | SD |
| 6 | 5 | 1.0120 | 0.1845 | 11 | 1.0029 | 0.1441 |
| 7 | 6 | 0.9715 | 0.1175 | 9 | 0.9300 | 0.1616 |
| 8 | 4 | 1.1346 | 0.0765 | 6 | 0.9942 | 0.1889 |
| 9 | 4 | 1.0406 | 0.0376 | 3 | 0.9863 | 0.1306 |
| 10 | 1147 | 0.9639 | 0.0880 | 201 | 0.9636 | 0.0910 |
| 11 | 1449 | 0.9646 | 0.0889 | 485 | 0.9650 | 0.0892 |
| 12 | 1837 | 0.9719 | 0.0889 | 807 | 0.9692 | 0.0875 |
| 13 | 2249 | 0.9722 | 0.0858 | 1053 | 0.9767 | 0.0874 |
| 14 | 6435 | 0.9715 | 0.0870 | 3347 | 0.9679 | 0.0858 |
| 15 | 6559 | 0.9739 | 0.0868 | 3434 | 0.9718 | 0.0854 |

Note: The primary outcome variable for the One Card Learning task is Accuracy (arcsine square-root transformation).

Table 4: CogState Pediatric Normative Data for the One Back Task.

| _ | Males | | | Females | | |
|-------------|-------|--------|--------|---------|--------|--------|
| Age (years) | N | М | SD | N | M | SD |
| 6 | 5 | 3.0924 | 0.0965 | 11 | 3.1386 | 0.1728 |
| 7 | 6 | 3.0799 | 0.0686 | 9 | 3.0789 | 0.0926 |
| 8 | 4 | 2.9574 | 0.0691 | 6 | 3.1290 | 0.1488 |
| 9 | 4 | 2.9524 | 0.0589 | 3 | 2.9646 | 0.1824 |
| 10 | 1278 | 2.9597 | 0.0984 | 218 | 2.9840 | 0.0990 |
| 11 | 1576 | 2.9225 | 0.0958 | 548 | 2.9405 | 0.0962 |
| 12 | 1973 | 2.8977 | 0.0962 | 879 | 2.9139 | 0.0972 |
| 13 | 2437 | 2.8824 | 0.0945 | 1130 | 2.8931 | 0.0938 |
| 14 | 7000 | 2.8673 | 0.0935 | 3604 | 2.8851 | 0.0930 |
| 15 | 7061 | 2.8547 | 0.0926 | 3663 | 2.8716 | 0.0952 |

Note: The primary outcome variable for the One Back task is Reaction Time (Log10 transformation).

Table 5: CogState Pediatric Normative Data for the Groton Maze Learning Test.

| _ | Males | | | Females | | |
|-------------|-------|----------|---------|---------|---------|---------|
| Age (years) | N | М | SD | N | М | SD |
| 6 | _ | _ | _ | 2 | 63.5000 | 16.2635 |
| 7 | 1 | 102.0000 | _ | _ | _ | _ |
| 8 | _ | _ | _ | 1 | 68.0000 | _ |
| 9 | 3 | 64.6667 | 24.0069 | 1 | 27.0000 | _ |
| 10 | 20 | 73.8500 | 31.0251 | 6 | 67.3333 | 25.5943 |
| 11 | 14 | 67.6429 | 22.4828 | 12 | 64.1667 | 14.9595 |
| 12 | 20 | 62.9500 | 18.9667 | 6 | 61.0000 | 14.0855 |
| 13 | 10 | 53.2000 | 19.0660 | 11 | 65.0000 | 15.7861 |
| 14 | 5 | 61.6000 | 16.7422 | 2 | 46.0000 | 19.7990 |
| 15 | _ | _ | _ | 1 | 39.0000 | _ |

Note: The primary outcome variable for the Groton Maze Learning Test is Total Errors.

Status: Approved, Date: 08 June 2020

# Appendix 2: Markedly Abnormal Laboratory Parameter Values

# Chemistry

| Laboratory Value<br>(SI Unit) | Lower Limit of<br>Normal(LLN)<br>Range | Upper Limit of<br>Normal(ULN)<br>Range | DNP<br>Recommended<br>Markedly<br>Abnormal:Low | DNP<br>Recommended<br>Markedly<br>Abnormal: High |
|---|---|---|---|---|
| Alanine Amino<br>Transferase – ALT<br>(SGPT)(U/L) | 1 | 30 | NA | ≥3 X ULN, OR<br>≥5 X ULN, OR<br>≥10 X ULN |
| Aspartate Amino<br>Transferase - AST<br>(SGOT)(U/L) | 0 | 35 | NA | ≥3 X ULN, OR<br>≥5 X ULN, OR<br>≥10 X ULN |
| Albumin(g/L) | <5 years:<br>29 | <5 years:<br>58 | <5 years:<br>≤20 | <5 years:<br>≥65 |
| | <u>≥5 years:</u><br>31 | <u>≥5 years:</u><br>54 | <u>≥5 years:</u><br>≤25 | <u>≥5 years:</u><br>≥ 60 |
| Alkaline<br>Phosphatase(U/L) | Females:<br>2-10 years:<br>100<br>11-17 years: | Females: 2-10 years: 320 11-17 years: | NA | > 3 X ULN |
| | 100<br><u>≥18 years:</u><br>30<br><i>Males:</i> | 320<br><u>≥18 years:</u><br>120<br><i>Males:</i> | | |
| | <u>2-10 years</u> :<br>100<br><u>11-17 years</u> :<br>100 | 2-10 years:<br>320<br>11-17 years:<br>390 | | |
| | <u>≥18 years:</u> 30 | <u>≥18 years:</u><br>120 | | |
| Ammonia(umol/L) | ≤18 years:<br>21 | ≤18 years:<br>50 | NA | ≥1.5 X ULN |
| | <u>&gt;18 years:</u><br>0 | >18 years:<br>35.7 | | |
| Bicarbonate/ | | _ | Value < 17, OR | _ |
| Laboratory Value<br>(SI Unit) | Lower Limit of<br>Normal (LLN)<br>Range | Upper Limit of<br>Normal(ULN)<br>Range | DNP<br>Recommended<br>Markedly<br>Abnormal:Low | DNP<br>Recommended<br>Markedly<br>Abnormal: High |
|---|---|---|---|---|
| CarbonDioxide<br>(CO2)(mmol/L) | 20 | 26 | (Value <17 and decrease from pre-treatment baseline >5 when pre-treatment baseline \( \geq 20 \) | ≥ <u>3</u> 1 |
| Bilirubin – Total<br>(umol/L) | 1.7 | 20.5 | NA | <u>&gt;</u> 41 |
| Blood Urea<br>Nitrogen (BUN)<br>(mmol/L) | 2.5 | 7.9 | NA | <u>&gt;</u> 16 |
| Calcium(mmol/L) | 2 | 2.6 | ≤ 1.7 | <u>≥</u> 3 |
| Chloride(mmol/L) | 96 | 109 | NA | <u>&gt;</u> 112 OR <u>≥</u> 115 |
| TotalCholesterol (mmol/L) | <18 years:<br>0 | <u>&lt;18 years:</u><br>5.18 | NA | ≥1.2 X ULN |
| | ≥18 years:<br>0 | <u>≥18 years:</u><br>6.2 | | |
| Creatinine (umol/L) | 2-12 years:<br>27<br>13-17 years:<br>44 | 2-12 years:<br>62<br>13-17 years:<br>88 | NA | ≥1.6 X ULN |
| | | <u>≥18 years:</u><br>Males<br>115<br>Females | | |

| | 44 | 106 | | |
|---|---|---|---|---|
| CreatineKinase | Females: | Females: | | |
| (CK) (U/L) – | <u>0-3 years</u> : | <u>0-3 years</u> : | <u>NA</u> | ≥1.6 X ULN |
| collected only in | 18 | 134 | | |
| TOPMAT-MIG- | <u>4-6 years</u> : | 4-6 years: | | |
| 3006 | 18 | 147 | | |
| | <u>7-9 years</u> :<br>18 | <u>8-9 years:</u><br>295 | | |
| | 10-12 years: | 10-12 years: | | |
| | 18 | 184 | | |
| | <u>13-15 years</u> : | <u>13-15 years</u> : | | |
| | 18 | 187 | | |
| | <u>16-17 years</u> : | <u>16-17 years</u> : | | |
| | 18 | 169 | | |
| | <u>≥18 years:</u><br>18 | ≥18 years:<br>169 | | |
| | Males: | Males: | | |
| | 0-3 years: | 0-3 years: | | |
| | 18 | 163 | | |
| | <u>4-6 years:</u> | <u>4-6 years:</u> | | |
| | 18 | 158 | | |
| | 7-9 years: | 7-9 years: | | |
| | 18 | 354 | | |
| | <u>10-12 years</u> :<br>18 | <u>10-12 years</u> :<br>363 | | |
| | 13-15 years: | 13-15 years: | | |
| | 18 | 363 | | |
| | <u>16-17 years</u> : | <u>16-17 years</u> : | | |
| | 18 | 408 | | |
| | ≥18 years: | ≥18 years: | | |
| | 18 | 198 | | |
| G-Glutamyl | <18 years: | <18 years: | | |
| Transferase(GGT) | 0 | 23 | NA | ≥3 X ULN |
| Glucose (mmol/L) | <16 years: | <16 years: | 40.0 W I I N | > 1.0 W I II N |
| | 3.3 | 5.8 | ≤0.8 X LLN | $\geq$ 1.2 X ULN |
| | <u>≥16 years:</u> 3.9 | ≥16 years:<br>6.4 | (e.g., $\leq$ 2.6 for $\leq$ 16 years and $\leq$ | (e.g., $\geq$ 7.0 for $\leq$ 16 years and $\geq$ 7.7 for $\geq$ |
| | 3.9 | 0.4 | 3.1 for > 16 | 16 years |
| | | | years | 10 30015 |
| | | | , | |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Phosphorus Inorg. (mmol/L) | <18 years:<br>1.03<br>≥18 years: | <18 years:<br>2.10<br>≥18 years: | < 0.8 X LLN | >1.4 X ULN |
|---|---|---|---|---|
| | 0.87 | 1.45 | | |
| Lactate<br>Dehydrogenase<br>(U/L) | <18 years:<br>150<br>≥18 years:<br>0 | <18 years:<br>300<br>≥18 years:<br>220 | NA | > 2 X ULN |
| Potassium<br>(mmol/L) | 3.5 | 5 | <u>≤</u> 3.0 | ≥ 5.7 |
| Sodium(mmol/L) | 135 | 148 | ≤127 | ≥158 |
| Total Protein (g/L) | <6 years:<br>49 | <6 years:<br>81 | ≤0.7 X LLN | ≥1.25 X ULN |
| | <u>≥6 years:</u><br>60 | <u>≥6 years:</u><br>80 | | |
| Triglycerides (mmol/L) | Females: 0-5 years: 0.3616 6-11 years: 0.3955 12-15 years: 0.4633 16-19 years: 0.452 Males: 0-5 years: 0.339 6-11 years: 0.3503 12-15 years: 0.4068 16-19 years: 0.452 | Females: 0-5 years: 1.1187 6-11 years: 1.2882 12-15 years: 1.5594 16-19 years: 1.4464 Males: 0-5 years: 0.9718 6-11 years: 1.2204 12-15 years: 1.5594 16-19 years: 1.8419 | NA | > 1.6 X ULN |
| Uric Acid<br>(umol/L) | 140 | 380 | ≤80 | ≥570 |

| Magnesium | Females: | Females: | < 0.5 | >2 |
|-----------|----------------------|----------------------|-------|-----|
| 8 | <u>1-3 years:</u> | <u>1-3 years:</u> | 10.5 | . 2 |
| | 0.7 | 0.98 | | |
| | <u>4-6 years</u> : | <u>4-6 years</u> : | | |
| | 0.7 | 0.90 | | |
| | <u>7-12 years</u> : | <u>7-12 years</u> : | | |
| | 0.7 | 0.90 | | |
| | <u>13-15 years</u> : | <u>13-15 years</u> : | | |
| | 0.66 | 0.94 | | |
| | <u>16-18 years</u> : | <u>16-18 years</u> : | | |
| | 0.62 | 0.90 | | |
| | Males: | Males: | | |
| | <u>1-3 years:</u> | <u>1-3 years:</u> | | |
| | 0.7 | 0.98 | | |
| | <u>4-6 years</u> : | <u>4-6 years</u> : | | |
| | 0.7 | 0.98 | | |
| | <u>7-12 years</u> : | <u>7-12 years</u> : | | |
| | 0.7 | 0.90 | | |
| | <u>13-15 years</u> : | <u>13-15 years</u> : | | |
| | 0.66 | 0.94 | | |
| | <u>16-18 years</u> : | <u>16-18 years</u> : | | |
| | 0.62 | 0.90 | | |

In addition, the MAL low and high for additional parameters will be as follows:

| Parameter | MAL low | MAL high |
|----------------------|-------------|----------|
| 25 Vitamin D (ng/ml) | <20 | >55 |
| 1, 25 D (pg/ml) | <15 | >90 |
| IGF-1 (nmol/L) | 2-8: <6 | >50 |
| | 9-10: <8 | >65 |
| | 11-12: <15 | >100 |
| | 13-16: <20 | >140 |
| PTH (pg/mL) | 2-7: <40 | >350 |
| | 8-10: <50 | >490 |
| | 11-12: <70 | >750 |
| | 13-16: <100 | >1100 |

The conversion factors for 25 Vitamin D, 1, 25 Vitamin D and PTH are listed below.

| Parameter | Units | Conversion factor |
|-----------------|-----------------|-------------------|
| 25 Vitamin D | nmol/L to ng/mL | 0.4 |
| 1, 25 Vitamin D | Pmol/L to pg/ml | 1.355 |
| PTH | Pmol/L to pg/mL | 9.434 |

## Hematology

| Laboratory<br>Value (SI Unit) | Lower Limit of<br>Normal(LLN)<br>Range | Upper Limit of<br>Normal (ULN)<br>Range | DNPRecommended<br>Markedly<br>Abnormal:Low | DNPRecommended<br>Markedly<br>Abnormal: High |
|---|---|---|---|---|
| Hemoglobin (g/L) | Females: 1-4 years: 109 5-10 years: 119 11-17 years: 119 ≥18 years: 119 Males: 1-4 years: 109 5-10 years: 119 11-17 years: | Females: 1-4 years: 150 5-10 years: 150 11-17 years: 150 ≥18 years: 155 Males: 1-4 years: 150 5-10 years: 150 11-17 years: | ≤90 | ≥180 |
| | 127<br>≥18 years:<br>132 | 170<br>≥18 years:<br>177 | | |

| Hematocrit | Females: | Females: | | |
|---|---|---|---|---|
| (proportion of 1.0) | 1-4 years: | 1-4 years: | <0.85 X LLN | ≥1.15 X ULN |
| | 0.31 | 0.44 | _ | _ |
| | 5-10 years: | 5-10 years: | | |
| | 0.35 | 0.44 | | |
| | <u>11-17 years</u> : | <u>11-17 years</u> : | | |
| | 0.34 | 0.44 | | |
| | ≥18 years:<br>0.35 | ≥18 years:<br>0.47 | | |
| | 0.35<br>Males: | 0.47<br>Males: | | |
| | 1-4 years: | <u>1-4 years:</u> | | |
| | 0.31 | 1-4 years.<br>0.44 | | |
| | <u>5-10 years</u> : | <u>5-10 years</u> : | | |
| | 0.35 | 0.44 | | |
| | <u>11-17 years</u> : | <u>11-17 years</u> : | | |
| | 0.37 | 0.48 | | |
| | ≥18 years:<br>0.40 | ≥18 years:<br>0.52 | | |
| RBC-Total | Females: | Females: | | |
| (10E12/L) | <u>1-4 years</u> : | <u>1-4 years</u> : | ≤0.85 X LLN | ≥1.15 X ULN |
| | 3.8 | 5.2 | | |
| | <u>5-10 years</u> : | <u>5-10 years</u> : | | |
| | 4.1 | 5.2 | | |
| | <u>11-17 years</u> :<br>3.9 | <u>11-17 years</u> :<br>5.1 | | |
| | ≥18 years: | ≥18 years: | | |
| | 4.2 | 5.4 | | |
| | Males: | Males: | | |
| | <u>1-4 years</u> : | <u>1-4 years</u> : | | |
| | 3.8 | 5.5 | | |
| | <u>5-10 years</u> : | <u>5-10 years</u> : | | |
| | 4.3 | 5.2 | | |
| | <u>11-17 years</u> : | <u>11-17 years</u> : | | |
| | 4.3 | 5.6 | | |
| | ≥18 years: | <u>≥18 years:</u> | | |
| | 4.5 | 6.2 | | |

| WBC – Total<br>(10E9/L) | 2-5 years:<br>5<br>6-17 years:<br>4.5<br>≥18 years:<br>4.5 | 2-5 years:<br>15.5<br>6-17 years:<br>13.5<br>≥18 years:<br>11 | < 0.85 X LLN | > 1.15 X ULN |
|---|---|---|---|---|
| Neutrophils—<br>WBCDifferential<br>Count(Proportion<br>of 1) | 0.38 | 0.80 | ≤0.15 | ≥0.90 |
| Lymphocytes—<br>WBCDifferential<br>Count(Proportion<br>of 1) | <u>0.15</u> | 0.40 | ≤0.10 | ≥0.60 |
| Monocytes –<br>WBCDifferential<br>Count(Proportion<br>of 1) | <u>0</u> | <u>0.13</u> | NA | ≥0.20 |
| Eosinophils—<br>WBCDifferential<br>Count(Proportion<br>of 1) | <u>0</u> | 0.08 | NA | ≥0.10 |
| Basophils – WBC<br>Differential Count<br>(Proportion of 1) | 0 | 0.02 | NA | ≥0.06 |
| PlateletCount (x10E9/L) | 150 | 350 | ≤0.75 X LLN | ≥1.3 X ULN |

## 11. URINALYSIS

| Laboratory<br>Value (SI Unit) | Lower Limit of<br>Normal(LLN)<br>Range | Upper Limit of<br>Normal(ULN)<br>Range | Markedly<br>Abnormal:Low | Markedly<br>Abnormal: High |
|---|---|---|---|---|
| РН | 4.5 | 8 | ≤4 | ≥8 |
| Specific Gravity | 1.007 | 1.03 | ≤1.001 | ≥1.035 |

## Appendix 3: AE of clinical interest

| AETERM | AEBODSYS in | AEDECOD (PT) In MedDRA |
|---|---|---|
| | MedDRA 22.0 | 22.1 |
| 5'nucleotidase increased | Investigations | 5'nucleotidase increased |
| Abulia | Psychiatric disorders | Abulia |
| Accommodation disorder | Eye disorders | Accommodation disorder |
| Acidosis | Metabolism and | Acidosis |
| | nutrition disorders | |
| Acidosis hyperchloraemic | Metabolism and | Acidosis hyperchloraemic |
| | nutrition disorders | |
| Acquired epidermolysis bullosa | Skin and | Acquired epidermolysis bullosa |
| | subcutaneous tissue | |
| | disorders | |
| Acquired pigmented | Injury, poisoning and | Acquired pigmented retinopathy |
| retinopathy | procedural | |
| | complications | |
| <b>Activation syndrome</b> | Psychiatric disorders | Activation syndrome |
| Acute generalised | Skin and | Acute generalised |
| exanthematous pustulosis | subcutaneous tissue | exanthematous pustulosis |
| | disorders | |
| Acute hepatic failure | Hepatobiliary | Acute hepatic failure |
| | disorders | |
| Renal failure acute | Renal and urinary | Acute kidney injury |
| | disorders | |
| Adjustment disorder with | Psychiatric disorders | Adjustment disorder with |
| anxiety | | anxiety |
| Adjustment disorder with | Psychiatric disorders | Adjustment disorder with |
| depressed mood | | depressed mood |
| Adjustment disorder with | Psychiatric disorders | Adjustment disorder with mixed |
| mixed anxiety and depressed | | anxiety and depressed mood |
| mood | | |
| Adjustment disorder with | Psychiatric disorders | Adjustment disorder with mixed |
| mixed anxiety and depressed | | anxiety and depressed mood |
| mood | | |
| Affect lability | Psychiatric disorders | Affect lability |
| Agitated depression | Psychiatric disorders | Agitated depression |
| Agitation | Psychiatric disorders | Agitation |
| Alanine aminotransferase | Investigations | Alanine aminotransferase |
| abnormal | | abnormal |
| Alanine aminotransferase | Investigations | Alanine aminotransferase |
| increased | | increased |
| Albumin urine present | Investigations | Albumin urine present |
| Alpha 1 foetoprotein abnormal | Investigations | Alpha 1 foetoprotein abnormal |
| Alpha 1 foetoprotein increased | Investigations | Alpha 1 foetoprotein increased |

| Alpha 1 globulin increased | Investigations | Alpha 1 globulin increased |
|---|---|---|
| Alpha 2 globulin increased | Investigations | Alpha 2 globulin increased |
| Alpha globulin increased | Investigations | Alpha globulin increased |
| Alpha-2 macroglobulin | Investigations | Alpha-2 macroglobulin |
| increased | Investigations | increased |
| Altered state of consciousness | Nervous system | Altered state of consciousness |
| Title ed state of consciousness | disorders | Aircrea state of consciousness |
| Altered visual depth | Eye disorders | Altered visual depth perception |
| perception | Lyc disorders | ritered visual depth perception |
| Amaurosis | Eye disorders | Amaurosis |
| Amaurosis fugax | Eye disorders | Amaurosis fugax |
| Ammonia abnormal | Investigations | Ammonia abnormal |
| Ammonia abnormal | Investigations | Ammonia abnormal |
| Ammonia abnormal Ammonia increased | Investigations | Ammonia increased |
| Ammonia increased | Investigations | Ammonia increased |
| Amnesia | Nervous system<br>disorders | Amnesia |
| CLLL | | |
| Global amnesia | Nervous system | Amnesia |
| | disorders | |
| Angle closure glaucoma | Eye disorders | Angle closure glaucoma |
| Anhedonia | Psychiatric disorders | Anhedonia |
| Anhidrosis | Skin and | Anhidrosis |
| | subcutaneous tissue | |
| | disorders | |
| Anorexia and bulimia | Psychiatric disorders | Anorexia and bulimia syndrome |
| syndrome | | |
| Anorexia and bulimia | Psychiatric disorders | Anorexia and bulimia syndrome |
| syndrome | | |
| Anorexia nervosa | Psychiatric disorders | Anorexia nervosa |
| Anorexia nervosa | Psychiatric disorders | Anorexia nervosa |
| Anterograde amnesia | Nervous system | Anterograde amnesia |
| | disorders | |
| Anticipatory anxiety | Psychiatric disorders | Anticipatory anxiety |
| Antidepressant therapy | Surgical and medical | Antidepressant therapy |
| | procedures | |
| Antimetropia | Eye disorders | Antimetropia |
| Anxiety | Psychiatric disorders | Anxiety |
| Anxiety disorder | Psychiatric disorders | Anxiety disorder |
| Apathy | Psychiatric disorders | Apathy |
| Dysphasia | Nervous system | Aphasia |
| | disorders | |
| Aphonia psychogenic | Nervous system | Aphonia psychogenic |
| | disorders | |
| Apocrine miliaria | Skin and | Apocrine miliaria |
| • | subcutaneous tissue | |
| | disorders | |
| L | 1 | |

| Apraxia | Nervous system | Apraxia |
|---|---|---|
| Ascites | disorders Gastrointestinal | Ascites |
| Ascites | disorders | Ascites |
| A | 3F-0 0 - 0F 0 - 0 | A |
| Aspartate aminotransferase | Investigations | Aspartate aminotransferase |
| abnormal | T (* (* | abnormal |
| Aspartate aminotransferase | Investigations | Aspartate aminotransferase |
| increased | <b>N</b> T | increased |
| Asterixis | Nervous system | Asterixis |
| | disorders | |
| Asterixis | Nervous system | Asterixis |
| | disorders | |
| Asthenia | General disorders and | Asthenia |
| | administration site | |
| | conditions | |
| Astigmatism | Eye disorders | Astigmatism |
| Attention deficit/hyperactivity | Psychiatric disorders | Attention deficit/hyperactivity |
| disorder | | disorder |
| Atypical attention deficit | Psychiatric disorders | Atypical attention deficit |
| syndrome | | syndrome |
| Autoimmune hepatitis | Hepatobiliary | Autoimmune hepatitis |
| | disorders | |
| Beta 2 microglobulin increased | Investigations | Beta 2 microglobulin increased |
| Beta globulin increased | Investigations | Beta globulin increased |
| Bile duct obstruction | Hepatobiliary | Bile duct obstruction |
| | disorders | |
| Bile duct pressure increased | Investigations | Bile duct pressure increased |
| Bile duct stenosis | Hepatobiliary | Bile duct stenosis |
| | disorders | |
| Bile duct stent insertion | Surgical and medical | Bile duct stent insertion |
| | procedures | |
| Bile output abnormal | Investigations | Bile output abnormal |
| Bile output decreased | Investigations | Bile output decreased |
| Biliary cirrhosis | Hepatobiliary | Biliary cirrhosis |
| | disorders | |
| Biliary dyskinesia | Hepatobiliary | Biliary dyskinesia |
| | disorders | |
| Biliary fibrosis | Hepatobiliary | Biliary fibrosis |
| | disorders | |
| Bilirubin conjugated abnormal | Investigations | Bilirubin conjugated abnormal |
| Bilirubin conjugated increased | Investigations | Bilirubin conjugated increased |
| Bilirubin excretion disorder | Hepatobiliary | Bilirubin excretion disorder |
| 1 11 1 32-3 2 - 37-3 | disorders | |
| Bilirubinuria | Renal and urinary | Bilirubinuria |
| | disorders | |
| Biopsy liver abnormal | Investigations | Biopsy liver abnormal |
| 2.5 psj ii vi asilvillai | | 210 poj mier admornia |

| Blepharospasm | Eye disorders | Blepharospasm |
|---|---|---|
| Blindness | Eve disorders | Blindness |
| Blindness cortical | Eye disorders | Blindness cortical |
| Blindness day | Eye disorders | Blindness day |
| Blindness transient | Eye disorders | Blindness transient |
| Blindness traumatic | Injury, poisoning and | Blindness traumatic |
| Dimuness truumute | procedural | Diffusess & unitable |
| | complications | |
| Blindness unilateral | Eye disorders | Blindness unilateral |
| Blister | Skin and | Blister |
| | subcutaneous tissue | |
| | disorders | |
| Blood alkaline phosphatase | Investigations | Blood alkaline phosphatase |
| abnormal | 8 | abnormal |
| Blood alkaline phosphatase | Investigations | Blood alkaline phosphatase |
| increased | | increased |
| Blood bicarbonate abnormal | Investigations | Blood bicarbonate abnormal |
| Blood bicarbonate decreased | Investigations | Blood bicarbonate decreased |
| Blood bilirubin abnormal | Investigations | Blood bilirubin abnormal |
| Blood bilirubin increased | Investigations | Blood bilirubin increased |
| Blood bilirubin unconjugated | Investigations | Blood bilirubin unconjugated |
| increased | | increased |
| Blood cholinesterase abnormal | Investigations | Blood cholinesterase abnormal |
| Blood cholinesterase decreased | Investigations | Blood cholinesterase decreased |
| Blood urine | Investigations | Blood urine |
| Blood urine present | Investigations | Blood urine present |
| Blunted affect | Psychiatric disorders | Blunted affect |
| Body height abnormal | Investigations | Body height abnormal |
| Body height below normal | Investigations | Body height below normal |
| Body height decreased | Investigations | Body height decreased |
| Body mass index decreased | Investigations | Body mass index decreased |
| <b>Body temperature decreased</b> | Investigations | Body temperature decreased |
| <b>Body temperature increased</b> | Investigations | <b>Body temperature increased</b> |
| Bone development abnormal | Musculoskeletal and | Bone development abnormal |
| | connective tissue | |
| | disorders | |
| Bone development abnormal | Musculoskeletal and | Bone development abnormal |
| | connective tissue | |
| | disorders | |
| Bone disorder | Musculoskeletal and | Bone disorder |
| | connective tissue | |
| | disorders | |
| Bone disorder | Musculoskeletal and | Bone disorder |
| | connective tissue | |
| | disorders | |

| Bone formation decreased | Musculoskeletal and connective tissue disorders | Bone formation decreased |
|---|---|---|
| Bone metabolism disorder | Musculoskeletal and connective tissue disorders | Bone metabolism disorder |
| Bone pain | Musculoskeletal and connective tissue disorders | Bone pain |
| Borderline glaucoma | Eye disorders | Borderline glaucoma |
| Borderline mental impairment | Nervous system disorders | Borderline mental impairment |
| Bradyphrenia | Psychiatric disorders | Bradyphrenia |
| Bromosulphthalein test abnormal | Investigations | Bromosulphthalein test abnormal |
| Budd-Chiari syndrome | Hepatobiliary<br>disorders | Budd-Chiari syndrome |
| Cachexia | Metabolism and nutrition disorders | Cachexia |
| Calculus bladder | Renal and urinary disorders | Calculus bladder |
| Calculus bladder | Renal and urinary disorders | Calculus bladder |
| Calculus prostatic | Reproductive system and breast disorders | Calculus prostatic |
| Calculus prostatic | Reproductive system and breast disorders | Calculus prostatic |
| Calculus ureteric | Renal and urinary disorders | Ureterolithiasis |
| Calculus urethral | Renal and urinary disorders | Calculus urethral |
| Calculus urinary | Renal and urinary disorders | Calculus urinary |
| Carbon dioxide decreased | Investigations | Carbon dioxide decreased |
| Cardiac arrest | Cardiac disorders | Cardiac arrest |
| Cardiac death | General disorders and administration site conditions | Cardiac death |
| Cardiac failure | Cardiac disorders | Cardiac failure |
| Cardiac failure acute | Cardiac disorders | Cardiac failure acute |
| Cardiac failure chronic | Cardiac disorders | Cardiac failure chronic |
| Cardiac failure congestive | Cardiac disorders | Cardiac failure congestive |
| Cardiac output decreased | Investigations | Cardiac output decreased |
| Cardiac ventriculogram abnormal | Investigations | Cardiac ventriculogram abnormal |

| | T 4: 4: | |
|---|---|---|
| Cardiac ventriculogram left | Investigations | Cardiac ventriculogram left |
| abnormal | | abnormal |
| Cells in urine | Investigations | Cells in urine |
| Change in sustained attention | Psychiatric disorders | Change in sustained attention |
| <b>Charles Bonnet syndrome</b> | Eye disorders | Charles Bonnet syndrome |
| Childhood disintegrative | Psychiatric disorders | Child-Pugh-Turcotte score |
| disorder | | increased |
| Child-Pugh-Turcotte score | Investigations | |
| increased | | |
| Chills | General disorders and | Chills |
| | administration site | |
| | conditions | |
| Chloropsia | Eye disorders | Chloropsia |
| Cholaemia | Hepatobiliary | Cholaemia |
| | disorders | |
| Cholelithiasis | Hepatobiliary | Cholelithiasis |
| Cholentinasis | disorders | Cholentinasis |
| Cholelithiasis obstructive | Hepatobiliary | Cholelithiasis obstructive |
| Cholentinasis obstructive | disorders | Cholenthiasis obstructive |
| Chalalith atomy | | Chalalith atomy |
| Cholelithotomy | Surgical and medical | Cholelithotomy |
| | procedures | |
| Cholestasis | Hepatobiliary | Cholestasis |
| | disorders | |
| Cholestatic liver injury | Hepatobiliary | Cholestatic liver injury |
| | disorders | |
| Cholestatic liver injury | Hepatobiliary | Cholestatic liver injury |
| | disorders | |
| Cholestatic pruritus | Skin and | Cholestatic pruritus |
| | subcutaneous tissue | |
| | disorders | |
| Chorioretinitis | Infections and | Chorioretinitis |
| | infestations | |
| Choroid tubercles | Infections and | Choroid tubercles |
| | infestations | |
| Choroiditis | Eye disorders | Choroiditis |
| Urine colour abnormal | Renal and urinary | Chromaturia |
| | disorders | |
| Chronic fatigue syndrome | General disorders and | Chronic fatigue syndrome |
| | administration site | , |
| | conditions | |
| Chronic hepatic failure | Hepatobiliary | Chronic hepatic failure |
| | disorders | |
| Chronic hepatitis | Hepatobiliary | Chronic hepatitis |
| - порини | disorders | om ome nepatitis |
| Ciliary muscle spasm | Eye disorders | Ciliary muscle spasm |
| Circumstantiality | Psychiatric disorders | Circumstantiality |
| Circumstantianty | 1 Sychian ic disorders | Circumstantianty |

| Clang associations | Psychiatric disorders | Clang associations |
|---|---|---|
| Cognitive disorder | Nervous system | Cognitive disorder |
| | disorders | |
| Cold sweat | Skin and | Cold sweat |
| | subcutaneous tissue | |
| | disorders | |
| Coma | Nervous system | Coma |
| | disorders | |
| Coma hepatic | Nervous system | Coma hepatic |
| | disorders | • |
| Communication disorder | Psychiatric disorders | Communication disorder |
| Completed suicide | Psychiatric disorders | Completed suicide |
| Confabulation | Psychiatric disorders | Confabulation |
| Confusional arousal | Psychiatric disorders | Confusional arousal |
| Confusional state | Psychiatric disorders | Confusional state |
| Confusional state | Psychiatric disorders | Confusional state |
| Conjunctival ulcer | Eye disorders | Conjunctival ulcer |
| Conjunctivitis | Infections and | Conjunctivitis |
| | infestations | 0.01134110017111111 |
| Consciousness fluctuating | Nervous system | Consciousness fluctuating |
| | disorders | g |
| Constricted affect | Psychiatric disorders | Constricted affect |
| Coprolalia | Psychiatric disorders | Coprolalia |
| Corneal deposits | Eye disorders | Corneal deposits |
| Corneal exfoliation | Eye disorders | Corneal exfoliation |
| Corneal oedema | Eye disorders | Corneal oedema |
| Corneal opacity | Eye disorders | Corneal opacity |
| Corneal perforation | Eye disorders | Corneal perforation |
| Creatine urine abnormal | Investigations | Creatine urine abnormal |
| Creatine urine decreased | Investigations | Creatine urine decreased |
| Creatine urine increased | Investigations | Creatine urine increased |
| Creatinine urine decreased | Investigations | Creatinine urine decreased |
| Creatinine urine increased | Investigations | Creatinine urine increased |
| Crocodile tears syndrome | Nervous system | Crocodile tears syndrome |
| , | disorders | |
| Crying | General disorders and | Crying |
| | administration site | |
| | conditions | |
| Cryptogenic cirrhosis | Hepatobiliary | Cryptogenic cirrhosis |
| | disorders | |
| Crystal urine | Investigations | Crystal urine |
| Crystal urine present | Investigations | Crystal urine present |
| Cyanopsia | Eye disorders | Cyanopsia |
| Cycloplegia | Eye disorders | Cycloplegia |
| Cysteine urine present | Investigations | Cysteine urine present |
| | Investigations | Cystine urine present |

| Daydreaming | Psychiatric disorders | Daydreaming |
|---|---|---|
| Deaf mutism | Congenital, familial | Deaf mutism |
| | and genetic disorders | |
| Decreased activity | General disorders and | Decreased activity |
| 2 001 000000 0001 1003 | administration site | |
| | conditions | |
| Anorexia | Metabolism and | Decreased appetite |
| THOTCALL | nutrition disorders | Decreased appeare |
| Anorexia | Metabolism and | Decreased appetite |
| Anorcaia | nutrition disorders | Decreased appetite |
| Decreased interest | Psychiatric disorders | Decreased interest |
| Dehydration Dehydration | Metabolism and | Dehydration Dehydration |
| Denyuration | nutrition disorders | Denyuration |
| Delirium | | Delirium |
| | Psychiatric disorders | |
| Depressed level of | Nervous system | Depressed level of consciousness |
| consciousness | disorders | D 1 1 |
| Depressed mood | Psychiatric disorders | Depressed mood |
| Depression | Psychiatric disorders | Depression |
| Depression postoperative | Injury, poisoning and | Depression postoperative |
| | procedural | |
| | complications | |
| Depression suicidal | Psychiatric disorders | Depression suicidal |
| Depressive symptom | Psychiatric disorders | Depressive symptom |
| Derailment | Psychiatric disorders | Derailment |
| Dermatitis bullous | Skin and | Dermatitis bullous |
| | subcutaneous tissue | |
| | disorders | |
| Dermatitis exfoliative | Skin and | Dermatitis exfoliative |
| | subcutaneous tissue | |
| | disorders | |
| Dermatitis exfoliative | Skin and | Dermatitis exfoliative |
| generalised | subcutaneous tissue | generalised |
| | disorders | |
| Detachment of retinal pigment | Eye disorders | Detachment of retinal pigment |
| epithelium | | epithelium |
| <b>Developmental coordination</b> | Nervous system | Developmental coordination |
| disorder | disorders | disorder |
| Developmental delay | General disorders and | Developmental delay |
| Ţ | administration site | |
| | conditions | |
| Diplopia | Eye disorders | Diplopia |
| Disorientation | Psychiatric disorders | Disorientation |
| Disorientation | Psychiatric disorders | Disorientation |
| Dissociative amnesia | Psychiatric disorders | Dissociative amnesia |
| Distractibility | Psychiatric disorders | Distractibility |
| - V | | - <del>/</del> |

| Disturbance in attention | Nervous system<br>disorders | Disturbance in attention |
|---|---|---|
| Disturbance in attention | Nervous system<br>disorders | Disturbance in attention |
| Drug eruption | Skin and subcutaneous tissue disorders | Drug eruption |
| Drug rash with eosinophilia and systemic symptoms | Skin and subcutaneous tissue disorders | Drug reaction with eosinophilia and systemic symptoms |
| Dry eye | Eye disorders | Dry eye |
| Keratoconjunctivitis sicca | Eye disorders | Dry eye |
| Keratoconjunctivitis sicca | Eye disorders | Dry eye |
| Dry skin | Skin and subcutaneous tissue disorders | Dry skin |
| <b>Duodenal varices</b> | Gastrointestinal disorders | <b>Duodenal varices</b> |
| Dwarfism | Musculoskeletal and connective tissue disorders | Dwarfism |
| Dysarthria | Nervous system<br>disorders | Dysarthria |
| Dysgraphia | Nervous system disorders | Dysgraphia |
| Dyshidrosis | Skin and subcutaneous tissue disorders | Dyshidrotic eczema |
| Dyshidrosis | Skin and subcutaneous tissue disorders | Dyshidrotic eczema |
| Dyslalia | Nervous system disorders | Dyslalia |
| Dysmetropsia | Eye disorders | Dysmetropsia |
| Dysphemia | Psychiatric disorders | Dysphemia |
| Dysphonia | Respiratory, thoracic and mediastinal disorders | Dysphonia |
| Dysphonia psychogenic | Nervous system disorders | Dysphonia psychogenic |
| Dysphoria | Psychiatric disorders | Dysphoria |
| Dysprosody | Nervous system<br>disorders | Dysprosody |
| Dyssomnia | Psychiatric disorders | Dyssomnia |
| Dysthymic disorder | Psychiatric disorders | Persistent depressive disorder |
| Echolalia | Psychiatric disorders | Echolalia |

| Electric shock | Injury, poisoning and | Electric shock |
|---|---|---|
| Dicetife shock | procedural | Licetic shock |
| | complications | |
| Electroconvulsive therapy | Surgical and medical | Electroconvulsive therapy |
| Dicetioconvalsive therapy | procedures | Liceti dedit varsive therapy |
| Electroencephalogram | Investigations | Electroencephalogram |
| abnormal | Investigations | abnormal |
| Emotional distress | Psychiatric disorders | Emotional distress |
| <b>Encephalopathy</b> | Nervous system | Encephalopathy |
| Encephalopathy | disorders | Encephalopathy |
| Epidermal necrosis | Skin and | Epidermal necrosis |
| Epidei mai necrosis | subcutaneous tissue | Epidei mai neci osis |
| | disorders | |
| Epidermolysis | Congenital, familial | Epidermolysis |
| Epidei morysis | and genetic disorders | Lpiuci morysis |
| Epidermolysis bullosa | Congenital, familial | Epidermolysis bullosa |
| Epidei moiysis bunosa | and genetic disorders | Epidei morysis bunosa |
| <b>Epiphyses delayed fusion</b> | Musculoskeletal and | Epiphyses delayed fusion |
| Epiphyses delayed fusion | connective tissue | Epiphyses delayed fusion |
| | disorders | |
| Erythema multiforme | Skin and | Erythema multiforme |
| Elythema mutulorme | subcutaneous tissue | El ythema multifol me |
| | disorders | |
| Erythropsia | Eye disorders | Erythropsia |
| Excessive eye blinking | Eye disorders | Excessive eye blinking |
| Exfoliative rash | Skin and | Exfoliative rash |
| Eximative rash | subcutaneous tissue | Eximative rash |
| | disorders | |
| Eye disorder | Eye disorders | Eye disorder |
| Eye pain | Eye disorders | Eye pain |
| Eyelid function disorder | Eye disorders | Eyelid function disorder |
| Eyelid ptosis | Eye disorders | Eyelid ptosis |
| Eyelid retraction | Eye disorders | Eyelid retraction |
| Failure to thrive | Metabolism and | Failure to thrive |
| ranuic to thrive | nutrition disorders | Tanuic to thrive |
| Fanconi syndrome | Congenital, familial | Fanconi syndrome |
| i ancom synarome | and genetic disorders | i ancom synarome |
| Fanconi syndrome acquired | Renal and urinary | Fanconi syndrome acquired |
| ancom synarome acquired | disorders | i ancom synarome acquired |
| Fanconi syndrome acquired | Renal and urinary | Fanconi syndrome acquired |
| ancom synarome acquired | disorders | i ancom synarome acquired |
| Fatigue | General disorders and | Fatigue |
| 1 uugue | administration site | - ungue |
| | conditions | |
| | Conultions | |

| Feeling cold | General disorders and | Feeling cold |
|---|---|---|
| | administration site | |
| | conditions | |
| Feeling drunk | General disorders and | Feeling drunk |
| | administration site | |
| B 1 | conditions | |
| Feeling guilty | Psychiatric disorders | Feeling guilty |
| Feeling hot | General disorders and administration site | Feeling hot |
| | conditions | |
| Feeling of body temperature | General disorders and | Feeling of body temperature |
| change | administration site | change |
| chunge | conditions | chunge |
| Feeling of despair | Psychiatric disorders | Feeling of despair |
| Feelings of worthlessness | Psychiatric disorders | Feelings of worthlessness |
| Flight of ideas | Psychiatric disorders | Flight of ideas |
| Floppy iris syndrome | Injury, poisoning and | Floppy iris syndrome |
| | procedural | |
| | complications | |
| Flushing | Vascular disorders | Flushing |
| Folliculitis | Infections and | Folliculitis |
| | infestations | |
| Fracture delayed union | Musculoskeletal and | Fracture delayed union |
| | connective tissue<br>disorders | |
| Fracture malunion | Musculoskeletal and | Fracture malunion |
| Tracture maiumon | connective tissue | Tracture maiumon |
| | disorders | |
| Fracture nonunion | Musculoskeletal and | Fracture nonunion |
| | connective tissue | |
| | disorders | |
| Fundoscopy | Investigations | Fundoscopy |
| Fundoscopy abnormal | Investigations | Fundoscopy abnormal |
| Galactose elimination capacity | Investigations | Galactose elimination capacity |
| test abnormal | | test abnormal |
| Galactose elimination capacity | Investigations | Galactose elimination capacity |
| test decreased | TT ( 1 'P' | test decreased |
| Gallbladder cholesterolosis | Hepatobiliary | Gallbladder cholesterolosis |
| Gallbladder disorder | disorders | Gallbladder disorder |
| Gandiadder disorder | Hepatobiliary<br>disorders | Gambiaduer disorder |
| Gallbladder enlargement | Hepatobiliary | Gallbladder enlargement |
| Gambiaddel emai gement | disorders | Gambiauuci emai gement |
| Gallbladder fistula | Hepatobiliary | Gallbladder fistula |
| | disorders | |
| | | 1 |

| Gallbladder mucocoele | Hepatobiliary | Gallbladder mucocoele |
|---|---|---|
| | disorders | |
| Gallbladder necrosis | Hepatobiliary | Gallbladder necrosis |
| | disorders | |
| Gallbladder non-functioning | Hepatobiliary | Gallbladder hypofunction |
| | disorders | |
| Gallbladder obstruction | Hepatobiliary | Gallbladder obstruction |
| | disorders | |
| Gallbladder oedema | Hepatobiliary | Gallbladder oedema |
| | disorders | |
| Gallbladder pain | Hepatobiliary | Biliary colic |
| | disorders | |
| Gamma-glutamyltransferase | Investigations | Gamma-glutamyltransferase |
| abnormal | | abnormal |
| Gamma-glutamyltransferase | Investigations | Gamma-glutamyltransferase |
| increased | | increased |
| Gastric varices | Gastrointestinal | Gastric varices |
| | disorders | |
| Generalised anxiety disorder | Psychiatric disorders | Generalised anxiety disorder |
| Genital ulceration | Reproductive system | Genital ulceration |
| | and breast disorders | |
| Gianotti-Crosti syndrome | Infections and | Gianotti-Crosti syndrome |
| | infestations | |
| Glare | Eye disorders | Glare |
| Glaucoma | Eye disorders | Glaucoma |
| Glaucomatous optic disc | Eye disorders | Glaucomatous optic disc |
| - | 1 * | - |
| atrophy | | atrophy |
| atrophy Globulin urine present | Investigations | atrophy Globulin urine present |
| atrophy Globulin urine present Globulins increased | Investigations Investigations | atrophy Globulin urine present Globulins increased |
| atrophy Globulin urine present Globulins increased Glucose urine | Investigations Investigations Investigations | atrophy Globulin urine present Globulins increased Glucose urine |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present | Investigations Investigations Investigations Investigations | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased | Investigations Investigations Investigations Investigations Investigations | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy | Investigations Investigations Investigations Investigations Investigations Investigations | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal | Investigations | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy | Investigations Hepatobiliary | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease | Investigations Hepatobiliary disorders | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal | Investigations Hepatobiliary disorders Musculoskeletal and | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease | Investigations Hepatobiliary disorders Musculoskeletal and connective tissue | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease Growth retardation | Investigations Hepatobiliary disorders Musculoskeletal and connective tissue disorders | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease Growth retardation |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease Growth retardation Guanase increased | Investigations Hepatobiliary disorders Musculoskeletal and connective tissue disorders Investigations | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease Growth retardation Guanase increased |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease Growth retardation | Investigations Hepatobiliary disorders Musculoskeletal and connective tissue disorders Investigations Renal and urinary | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease Growth retardation |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease Growth retardation Guanase increased Haematuria | Investigations Hepatobiliary disorders Musculoskeletal and connective tissue disorders Investigations Renal and urinary disorders | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease Growth retardation Guanase increased Haematuria |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease Growth retardation Guanase increased Haematuria Haemoglobin urine | Investigations Hepatobiliary disorders Musculoskeletal and connective tissue disorders Investigations Renal and urinary disorders Investigations | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease Growth retardation Guanase increased Haematuria Haemoglobin urine |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease Growth retardation Guanase increased Haematuria Haemoglobin urine Haemoglobin urine present | Investigations Hepatobiliary disorders Musculoskeletal and connective tissue disorders Investigations Renal and urinary disorders Investigations Investigations Investigations Investigations | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease Growth retardation Guanase increased Haematuria Haemoglobin urine Haemoglobin urine present |
| atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease Growth retardation Guanase increased Haematuria Haemoglobin urine | Investigations Hepatobiliary disorders Musculoskeletal and connective tissue disorders Investigations Renal and urinary disorders Investigations | atrophy Globulin urine present Globulins increased Glucose urine Glucose urine present Glyceric acid urine increased Gonioscopy Gonioscopy abnormal Granulomatous liver disease Growth retardation Guanase increased Haematuria Haemoglobin urine |

| Haemorrhagic hepatic cyst | Hepatobiliary<br>disorders | Haemorrhagic hepatic cyst |
|---|---|---|
| Halo vision | Eye disorders | Halo vision |
| Heat exhaustion | Injury, poisoning and procedural complications | Heat exhaustion |
| Heat illness | Injury, poisoning and procedural complications | Heat illness |
| Heat oedema | Injury, poisoning and procedural complications | Heat oedema |
| Heat stroke | Injury, poisoning and procedural complications | Heat stroke |
| Hemianopia | Nervous system disorders | Hemianopia |
| Hemianopia heteronymous | Nervous system disorders | Hemianopia heteronymous |
| Hemianopia homonymous | Nervous system disorders | Hemianopia homonymous |
| Hemiapraxia | Nervous system disorders | Hemiapraxia |
| Hepaplastin abnormal | Investigations | Hepaplastin abnormal |
| Hepaplastin decreased | Investigations | Hepaplastin decreased |
| Hepatic atrophy | Hepatobiliary disorders | Hepatic atrophy |
| Hepatic calcification | Hepatobiliary<br>disorders | Hepatic calcification |
| Hepatic cirrhosis | Hepatobiliary disorders | Hepatic cirrhosis |
| Hepatic congestion | Hepatobiliary disorders | Hepatic congestion |
| Hepatic encephalopathy | Nervous system disorders | Hepatic encephalopathy |
| Hepatic encephalopathy | Surgical and medical | Hepatic encephalopathy |
| prophylaxis | procedures | prophylaxis |
| Hepatic enzyme abnormal | Investigations | Hepatic enzyme abnormal |
| Hepatic enzyme decreased | Investigations | Hepatic enzyme decreased |
| Hepatic enzyme increased | Investigations | Hepatic enzyme increased |
| Hepatic failure | Hepatobiliary<br>disorders | Hepatic failure |
| Hepatic fibrosis | Hepatobiliary<br>disorders | Hepatic fibrosis |
| Hepatic function abnormal | Hepatobiliary<br>disorders | Hepatic function abnormal |

| Hepatic haemorrhage | Hepatobiliary | Hepatic haemorrhage |
|---|---|---|
| Transition in the | disorders | The state of the s |
| Hepatic hydrothorax | Respiratory, thoracic | Hepatic hydrothorax |
| ı v | and mediastinal | |
| | disorders | |
| Hepatic infarction | Hepatobiliary | Hepatic infarction |
| - | disorders | |
| Hepatic infiltration | Hepatobiliary | Hepatic infiltration eosinophilic |
| eosinophilic | disorders | |
| Hepatic lesion | Hepatobiliary | Hepatic lesion |
| | disorders | |
| Hepatic mass | Hepatobiliary | Hepatic mass |
| | disorders | |
| Hepatic necrosis | Hepatobiliary | Hepatic necrosis |
| | disorders | |
| Hepatic pain | Hepatobiliary | Hepatic pain |
| | disorders | |
| Hepatic steatosis | Hepatobiliary | Hepatic steatosis |
| | disorders | |
| Cytolytic hepatitis | Hepatobiliary | Hepatitis |
| | disorders | |
| Hepatitis | Hepatobiliary | Hepatitis |
| | disorders | |
| Hepatitis acute | Hepatobiliary | Hepatitis B |
| | disorders | |
| Hepatitis fulminant | Hepatobiliary | Hepatitis chronic active |
| | disorders | |
| Hepatitis toxic | Hepatobiliary | Hepatitis toxic |
| | disorders | |
| Hepatobiliary disease | Hepatobiliary | Hepatobiliary disease |
| | disorders | |
| Hepatobiliary scan abnormal | Investigations | Hepatobiliary scan abnormal |
| Hepatocellular foamy cell | Hepatobiliary | Hepatocellular foamy cell |
| syndrome | disorders | syndrome |
| Hepatocellular injury | Hepatobiliary | Hepatocellular injury |
| TT 4 | disorders | |
| Hepatomegaly | Hepatobiliary | Hepatomegaly |
| W4 | disorders | Transferrale 1 |
| Hepatopulmonary syndrome | Respiratory, thoracic | Hepatopulmonary syndrome |
| | and mediastinal | |
| Honotowonal fallows | disorders | Honotowonal fallows |
| Hepatorenal failure | Hepatobiliary | Hepatorenal failure |
| Honotowonal averdesees | disorders | Hanatawanal avy duama |
| Hepatorenal syndrome | Hepatobiliary | Hepatorenal syndrome |
| | disorders | |

| Hepatosplenomegaly | Hepatobiliary<br>disorders | Hepatosplenomegaly |
|---|---|---|
| Hepatotoxicity | Hepatobiliary<br>disorders | Hepatotoxicity |
| Hidradenitis | Skin and subcutaneous tissue disorders | Hidradenitis |
| Hippus | Eye disorders | Hippus |
| Holmes-Adie pupil | Eye disorders | Holmes-Adie pupil |
| Homocysteine urine | Investigations | Homocysteine urine |
| Homocysteine urine present | Investigations | Homocysteine urine present |
| Hot flush | Vascular disorders | Hot flush |
| Hydrocholecystis | Hepatobiliary<br>disorders | Hydrocholecystis |
| Hydronephrosis | Renal and urinary disorders | Hydronephrosis |
| Hydronephrosis repair | Surgical and medical procedures | Hydronephrosis repair |
| Hyperammonaemia | Metabolism and nutrition disorders | Hyperammonaemia |
| Hyperammonaemic | Nervous system | Hyperammonaemic |
| encephalopathy | disorders | encephalopathy |
| Hyperbilirubinaemia | Hepatobiliary<br>disorders | Hyperbilirubinaemia |
| Hypercalcaemia | Metabolism and nutrition disorders | Hypercalcaemia |
| Hypercalcaemic nephropathy | Renal and urinary | Hypercalcaemic nephropathy |
| Hypercalciuria | Renal and urinary disorders | Hypercalciuria |
| Hypercholia | Hepatobiliary<br>disorders | Hypercholia |
| Hypergammaglobulinaemia | Blood and lymphatic system disorders | Hypergammaglobulinaemia |
| Hyperglobulinaemia | Blood and lymphatic system disorders | Hyperglobulinaemia |
| Hyperhidrosis | Skin and subcutaneous tissue disorders | Hyperhidrosis |
| Hypermetropia | Eye disorders | Hypermetropia |
| Hyperplastic cholecystopathy | Hepatobiliary<br>disorders | Hyperplastic cholecystopathy |
| Hyperpyrexia | General disorders and administration site conditions | Hyperpyrexia |

| Hypersomnia | Nervous system<br>disorders | Hypersomnia |
|---|---|---|
| Hyperthermia | General disorders and administration site conditions | Hyperthermia |
| Hyperthermia malignant | General disorders and administration site conditions | Hyperthermia malignant |
| Hypertransaminasaemia | Hepatobiliary disorders | Hypertransaminasaemia |
| Hyperventilation | Respiratory, thoracic and mediastinal disorders | Hyperventilation |
| Hyphaema | Eye disorders | Hyphaema |
| Hypoalbuminaemia | Metabolism and nutrition disorders | Hypoalbuminaemia |
| Hypohidrosis | Skin and subcutaneous tissue disorders | Hypohidrosis |
| Hypophosphataemia | Metabolism and nutrition disorders | Hypophosphataemia |
| Hypophosphataemic rickets | Musculoskeletal and connective tissue disorders | Hypophosphataemic osteomalacia |
| Hypophosphatasia | Congenital, familial and genetic disorders | Hypophosphatasia |
| Hyposomnia | Psychiatric disorders | Hyposomnia |
| Hypothermia | General disorders and administration site conditions | Hypothermia |
| <b>Icterus index increased</b> | Investigations | Icterus index increased |
| Illogical thinking | Psychiatric disorders | Illogical thinking |
| Impaired self-care | General disorders and administration site conditions | Impaired self-care |
| Incoherent | Nervous system disorders | Incoherent |
| Initial insomnia | Psychiatric disorders | Initial insomnia |
| Intentional self-injury | Psychiatric disorders | Intentional self-injury |
| Intentional self-injury | Psychiatric disorders | Intentional self-injury |
| Iridoplegia | Eye disorders | Iridoplegia |
| Iritis | Eye disorders | Iritis |
| Ischaemic hepatitis | Hepatobiliary disorders | Ischaemic hepatitis |
| Jaundice | Hepatobiliary disorders | Jaundice |

| Jaundice cholestatic | Hepatobiliary | Jaundice cholestatic |
|---|---|---|
| | disorders | |
| Jaundice hepatocellular | Hepatobiliary | Jaundice hepatocellular |
| - | disorders | - |
| Judgement impaired | Nervous system | Judgement impaired |
| | disorders | |
| Kayser-Fleischer ring | Eye disorders | Kayser-Fleischer ring |
| Keratitis | Eye disorders | Keratitis |
| Kussmaul respiration | Respiratory, thoracic | Kussmaul respiration |
| | and mediastinal | |
| | disorders | |
| Lack of spontaneous speech | Psychiatric disorders | Lack of spontaneous speech |
| Lacrimal disorder | Eye disorders | Lacrimal disorder |
| Lacrimation decreased | Eye disorders | Lacrimation decreased |
| Lacrimation increased | Eye disorders | Lacrimation increased |
| Lactic acidosis | Metabolism and | Lactic acidosis |
| | nutrition disorders | |
| Expressive language disorder | Nervous system | Language disorder |
| | disorders | |
| Mixed receptive-expressive | Nervous system | Language disorder |
| language disorder | disorders | |
| Laurence-Moon-Bardet-Biedl | Congenital, familial | Laurence-Moon-Bardet-Biedl |
| syndrome | and genetic disorders | syndrome |
| Learning disability | Social circumstances | Learning disability |
| Learning disorder | Psychiatric disorders | Learning disorder |
| Lenticular opacities | Eye disorders | Lenticular opacities |
| Lethargy | Nervous system | Lethargy |
| | disorders | |
| Leucine aminopeptidase | Investigations | Leucine aminopeptidase |
| increased | D 11 1 1 | increased |
| Libido decreased | Psychiatric disorders | Libido decreased |
| Libido disorder | Psychiatric disorders | Libido disorder |
| Libido increased | Psychiatric disorders | Libido increased |
| Lip exfoliation | Gastrointestinal | Lip exfoliation |
| T · A | disorders | 1:4 |
| Listless | Psychiatric disorders | Listless |
| Liver disorder | Hepatobiliary | Liver disorder |
| Liver from attended at | disorders | Times from Alice 4 and al |
| Liver function test abnormal | Investigations | Liver function test abnormal Liver induration |
| Liver induration | Hepatobiliary disorders | Liver induration |
| Liver injury | Hepatobiliary | Liver injury |
| | disorders | |
| Liver palpable subcostal | Investigations | Liver palpable |
| Liver tenderness | Hepatobiliary | Liver tenderness |
| | disorders | |
| | disorders | |

| Cluttering | Psychiatric disorders | Logorrhoea |
|---|---|---|
| Loose associations | Psychiatric disorders | Loose associations |
| Loss of consciousness | Nervous system | Loss of consciousness |
| 2000 01 0010010 10010 | disorders | |
| Loss of libido | Psychiatric disorders | Loss of libido |
| Loss of visual contrast | Eye disorders | Loss of visual contrast |
| sensitivity | | sensitivity |
| Low cardiac output syndrome | Cardiac disorders | Low cardiac output syndrome |
| Lupoid hepatic cirrhosis | Hepatobiliary | Lupoid hepatic cirrhosis |
| | disorders | |
| Macular cyst | Eye disorders | Macular cyst |
| Macular degeneration | Eye disorders | Macular degeneration |
| Macular hole | Eye disorders | Macular hole |
| Macular ischaemia | Eye disorders | Macular ischaemia |
| Macular oedema | Eye disorders | Macular oedema |
| Macular opacity | Eye disorders | Macular opacity |
| Macular pseudohole | Eye disorders | Macular pseudohole |
| Macular scar | Eye disorders | Macular scar |
| Macular vasospasm | Eye disorders | Macular vasospasm |
| Maculopathy | Eye disorders | Maculopathy |
| Major depression | Psychiatric disorders | Major depression |
| Memory impairment | Nervous system | Memory impairment |
| | disorders | |
| Menopausal depression | Psychiatric disorders | Menopausal depression |
| Mental impairment | Nervous system | Mental impairment |
| | disorders | |
| Mental retardation | Nervous system | Intellectual disability |
| | disorders | |
| Metabolic acidosis | Metabolism and | Metabolic acidosis |
| | nutrition disorders | |
| Metamorphopsia | Eye disorders | Metamorphopsia |
| Microlithiasis | General disorders and | Lithiasis |
| | administration site | |
| | conditions | |
| Middle insomnia | Psychiatric disorders | Middle insomnia |
| Mikulicz's disease | Gastrointestinal | Mikulicz's disease |
| | disorders | |
| Mikulicz's syndrome | Gastrointestinal | Mikulicz's syndrome |
| | disorders | |
| Mild mental retardation | Nervous system | Intellectual disability |
| 3.500 | disorders | 1200 |
| Milia | Skin and | Milia |
| | subcutaneous tissue | |
| | disorders | |

| Heat rash | Skin and | Miliaria |
|---|---|---|
| | subcutaneous tissue | |
| | disorders | |
| Miosis | Eye disorders | Miosis |
| Mitochondrial aspartate | Investigations | Mitochondrial aspartate |
| aminotransferase increased | 111 ( 03 01 9 11 0 11 3 | aminotransferase increased |
| Mixed hepatocellular | Neoplasms benign, | Mixed hepatocellular |
| cholangiocarcinoma | malignant and | cholangiocarcinoma |
| enoungioeur enronnu | unspecified (incl cysts | enoungioeur emoniu |
| | and polyps) | |
| Mixed liver injury | Hepatobiliary | Mixed liver injury |
| | disorders | |
| Moderate mental retardation | Nervous system | Intellectual disability |
| 1710 del del meneral l'ettal dution | disorders | |
| Molar ratio of total branched- | Investigations | Molar ratio of total branched- |
| chain amino acid to tyrosine | | chain amino acid to tyrosine |
| Mood altered | Psychiatric disorders | Mood altered |
| Mood swings | Psychiatric disorders | Mood swings |
| Morose | Psychiatric disorders | Morose |
| Mouth ulceration | Gastrointestinal | Mouth ulceration |
| | disorders | |
| Mucocutaneous ulceration | Skin and | Mucocutaneous ulceration |
| | subcutaneous tissue | |
| | disorders | |
| Mucosa vesicle | General disorders and | Mucosa vesicle |
| | administration site | |
| | conditions | |
| Mucosal erosion | General disorders and | Mucosal erosion |
| | administration site | |
| | conditions | |
| Mucosal exfoliation | General disorders and | Mucosal exfoliation |
| | administration site | |
| | conditions | |
| Mucosal necrosis | General disorders and | Mucosal necrosis |
| | administration site | |
| | conditions | |
| Mucosal ulceration | General disorders and | Mucosal ulceration |
| | administration site | |
| | conditions | |
| Musculoskeletal chest pain | Musculoskeletal and | Musculoskeletal chest pain |
| | connective tissue | |
| | disorders | |
| Musculoskeletal pain | Musculoskeletal and | Musculoskeletal pain |
| | connective tissue | |
| 75.0 | disorders | 77. |
| Mutism | Psychiatric disorders | Mutism |

| Mydriasis | Eye disorders | Mydriasis |
|---|---|---|
| Myopia | Eye disorders | Myopia |
| Necrotising retinitis | Eye disorders | Necrotising retinitis |
| Negative cardiac inotropic effect | Cardiac disorders | Negative cardiac inotropic effect |
| Negative thoughts | Psychiatric disorders | Negative thoughts |
| Neglect of personal appearance | Psychiatric disorders | Neglect of personal appearance |
| Neologism | Psychiatric disorders | Neologism |
| Nephrocalcinosis | Renal and urinary | Nephrocalcinosis |
| • | disorders | ' |
| Nephrocalcinosis | Renal and urinary | Nephrocalcinosis |
| 1 | disorders | |
| Nephrolithiasis | Renal and urinary | Nephrolithiasis |
| • | disorders | ' |
| Nephrolithiasis | Renal and urinary | Nephrolithiasis |
| | disorders | |
| Nervousness | Psychiatric disorders | Nervousness |
| Neurodevelopmental disorder | Psychiatric disorders | Neurodevelopmental disorder |
| Neuroleptic malignant | Nervous system | Neuroleptic malignant |
| syndrome | disorders | syndrome |
| Night blindness | Eye disorders | Night blindness |
| Night sweats | Skin and | Night sweats |
| 1 (1 <b>9</b> 110 5 ((1000) | subcutaneous tissue | |
| | disorders | |
| Nikolsky's sign | Skin and | Nikolsky's sign |
| - ·, | subcutaneous tissue | · |
| | disorders | |
| Nitrite urine | Investigations | Nitrite urine |
| Nitrite urine present | Investigations | Nitrite urine present |
| Nodular regenerative | Hepatobiliary | Nodular regenerative |
| hyperplasia | disorders | hyperplasia |
| Normal tension glaucoma | Eye disorders | Normal tension glaucoma |
| Obsessive rumination | Psychiatric disorders | Obsessive rumination |
| Ocular hypertension | Eye disorders | Ocular hypertension |
| Ocular icterus | Eye disorders | Ocular icterus |
| Oculomucocutaneous | Skin and | Oculomucocutaneous syndrome |
| syndrome | subcutaneous tissue | • |
| | disorders | |
| Oedema due to cardiac disease | General disorders and | Oedema due to cardiac disease |
| | administration site | |
| | conditions | |
| Oedema due to hepatic disease | General disorders and | Oedema due to hepatic disease |
| | administration site | • |
| | conditions | |
| Oesophageal varices | Gastrointestinal | Oesophageal varices |
| haemorrhage | disorders | haemorrhage |
| <del></del> | | |

63

| Open angle glaucoma | Eye disorders | Open angle glaucoma |
|---|---|---|
| Ophthalmoplegia | Eye disorders | Ophthalmoplegia |
| Optic atrophy | Eye disorders | Optic atrophy |
| Optic disc disorder | Eye disorders | Optic disc disorder |
| Optic disc drusen | Eye disorders | Optic disc drusen |
| Optic discs blurred | Eye disorders | Optic discs blurred |
| Optic ischaemic neuropathy | Eye disorders | Optic ischaemic neuropathy |
| Optic nerve cupping | Eye disorders | Optic nerve cupping |
| Optic nerve disorder | Eye disorders | Optic nerve disorder |
| Optic nerve infarction | Eye disorders | Optic nerve infarction |
| Optic neuritis | Nervous system | Optic neuritis |
| opere neuritis | disorders | opere neurous |
| Optic neuropathy | Eye disorders | Optic neuropathy |
| Oral mucosal exfoliation | Gastrointestinal | Oral mucosal exfoliation |
| | disorders | |
| Oropharyngeal blistering | Respiratory, thoracic | Oropharyngeal blistering |
| | and mediastinal | |
| | disorders | |
| Oscillopsia | Eye disorders | Oscillopsia |
| Osteomalacia | Musculoskeletal and | Osteomalacia |
| | connective tissue | |
| | disorders | |
| Osteoporosis | Musculoskeletal and | Osteoporosis |
| | connective tissue | |
| | disorders | |
| Osteoporosis-pseudoglioma | Congenital, familial | Osteoporosis-pseudoglioma |
| syndrome | and genetic disorders | syndrome |
| Osteoporotic fracture | Musculoskeletal and | Osteoporotic fracture |
| | connective tissue | |
| | disorders | |
| Papilloedema | Eye disorders | Papilloedema |
| Paracentesis eye | Investigations | Paracentesis eye |
| Paracentesis eye abnormal | Investigations | Paracentesis eye abnormal |
| Paralytic lagophthalmos | Eye disorders | Paralytic lagophthalmos |
| Paramnesia | Psychiatric disorders | Paramnesia |
| Pars plana cyst | Eye disorders | Pars plana cyst |
| Malignant myopia | Eye disorders | Pathologic myopia |
| Pathological fracture | Musculoskeletal and | Pathological fracture |
| | connective tissue | |
| | disorders | |
| Pemphigoid | Skin and | Pemphigoid |
| | subcutaneous tissue | |
| | disorders | |
| Pemphigus | Skin and | Pemphigus |
| | subcutaneous tissue | |
| | disorders | |

| Penile exfoliation | Reproductive system | Penile exfoliation |
|---|---|---|
| | and breast disorders | 1 011110 01110111101 |
| Perihepatic discomfort | Hepatobiliary | Perihepatic discomfort |
| 1 | disorders | • |
| Perihepatitis gonococcal | Infections and | Perihepatitis gonococcal |
| | infestations | |
| Perseveration | Psychiatric disorders | Perseveration |
| pH urine abnormal | Investigations | pH urine abnormal |
| pH urine decreased | Investigations | pH urine decreased |
| pH urine increased | Investigations | pH urine increased |
| Phonological disorder | Psychiatric disorders | Speech sound disorder |
| Photophobia | Eye disorders | Photophobia |
| Phosphenes | Eye disorders | Photopsia |
| Photopsia | Eye disorders | Photopsia |
| Poor quality sleep | Nervous system | Poor quality sleep |
| | disorders | |
| Poor weight gain neonatal | Pregnancy, | Poor weight gain neonatal |
| | puerperium and | |
| | perinatal conditions | |
| Porcelain gallbladder | Hepatobiliary | Porcelain gallbladder |
| | disorders | |
| Portal hypertension | Hepatobiliary | Portal hypertension |
| | disorders | |
| Portal triaditis | Hepatobiliary | Portal tract inflammation |
| | disorders | |
| Portal vein flow decreased | Investigations | Portal vein flow decreased |
| Portal vein pressure increased | Investigations | Portal vein pressure increased |
| Portopulmonary hypertension | Respiratory, thoracic | Portopulmonary hypertension |
| | and mediastinal | |
| D 4 4 1 | disorders | D : 411 |
| Postpartum depression | Psychiatric disorders | Perinatal depression |
| Poverty of speech | Psychiatric disorders | Poverty of speech |
| Poverty of thought content | Psychiatric disorders | Poverty of thought content |
| Presbyopia | Eye disorders | Presbyopia |
| Pressure of speech | Psychiatric disorders | Pressure of speech |
| Profound mental retardation | Nervous system | Intellectual disability |
| Protein urine | disorders | Protein urine |
| | Investigations | |
| Protein urine present | Investigations Museulaskalatal and | Protein urine present |
| Pseudarthrosis | Musculoskeletal and | Pseudarthrosis |
| | connective tissue | |
| Decude blankamentasis | disorders Evo disorders | Deauda blanhavantasia |
| Pseudo-blepharoptosis Pseudopapilloodoma | Eye disorders | Pseudo-blepharoptosis Pseudopapilloadoma |
| Pseudopapilloedema Psychomotor hyperactivity | Eye disorders Norvous system | Pseudopapilloedema Psychomotor hyperactivity |
| 1 Sychomotor hyperactivity | Nervous system<br>disorders | 1 Sychomotor hyperactivity |
| | uisoruers | |

| Psychomotor retardation | Psychiatric disorders | Psychomotor retardation |
|---|---|---|
| Psychomotor skills impaired | Nervous system | Psychomotor skills impaired |
| | disorders | |
| Psychosocial support | Surgical and medical | Psychosocial support |
| | procedures | |
| Psychotherapy | Surgical and medical | Psychotherapy |
| | procedures | |
| Pupil fixed | Eye disorders | Pupil fixed |
| Pupillary deformity | Eve disorders | Pupillary deformity |
| Pupillary disorder | Eye disorders | Pupillary disorder |
| Pupillary reflex impaired | Eye disorders | Pupillary reflex impaired |
| Pupillotonia | Eye disorders | Pupillotonia Pupillotonia |
| Pupils unequal | Eve disorders | Pupils unequal |
| Pyrexia | General disorders and | Pyrexia Pyrexia |
| Julian | administration site | 1 y CAIU |
| | conditions | |
| Rash maculo-papular | Skin and | Rash maculo-papular |
| Rash maculo papulai | subcutaneous tissue | Rush maculo papalar |
| | disorders | |
| Rash pustular | Infections and | Rash pustular |
| Rush pustulai | infestations | Rush pustular |
| Reading disorder | Psychiatric disorders | Reading disorder |
| Red blood cells urine | <b>Investigations</b> | Red blood cells urine |
| Red blood cells urine positive | Investigations | Red blood cells urine positive |
| Refraction disorder | Eye disorders | Refraction disorder |
| Renal colic | Renal and urinary | Renal colic |
| Kenar conc | disorders | Renai cone |
| Renal failure | Renal and urinary | Renal failure |
| Kenai ianui e | disorders | Kenai ianui e |
| Renal function test abnormal | Investigations | Renal function test abnormal |
| Renal pain | Renal and urinary | Renal pain |
| Kenai pam | disorders | Kenai pam |
| Renal tubular acidosis | Renal and urinary | Renal tubular acidosis |
| Renai tubulai acidosis | disorders | Renai tubulai acidosis |
| Repetitive speech | Nervous system | Repetitive speech |
| Repetitive specen | disorders | repetitive specen |
| Residual urine volume | Investigations | Residual urine volume |
| decreased | in consations | decreased |
| Residual urine volume | Investigations | Residual urine volume increased |
| increased | in testigations | residual arme volume mercascu |
| Respiration abnormal | Respiratory, thoracic | Respiration abnormal |
| 200pm and annormal | and mediastinal | |
| | disorders | |
| Retinal artery spasm | Eye disorders | Retinal artery spasm |
| Retinal artery stenosis | Eye disorders | Retinal artery stenosis |
| Retinal cyst | Eye disorders | Retinal cyst |
| ixtinai cyst | Lyc districts | ixemai cyst |

| Retinal degeneration | Eye disorders | Retinal degeneration |
|---|---|---|
| Retinal depigmentation | Eye disorders | Retinal depigmentation |
| Retinal deposits | Eye disorders | Retinal deposits |
| Retinal detachment | Eye disorders | Retinal detachment |
| Retinal disorder | Eye disorders | Retinal disorder |
| Retinal dystrophy | Eye disorders | Retinal dystrophy |
| Retinal haemorrhage | Eye disorders | Retinal haemorrhage |
| Retinal infarction | Eye disorders | Retinal infarction |
| Retinal infiltrates | Eye disorders | Retinal infiltrates |
| Retinal ischaemia | Eye disorders | Retinal ischaemia |
| Retinal oedema | Eye disorders | Retinal oedema |
| Retinal pallor | Eye disorders | Retinal pallor |
| Retinal pigment epitheliopathy | Eye disorders | Retinal pigment epitheliopathy |
| Retinal pigmentation | Eye disorders | Retinal pigmentation |
| Retinal scar | Eye disorders | Retinal scar |
| Retinal tear | Eye disorders | Retinal tear |
| Retinal toxicity | Eye disorders | Retinal toxicity |
| Retinal vascular occlusion | Eye disorders | Retinal vascular occlusion |
| Retinal vascular thrombosis | Eye disorders | Retinal vascular thrombosis |
| Retinal vasculitis | Eye disorders | Retinal vasculitis |
| Retinal vein occlusion | Eye disorders | Retinal vein occlusion |
| Retinal vein thrombosis | Eye disorders | Retinal vein thrombosis |
| Retinitis | Infections and | Retinitis |
| | infestations | |
| Retinogram | Investigations | Retinogram |
| Retinogram abnormal | Investigations | Retinogram abnormal |
| Retinol binding protein | Investigations | Retinol binding protein |
| decreased | _ | decreased |
| Retinoschisis | Eye disorders | Retinoschisis |
| Retinoschisis congenital | Congenital, familial | Retinoschisis congenital |
| _ | and genetic disorders | _ |
| Retrograde amnesia | Nervous system | Retrograde amnesia |
| | disorders | |
| Retrograde portal vein flow | Hepatobiliary | Retrograde portal vein flow |
| | disorders | |
| Reye's syndrome | Hepatobiliary | Reye's syndrome |
| | disorders | |
| Scintillating scotoma | Eye disorders | Scintillating scotoma |
| Screaming | Psychiatric disorders | Screaming |
| Sedation | Nervous system | Sedation |
| | disorders | |
| Selective mutism | Psychiatric disorders | Selective mutism |
| Self esteem decreased | Psychiatric disorders | Self esteem decreased |
| Self injurious behaviour | Psychiatric disorders | Intentional self-injury |
| Self-injurious ideation | Psychiatric disorders | Self-injurious ideation |
| J | J | |

| Severe mental retardation | Nervous system disorders | Intellectual disability |
|---|---|---|
| Sicca syndrome | Musculoskeletal and connective tissue disorders | Sjogren's syndrome |
| Sjogren's syndrome | Musculoskeletal and connective tissue disorders | Sjogren's syndrome |
| Skin erosion | Skin and subcutaneous tissue disorders | Skin erosion |
| Skin exfoliation | Skin and subcutaneous tissue disorders | Skin exfoliation |
| Skin necrosis | Skin and subcutaneous tissue disorders | Skin necrosis |
| Somnolence | Nervous system disorders | Somnolence |
| Speech disorder | Nervous system<br>disorders | Speech disorder |
| Speech disorder developmental | Nervous system<br>disorders | Speech disorder developmental |
| Spider naevus | Skin and subcutaneous tissue disorders | Spider naevus |
| Stag horn calculus | Renal and urinary disorders | Stag horn calculus |
| Stag horn calculus | Renal and urinary disorders | Stag horn calculus |
| Stevens-Johnson syndrome | Skin and subcutaneous tissue disorders | Stevens-Johnson syndrome |
| Stomatitis | Gastrointestinal disorders | Stomatitis |
| Strabismus | Eye disorders | Strabismus |
| Stupor | Nervous system disorders | Stupor |
| Subacute hepatic failure | Hepatobiliary<br>disorders | Subacute hepatic failure |
| Subacute myelo- | Nervous system | Subacute myelo- |
| opticoneuropathy | disorders | opticoneuropathy |
| Subretinal fibrosis | Eye disorders | Subretinal fibrosis |
| Sudden cardiac death | General disorders and administration site conditions | Sudden cardiac death |

| Sudden visual loss | Eye disorders | Sudden visual loss |
|---|---|---|
| Suicidal behaviour | Psychiatric disorders | Suicidal behaviour |
| Suicidal ideation | Psychiatric disorders | Suicidal ideation |
| Suicide attempt | Psychiatric disorders | Suicide attempt |
| Sweat discolouration | Skin and | Sweat discolouration |
| S Weat discolour delon | subcutaneous tissue | Sweat alsolidar attor |
| | disorders | |
| Sweat gland disorder | Skin and | Sweat gland disorder |
| | subcutaneous tissue | |
| | disorders | |
| Synostosis | Musculoskeletal and | Synostosis |
| · | connective tissue | ľ |
| | disorders | |
| Taciturnity | Psychiatric disorders | Taciturnity |
| Tangentiality | Psychiatric disorders | Tangentiality |
| Tear discolouration | Eye disorders | Tear discolouration |
| Tearfulness | Psychiatric disorders | Tearfulness |
| Temperature intolerance | General disorders and | Temperature intolerance |
| | administration site | |
| | conditions | |
| Temperature regulation | General disorders and | Temperature regulation |
| disorder | administration site | disorder |
| | conditions | |
| Temperature regulation | General disorders and | Temperature regulation |
| disorder | administration site | disorder |
| | conditions | |
| Terminal insomnia | Psychiatric disorders | Terminal insomnia |
| Thinking abnormal | Psychiatric disorders | Thinking abnormal |
| Thought blocking | Psychiatric disorders | Thought blocking |
| Thought withdrawal | Psychiatric disorders | Thought withdrawal |
| Tongue exfoliation | Gastrointestinal | Tongue exfoliation |
| | disorders | |
| Total bile acids increased | Investigations | Total bile acids increased |
| Toxic epidermal necrolysis | Skin and | Toxic epidermal necrolysis |
| | subcutaneous tissue | |
| | disorders | |
| Toxic skin eruption | Skin and | Toxic skin eruption |
| | subcutaneous tissue | |
| | disorders | |
| Transaminases abnormal | Investigations | Transaminases abnormal |
| Transaminases increased | Investigations | Transaminases increased |
| Tunnel vision | Nervous system | Tunnel vision |
| Y11 (1 009 1 | disorders | XII (1 009 1 |
| Uhthoff's phenomenon | Nervous system | Uhthoff's phenomenon |
| | disorders | |

| Ultrasound biliary tract | Investigations | Ultrasound biliary tract |
|---|---|---|
| abnormal | investigations | abnormal |
| Ultrasound bladder abnormal | Investigations | Ultrasound bladder abnormal |
| Ultrasound eye abnormal | Investigations | Ultrasound eye abnormal |
| Ultrasound kidney abnormal | Investigations | Ultrasound kidney abnormal |
| Ultrasound liver abnormal | Investigations | Ultrasound liver abnormal |
| Underweight | Metabolism and | Underweight |
| onder weight | nutrition disorders | onder weight |
| Urea urine abnormal | Investigations | Urea urine abnormal |
| Urea urine decreased | Investigations | Urea urine decreased |
| Urea urine increased | Investigations | Urea urine increased |
| Urine abnormality | Renal and urinary | Urine abnormality |
| | disorders | of the abhormancy |
| Urine albumin/creatinine ratio | Investigations | Urine albumin/creatinine ratio |
| abnormal | | abnormal |
| Urine albumin/creatinine ratio | Investigations | Urine albumin/creatinine ratio |
| decreased | in vestigations | decreased |
| Urine albumin/creatinine ratio | Investigations | Urine albumin/creatinine ratio |
| increased | | increased |
| Urine bilirubin increased | Investigations | Urine bilirubin increased |
| Urine calcium decreased | Investigations | Urine calcium decreased |
| Urine calcium increased | Investigations | Urine calcium increased |
| Urine calcium/creatinine ratio | Investigations | Urine calcium/creatinine ratio |
| decreased | | decreased |
| Urine calcium/creatinine ratio | Investigations | Urine calcium/creatinine ratio |
| increased | 8 | increased |
| Urine flow decreased | Renal and urinary | Urine flow decreased |
| | disorders | |
| Urine homocystine present | Investigations | Urine homocystine present |
| Urine ketone body | Investigations | Urine ketone body |
| Urine ketone body present | Investigations | Urine ketone body present |
| Urine lactic acid decreased | Investigations | Urine lactic acid decreased |
| Urine lactic acid increased | Investigations | Urine lactic acid increased |
| Urine nitrogen | Investigations | Urine nitrogen |
| Urine odour abnormal | Renal and urinary | Urine odour abnormal |
| | disorders | |
| Urine osmolarity decreased | Investigations | Urine osmolarity decreased |
| Urine osmolarity increased | Investigations | Urine osmolarity increased |
| Urine output decreased | Investigations | Urine output decreased |
| Urine output increased | Investigations | Urine output increased |
| Urine oxalate decreased | Investigations | Urine oxalate decreased |
| Urine oxalate increased | Investigations | Urine oxalate increased |
| Urine phosphate abnormal | Investigations | Urine phosphorus abnormal |
| Urine phosphate decreased | Investigations | Urine phosphorus decreased |
| Iluino muotoin/ouootinino votio | Investigations | II-ing nuctain/augatining uatio |
|---|---|---|
| Urine protein/creatinine ratio abnormal | Investigations | Urine protein/creatinine ratio abnormal |
| | Investigations | |
| Urine protein/creatinine ratio | Investigations | Urine protein/creatinine ratio decreased |
| decreased | Investigations | |
| Urine protein/creatinine ratio | Investigations | Urine protein/creatinine ratio |
| increased | T 4: 4: | increased |
| Urine sodium abnormal | Investigations | Urine sodium abnormal |
| Urine sodium decreased | Investigations | Urine sodium decreased |
| Urine sodium increased | Investigations | Urine sodium increased |
| Urine transitional cells present | Investigations | Urine transitional cells present |
| Urine uric acid abnormal | Investigations | Urine uric acid abnormal |
| Urine uric acid decreased | Investigations | Urine uric acid decreased |
| Urine uric acid increased | Investigations | Urine uric acid increased |
| Urine viscosity abnormal | Investigations | Urine viscosity abnormal |
| Urine viscosity decreased | Investigations | Urine viscosity decreased |
| Urine viscosity increased | Investigations | Urine viscosity increased |
| Urobilin urine present | Investigations | Urobilinogen urine increased |
| Uveitis | Eye disorders | Uveitis |
| Vaginal exfoliation | Reproductive system | Vaginal exfoliation |
| | and breast disorders | |
| Vaginal ulceration | Reproductive system | Vaginal ulceration |
| | and breast disorders | |
| Varices oesophageal | Gastrointestinal | Varices oesophageal |
| | disorders | |
| Caput medusae | Gastrointestinal | Varicose veins of abdominal |
| | disorders | wall |
| Vasodilatation | Vascular disorders | Vasodilatation |
| Venoocclusive liver disease | Hepatobiliary | Venoocclusive liver disease |
| | disorders | |
| Venous stasis retinopathy | Eye disorders | Venous stasis retinopathy |
| Verbigeration | Psychiatric disorders | Verbigeration |
| Vision abnormal neonatal | Eye disorders | Vision abnormal neonatal |
| Vision blurred | Eye disorders | Vision blurred |
| Visual acuity reduced | Eye disorders | Visual acuity reduced |
| Visual brightness | Eye disorders | Visual brightness |
| Visual evoked potentials | Investigations | Visual evoked potentials |
| Visual evoked potentials Visual evoked potentials | Investigations | Visual evoked potentials Visual evoked potentials |
| abnormal | in Conguitons | abnormal |
| Scotoma | Nervous system | Visual field defect |
| ~ Cooling | disorders | , asami nicia acicci |
| Visual field defect | Nervous system | Visual field defect |
| , isum neid delect | disorders | , as and a second delect |
| Visual field tests | Investigations | Visual field tests |
| Visual field tests abnormal | Investigations | Visual field tests abnormal |
| Visual impairment | Eye disorders | Visual impairment |
| v isuai impan ment | Lyc districts | v isuai impan ment |

| Visual pathway disorder | Nervous system<br>disorders | Visual pathway disorder |
|---|---|---|
| Vitreous abscess | Infections and infestations | Vitreous abscess |
| Vitreous detachment | Eye disorders | Vitreous detachment |
| Vitritis | Eye disorders | Vitritis |
| Vulval ulceration | Reproductive system and breast disorders | Vulval ulceration |
| Vulvovaginal ulceration | Reproductive system and breast disorders | Vulvovaginal ulceration |
| Weight abnormal | Investigations | Weight abnormal |
| Weight decrease neonatal | Pregnancy, puerperium and perinatal conditions | Weight decrease neonatal |
| Weight decreased | Investigations | Weight decreased |
| Weight fluctuation | Metabolism and nutrition disorders | Weight fluctuation |
| Weight gain poor | Metabolism and nutrition disorders | Weight gain poor |
| White blood cells urine | Investigations | White blood cells urine |
| White blood cells urine positive | Investigations | White blood cells urine positive |
| X-ray hepatobiliary abnormal | Investigations | X-ray hepatobiliary abnormal |
| X-ray hepatobiliary abnormal | Investigations | X-ray hepatobiliary abnormal |
| Yellow skin | Skin and | Yellow skin |
| | subcutaneous tissue<br>disorders | |

## Appendix 4: Vineland scores

### **OVERVIEW**

The Vineland Adaptive Behavior Scale is a composite of four Vineland domains:

- Communications (Receptive, Expressive, Written)
- Daily Living Skills (Personal, Domestic, Community)
- Socialization (Interpersonal Relationships, Play and Leisure Time, Coping Skills)
- Motor Skills (Gross, Fine)

Reference: Vineland Adaptive Behavior Scales, Interview Edition, Survey Form Manual, S. Sparrow et al, 1984.

The KVINLAND.XPT dataset includes standard scores, age-equivalences, the adaptive levels for subdomains, domains, and adaptive Behavior Composite, and percentile ranks for domains and adaptive behavior composite. These variables are based on the 1984 Vineland scale analyses from the Vineland Interview Edition.

Standard scores (mean 100, SD=15) were analyzed for each of the four adaptive behavior domains and the Adaptive Behavior composite. The standard score is "based on the performance of a representative national standardization sample of 3000 individuals between birth and age 18-11-30" (p. 116).

## STANDARD SCORES

As stated in the Vineland manual (p. 116), "standard scores express in standard deviation units the extent to which the individual's score exceeds or falls below the mean score of persons the same age with whom the instrument was standardized. Adaptive Behavior Composite and adaptive behavior domain standard scores range from 20 to 160, or 5.5 SD below the mean to 4 SD above the mean ... Standard scores have the advantage of being equal units across the full range of scores The difference in performance between standard scores of 100 and 115 is the same as that between 130 and 145. Because they are of equal units, standard scores can easily be manipulated statistically."

## PERCENTILE RANKS

As stated in Vineland manual (p. 117), "although standard scores are superior to percentile ranks in a psychometric sense, they are not easily understood by many people. Percentile ranks aid in giving meaning to standard scores. Percentile ranks range from 0.1 to 99.9. A percentile rank of 50 indicates median performance ... The chief advantage of percentile ranks is that they are easily understood. A major limitation is that unlike standard score units, percentile rank units are unequal ... The difference between percentile ranks of 50 and 55 is much smaller than the difference of percentile ranks of 90 and 95. This occurs because percentile ranks are compressed near the center of the distribution and less heavily concentrated at the extremes."

## ADAPTIVE LEVELS

Adaptive levels are a categorical representation of the standard scores (p. 118):

 $Adaptive\,Level\,Standard\,Score\,Percentile\,Rank$ 

 $High \ge 131 \ge 98$ 

Moderately High 116-130 85-97 Adequate 85-115 16-84 Moderately Low 70-84 3-15 Low  $\leq 69 \leq 2$ 

## AGE EQUIVALENTS

As described on page 119, the age equivalent represents the raw score that was the average of individuals of a given chronological age in the national standardization sample. They are not used for statistical analysis because the scale units are unequal. In the communication domain, for example, performance increases more between the ages of 2 and 3 than between 10 and 11, for example.

## **VARIABLES IN KVINLAND.XPT**

## 12. VARIABLE DESCRIPTION

VNSS Standard score. Standard scores of '<20' are set to 19. Standard scores of 'Above 160' are set to 161.

VNSS\_PRORATED Standard score - prorated. For adaptive behavior composite scores, VNSS\_PRORATED not equal to VNSS means that the

standard score was prorated. VNSS\_PRORATED equal to VNSS means the score was not prorated. VNSS\_PRORATED is missing (not applicable) for the adaptive behavior composite. The Vineland manual describes the rules for prorating on pages 89 and 107.

VNP Percentile rank

VN AL Adaptive level

VN\_AE Age equivalent. VN\_AE is computed using methods given on p. 101 of the Vineland manual (median used only if one or more

subdomain age equivalents are below 0-1 and above 18-11).

VNSCORE Raw score. For domain totals (VNEXAMC=100) VNSCORE is the raw score total for that domain. The raw score total is

undefined for adaptive behavior composite

Records for domain and ADAPTIVE BEHAVIOR COMPOSITE results are derived. These records are identified as follows:

- VNEXAMC=100: domain scores
- VNEXAMC=101: adaptive behavior composite scores

## Composite score

The composite score will be the sum of 4 standardized domain scores. If a subject has only 3 domains, then the standardized score for the missing domain will be prorated and the composite score will be calculated as sum of 4 domains. If a subject has less than 3 domains, then the composite score will not be calculated.

### SAS code:

```
/* Program: vineland.sas
Author: Dr. PPD , University of Texas PPD
```

Purpose: The program implements the 1984 Vineland scale analyses from the Vineland Interview Edition) to calculate standard score,

 $\,$  age-equivalence, the Adaptive Levels for Subdomains and Domains and Adaptive Behavior Composite, and percentile ranks

for Domains and Adaptive Behavior Composite to Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (J&J PRD)

for use in analyzing Vineland data in any J&JPRD study.

Vineland variables:

```
The output dataset contains all variables in the input dataset.
addition, the following variables are created:
   - VNSS:
                    standard score
   - VN AL:
                    adaptive level
   - VN_AE: age equivalent.

- VNSS_PRORATED: standard score - prorated. For adaptive behavior
composite scores, VNSS PRORATED ^= VNSS means the score was
                     prorated, and VNSS PRORATED = VNSS means the score was
not prorated. VNSS PRORATED is missing (not applicable) for
                     the adaptive behavior composite.
   - VNP:
                     percentile rank
                     raw score. For domain totals (VNEXAMC=100) VNSCORE is
   - VNSCORE:
the raw score total for that domain. The raw score total is
                     undefined for adaptive behavior composite
   Records Created:
   The program adds records for domain and ADAPTIVE BEHAVIOR COMPOSITE
results. The records are identified as follows:
   - VNEXAMC=100:
                  domain scores
   - VNEXAMC=101: adaptive behavior composite scores
   Supporting Data Files:
   The program expects the seven lookup data sets to be associated with a SAS
libname of "NORMDATA". These datasets are:
   - vineland table1.sas7bdat
   - vineland table2.sas7bdat
   - vineland table5 2.sas7bdat
   - vineland table6.sas7bdat
   - vineland table8.sas7bdat
   - vineland table10.sas7bdat
   - vineland table11.sas7bdat
   Notes:
   - Standard scores of '<20' are set to 19.
   - Standard scores of 'Above 160' are set to 161.
   - The program assumes that the combination of SUBJECT and VNDT uniquely
identify each record.
   - VN AE is computed using methods given on p. 101 of the Vineland manual
(median used only if one or more subdomain age
      equivalents are below 0-1 and above 18-11).
   Modified: M. Todd 21-Sep-2007 - added header block and macro parameters
(INDATA and OUTDATA).
* /
%macro vineland (indata=,
                outdata=);
%let sortby=SUBJECT VNDT VNMAINC VNSEQ;
datavineland 1(index=(complex=(&sortby))); length
 vnmain $40; set
  &indata(rename=(vnscore= vnscore));
  length vnscore 3; vnscore=left( vnscore);
  drop vnscore; run;
proc means data=vineland 1 noprint nway;
```

```
class SUBJECT VNDT VNMAIN VNMAINC agevisit; var
  vnscore:
  output out=vineland 2 n=n within domain sum=vnscore;
  where vnexam ne "DO\overline{\text{N}}'T K\overline{\text{NOW}}" and \overline{\text{VNSCORE}} NE . and agevisit ne .; run;
proc sort data=vineland 1 out=vineland dk too high(keep=subject vndt vnmain);
  by subject vndt vnmain;
  where vnexam="DON'T KNOW" and VNSCORE>=5;
run:
data vineland 3; merge
  vineland 2
        vineland dk too high (in=indk);
  by subject vndt vnmain;
  if indk then delete;
  if (vnmain in ('COMMUNICATION' 'DAILY LIVING SKILLS' 'SOCIALIZATION') and
n within domain=3) or
     (vnmain='MOTOR SKILLS' and n within domain=2);
run;
proc sql noprint;
  create table vineland 4 as
    select a.*, b. standscore as vnss
    from vineland 3 a left join
    normdata.vineland table1b
    on b.agemin <= agevisit <= b.agemax and a.vnscore=b.raw and a.vnmain=b.domain
    order by subject, vndt, vnmainc;
proc means data=vineland 4 noprint nway;
  class subject vndt agevisit;
  var vnss;
  output out=vineland_5(drop=_:) n=n_domains sum=sum_ss_across_domains;
run;
data vineland 5a; set
  vineland 5;
  if (n domains=3 and 0 \le agevisit \le 71) or (n domains=2 and agevisit>71) and
sum ss across domains ne . then
    prorated flag='X';
run;
proc sql noprint;
  create table vineland 5b as
  select a.*, case when prorated flag='X' and n domains=3 then
prorated sum for 4 domains
                   when prorated flag='X' and n domains=2 then
prorated sum for 3 domains
                   else . end as prorated sum from
    vineland 5a a left join
    normdata.vineland table5 2b
    on a.sum ss across domains=b.actual;
quit;
data vineland 5c; set
  vineland 5b;
  if prorated sum ne . then do;
    sum_ss_across_domains=prorated_sum;
    n_domains=n_domains+1;
  end;
  drop prorated sum; run;
```

```
proc sql noprint;
  create table vineland 6 as
    select a.*, b.domain as vnmain, b.ss as vnss
    from vineland 5c a left join
    normdata.vineland table2b
    onb.ndomain=a.n domains and b.minsum <= a.sum ss across domains <= b.maxSUM
    where (n domains=4 and 0 \le agevisit \le 71) or (n domains=3 and agevisit>51)
order by subject, vndt; quit;
proc sort data=vineland 1 out=vnunique nodupkey; by
  subject vndt;
run;
data combined1;
  merge vineland 4 (in=ins keep=subject vndt vnmain vnmainc vnss vnscore)
        vnunique(drop=vnmain vnmainc vnscore);
  by subject vndt; if
  ins; vnexamc=100;
  vnseq=vnmainc+1-.001;
  vnexam=vnmain;
run;
data combined2;
  merge vineland 6(in=ins keep=subject vndt vnmain vnss prorated flag)
        vnunique(drop=vnmain);
  by subject vndt; if
  ins; vnexam=vnmain;
  vnmainc=5;
  vnexamc=101;
  vnseq=5.1;
  vnscore=.;
run;
data combined3;
  set vineland 1
      combined1
      combined2;
run;
proc sql noprint;
  create table vineland 7 as
    select a.*, b. adaptive level as vn al, c. adaptive level as vn al2, d.ae as
vn ae, e.ae as vn ae2
    from combined3 a left
    join
    normdata.vineland table6b
    on b.domain=a.vnmain and b.subdomain=a.vnexam and
b.agemin<=a.agevisit<=b.agemax and b.minraw<=a.vnss<=b.maxraw
    left join normdata.vineland table8
    on c.domain=a.vnmain and c.subdomain=a.vnexam and
c.agemin <= a.agevisit <= c.agemax and c.minraw <= a.vnscore <= c.maxraw
    left join normdata.vineland table10
    on a.vnmain=d.domain and a.vnexam=d.domain and a.vnscore=d.raw left
    join
    normdata.vineland table11e
    on a.vnmain=e.domain and a.vnexam=e.subdomain and a.vnscore=e.raw
    order by subject, vndt, vnmainc, vnseq;
```

```
quit;
data &outdata;
 set vineland 7; by
 subject vndt;
 length avg method $6;
 retain ael ae2 ae3 ae4 avg method;
    if first.vndt then do;
      ae1=.; ae2=.; ae3=.; ae4=.; avg method='MEAN'; count=1;
    end;
    array ae(4) _ae1 _ae2 _ae3 _ae4;
    length vnss prorated 3;
    if vn ae2 ne '' then vn ae=vn ae2;
    if vn al2 ne '' then vn al=vn al2;
    if vnmain=vnexam and vnmain ne 'ADAPTIVE BEHAVIOR COMPOSITE' then do;
      if vn ae ne '' then do;
        if index(vn ae,'>') or index(vn ae,'<') then do;</pre>
           avg method='MEDIAN';
          if index(vn ae,'>') then ae( count)=228;
          else ae( count) = .1;
        end:
        else do;
          ae( count) = 12 * scan(vn ae, 1, '-') + scan(vn ae, 2, '-');
        count+1;
      end;
    end;
    if vnmain='ADAPTIVE BEHAVIOR COMPOSITE' then do;
      vnss prorated=vnss;
      if prorated flag='X' then vnss=.;
      if avg method='MEAN' then ae avg=round(mean(of ae1- ae4));
      else _ae_avg=median(of ae1- ae4);
      if ae avg=.1 then vn ae='<0-1';
            vn ae=cats(int( ae avg/12),'-',int(mod( ae avg,12)));
    end;
     ss=vnss;
    if vnss=. then _ss=vnss_prorated;
    if ss ne . then vnp=probnorm((ss-100)/15);
            52<= ss<=61 or 139<= ss<=148 then vnp=round(vnp,.001);
    else if 62 \le s \le 138 then vnp = round(vnp, .01);
    format vnp percent7.1;
    label vnss='VINELAND Standard Score'
          vnss prorated='VINELAND Standard Score - Prorated'
          vn ae='VINELAND Age Equivalent'
          vnp ='VINELAND Percentile'
          vn al='VINELAND Adaptive Level';
    drop vn ae2 vn al2 prorated flag :;
  run;
  proc sql noprint;
  drop table COMBINED1, COMBINED2, COMBINED3, VINELAND 1, VINELAND 2,
  VINELAND 3, VINELAND 4, VINELAND 5,
```

```
VINELAND_5A, VINELAND_5B, VINELAND_5C, VINELAND_6, VINELAND_7, VINELAND_DK_TOO_HIGH, VNUNIQUE; quit; %mend vineland;
```

### Appendix 5: CBCL scoring instruction



# INSTRUCTIONS FOR HAND SCORING THE 2001 CBCL/6-18, YSR, AND TRF ON THE 2001 PROFILES

Note. There are some small differences between the hand-scored and computer-scored data entry formats, but they produce the same results. Be sure to use the CBCL and TRF profile forms appropriate for the child's gender. For information on computer-scoring programs, check our web site: www.ASEBA.org

#### Scoring the CBCL and YSR Competence Scales

#### ACTIVITIES SCALE

Do *not* score if data are missing for more than 1 of the 6 scores indicated beside the Roman numerals below. The Roman numerals correspond to those on pages 1 and 2 of the CBCL and YSR and on the profile scoring form. If a respondent checked more than 1 box where only 1 should be checked, score the box closest to "average."

I-A. # of sports.

- If respondent checked box for *None*—enter 0 below profile
  If respondent reported: 1 sport—enter 1 below profile
  2 sports—enter 2 below profile
  3 or more sports—enter 3 below profile
- I-B. Mean of participation & skill in sports.

If respondent checked box for *None*—enter 0 below profile
For each response of *less than average* or *below average*—score 0

average—score 1

more than average or above average—score 2

Excluding blanks and "don't know" responses, compute the *mean* of these scores by summing them and dividing by the number of scores you have summed. Enter this mean on the profile.

II-A. # of other activities.

If respondent checked box for *None*—enter 0 below profile
If respondent reported: 1 activity—enter 1 below profile
2 activities—enter 2 below profile
3 or more activities—enter 3 below profile

Do not count listening to radio or TV, goofing off, or the like as activities.

II-B. Mean of participation & skill in activities. Compute in the same way as specified in I-B for sports.

IV-A. # of jobs.

If respondent checked box for *None*—enter 0 below profile
If respondent reported: 1 job—enter 1 below profile
2 jobs—enter 2 below profile
3 or more jobs—enter 3 below profile

ASEBA, 1 South Prospect Street, Burlington, VT 05401-3456 www.aseba.org; E-mail: Mail@ASEBA.org; Fax: (802) 264-6433

IV-B..Mean job quality. Compute as specified in 1-B.

Total score for Activities Scale. Sum the 6 scores just entered for the items of the Activities scale. If missing data prevent computation of 1 score, substitute the *mean* of the other 5 scores for the missing score in computing the total. Ifitem I-B, II-B, or IV-B is missing and the mean of the other 5 scores exceeds 2.0, round it down to 2.0. Round off total to nearest .5.

SOCIAL SCALE

Do not score if data are missing for more than 1 of the 6 scores.

III-A. # of organizations. If respondent checked box for None-enter 0 below profile

If respondent reported: I-enter 1below profile

2-enter 2 below profile

3 or more--enter 3 below profile

III-B. Mean of participation in organizations. Compute as specified in I-B.

V-1.#offriends. If respondent checked box for *None-enter* 0 below profile

I-enter 1below profile

2 or 3-enter 2 below profile

4 or more-enter 3 below profile

V-2. Contacts with friends. (Item V-2 can be scored 1or 2 even if no close friends were reported in item V-1.)

If respondent checked less than I-enter 0 below profile

Ior2-enter 1 below profile

3 or more-enter 2 below profile

VI-A. Behavior with others (items a, b, & c). If the respondent checked worse-score 0

average-score I

better-score 2

Excluding any items for which the respondent did not check a box, compute the *mean* of these scores and enter-it below the profile.

VI-B. Does things alone (item d). 
If the respondent checked worse-enter 0 below profile

. < Iverage---enter 1below profile

better-enter 2 below profile

Total score for Social Scale. Sum the 6 scoresjust entered for the items of the Social scale. Ifinissing data prevent computation of 1 score, substitute the *mean* of the other 5 scores for the missing score in computing the total. If item 111-B, V-2, VI-A, or VI-B is missing and the mean of the other 5 scores exceeds 2.0, round it down to 2.0. Round off total to nearest .5.

#### CBCL SCHOOL SCALE

Do *not* score if the child does not attend school or if data are missing for any of the 4 scores indicated below for items VII-1 through VII-4, which appear on Page 2 of the CBCL and on the *School* scale of the profile scoring form.

VII-1. Academic performance. For each academic subject checked by respondent:

failing- score 0 below average-score 1 average-score 2 above average-score 3

Enter the *mean* of these scores on the profile. (Academic subjects include reading, writing, arithmetic, spelling, science, English, foreign language, history, social stildies, and similar subjects. Do *not* count physical education, ali, music, home economics, driver education, industrial arts, typing, or the like.)

VII-2. Special services, special class, or special school.

For any type of remedial special services, class, or school (for retarded, emotionally disturbed, learning diability, perceptual-motor handicapped, reading readiness, resource room, behavior problems, etc):

-enter 0 below profile

not in relnedial class-enter 1below profile

VII-3. Repeated grade.

If any grades were repeated-enter 0 below profile no grades repeated-enter 1 below profile

VII-4. School problems.

If the respondent entered any school problem that was present in the last 6 mouths but was not already scored above: -enter 0 below profile

no problem beside those scored above---enter 1below profile

Total score for School Scale. Sum the 4 scoresjust entered on the *School* scale of the profile, unless any score is missing. After computing the total, round off to the nearest .5.

#### CBCL TOTAL COMPETENCE SCORE

Compute the Total Competence score by summing the total scores for the Activities, Social, and School scales. Do *not* compute a Total Competence score if any of these 3 scale scores is inissing. *T scores* for Total Competence scores are listed in the box to the right of the profile. Circle the child's Total Competence score in the column for the child's age. After you circle the child's raw score, look to the right to find the *T* score.

#### YSR ACADEMIC PERFORMANCE

Compute in the same way as specified in VII-I for CBCL Academic Performance.

#### YSR TOTAL COMPETENCE SCORE

Sum the total scores for Activities, Social, and Academic Performance. Do 11oi- ompute a Total Competence score if any of these 3 scores is missing. T scores for Total Competence scores are in the box to the right of the profile. Circle the youth's Total Competence raw score in the column for the youth's gender. After you circle the youth's raw score, look to the right to find the T score.

#### Scoring the TRFA cademic Performance mid Adaptive Functioning

Item VII. For each academic subject, score the teacher's ratings as follows:

Far below grade = 1

Somewhat below grade = 2

At grade level = 3

Somewhat above grade = 4

Far above grade = 5

If a teacher checked two boxes for one subject, use the mean of the two scores assigned to these boxes.

Enter the *mean* of the teacher's ratings for all academic subjects beneath the heading *Academic Performance* on the profile. (Academic subjects include reading, writing, arithmetic, spelling, science, English, foreign language, history, social studies, computer programming, etc. Do *not* count physical education, art, music, home economics, driver education, industrial art.s, typing, or the like.)

Iten1 VIII. For each of the questions 1-4, score the teacher's ratings as follows:

Much less = 1

.S Somewhat less =

2 Slightly less = 3

About ave 1 · age=4

Slightly more = 5

Somewhat more = 6

Much more = 7

Enter the score for each rating beneath the appropriate heading on the profile.

Sum of Items VIII. 1-4. Sum the scores for Items VIII. 1,2, 3, and 4. Enter this sum beneath the appropriate heading on the profile. Do *not* compute this sum if any of the 4 items is missing.

#### Scoring the CBCL/6-18, YSR, and TRF Problem Scales

Do *not* score the problem scales if data are missing for more than 8 items, not counting open-ended items 56h and 113, or YSR socially desirable items 6, 15, 49, 59, 60, 73, 80, 88, 92, 98, 106, 107, 108, 109. If TRF items 56a-56g were left blank, score them 0.

#### TRANSFERRING PROBLEM ITEM SCORES TO THE PROFILES

Templates. Templates are available to aid in transferring data from the school-age fonns to the profiles. Different templates are needed for the CBCL/6-18, YSR, and TRF. To transfer problem item scores onto the profile, place the Page 3 template on Page 3 of the form. For each problem item, the template indicates whether the item's score is to be entered on a syndrome scale or on the OTHER PROBLEMS list of the profile of empirically based syndromes. The template also indicates the DSMcoriented scale on which to score each item. Repeat using the Page 4 template pn Page 4 of the form.

*Item Seo.res.* For each problem item, print the respondent's 0, 1, or 2 response in the appropriate space beside the item on the profile form. If the respondent circled two numbers for an item, print 1 beside the item on the profile form. Comments written by the respondent should be used in judging whether items deserve to be scored, with the following guidelines:

For each problem reported by the respondent, only the item that most specifically describes the problem should be scored. If the respondent's comments show that more than

- one item has been scored for a particular problem, or if the respondent wrote in a problem for item 56h or 113 that is specifically covered elsewhere, score only the most specific item.
- 2. For items on which the respondent noted "used to do this," score as the respondent scored it, unless it clearly occurred earlier than the 6 months specified in the instructions for the CBCL and YSR, or 2 months for the TRF.
- 3. When in doubt, score the item the way the respondent scored it, except on the following items:

CBCL & TRF 9.-0bsessions--exclude anything that is clearly *11ot* obsessional; e.g., do *not* score "won't take no for an answer."

- YSR 9. Can't get mind off certain thoughts-On the YSR, this item is *11ot* restricted to obsessions. Itcan include almost anything the youth lists here except problems that are specifically listed elsewhere. If the youth wrote "sex" for this item, for example, it would be more appropriately scored on Item 96, *1 think about sex too much*. Ifnot covered by another item, responses that might be considered normal for the youth's age should be scored the way the youth scored them; e.g., "cars,""girls,""boys."
- YSR 40. Hears sounds and 70. Sees things core experiences such as "ringing in ears" and "spots befoleeyes" the way the youth scored them; do not score experiences while under the influence of drugs or alcohol.
- 46. Nervous movements-if "can't sit still" or anything entirely covered by item 10 is entered here, score only item 10.
- 56d. Problems with eyes-do *not* score "wears glasses," "near-sighted," and other visual problems having an organic basis.
- CBCL & TRF 66. Compulsions--Oo not score noncompulsive behavior; e.g., "keeps hitting brother."
- YSR 66. Repeats actions-On the YSR, this item is *not* restricted to compulsions. It can include almost anything the youth lists here except problems that are specifically listed elsewhere. Speech repetitions or stammers, for example, would be more appropriately scored on Item 79. Speech problem.
- CBCL 72. Sets fires-score playing with matches or lighter if parent reported it.
- 77. Sleeps more than most--Oo not s.core "wants to stay in bed,"but score difficulties in waking child.
- 83. Stores up too many things-do not Score hobby collections, such as stamps, dolls.
- 84. Strangebehavior and 85. Strange ideas-if what the respondent describes is specifically covered by anotheritern, scorethen lore specificitem instead.
- CBCL & YSR 105. Drugs-if alcohol or tobacco are entered here, score item 2 or 99, if they are not already scored.
- TRF 105. Drugs-iftobacco is entered here, score item 99, if it is not already scored.
- 113. Additional problems-score only if *not* specifically covered by another item; if respondent listed inore than 1"other" item, count only highest toward total problem score. For example, if a respondent

scored one additional problem "2" and another additional problem "1," add 2 to the total problem score.

Syndrome and DSM-Oriented Scale Scores. To obtain the total raw score for each scale, sum the 1s and 2s you have entered for the scale. The OTHER PROBLEMS do not form a scale, but should be summed to help in computing the Total Problems score, as described later.

#### GRAPHIC DISPLAY AND T SCORES

To complete the graphic displays for the syndrome and DSM-oriented scales, circle the number above each scale that equals the total score obtained for that scale. Be sure to circle the 11umber i11 the co/um11 approp1; iatefor the child's age a11d gende1: Then draw a line to connect the circled numbers. Percentiles based on the normative sample can be read from the left side of the graphic display. Tscores can be read from the right side.

#### INTERNALIZING, EXTERNALIZING, TOTAL PROBLEMS

Computatio11 of Scores. On the profile of syndrome scales, look to the right of the graphic display. You will see a column headed Computatio11s. Under Computatio11s, enter the raw scores that you have obtained for each of the syndrome scales and for the OTHER PROBLEMS as follows:

- 1. Enter the scores for the 3 leftmost syndrome scales in the spaces provided.
- 2 Enter their sum in the box marked Illterllal (a).
- 3. Enter the scores for the 2 rightmost syndrome scales in the spaces provided.
- 4. Enter their sum in the box marked External (b).
- 5. Enter the total score for the 3 middle syndrome scales and *OTHER PROBLEMS* in the spacesprovided.
- 6. Entel the sum of scores from # 5 in the box marked (c).
- 7. Enter the sum of scores from boxes (tt), (b), and (c) in the box marked Totttl.

TScores. Obtain Tscores for Internalizing, Externalizing, and Total Problems as follows:

- 1. Look in the appropriate columns of the large box on the right side of the profile forn1.
- 2 In the appropriate column under the heading *Internalizing*, circle the raw score that corresponds to the score you have entered in the box beside *Internal*.
- 3. Look to the right in the III ternalizi11g column headed Tand circle the Tscore that corresponds to the Internalizing raw score that you have obtained.
- 4. Enter this Tscore in the box marked Internal Tunder the Computtitio11s heading.
- 5. Look under the *Exterl1alizi11g* and *Total Problems* headings to obtain *T* scores-in the same way as was done for Internalizing; enter the *Externalizing* and *Totttl Problems T* scores in the appropriate boxes.



| 32. Must be perfect | _7S.Shy,timid<br>_102.Lacks | _56b. Headaches,<br>_56e. Nausea | :W.Others out to<br>— get hlm | 58. Picksskin<br>_ 59.Sexpartspublic | _13. Confused<br>_17.Daydreams | 63. Prefers older kids<br>_67.Runsaway | 22. Disobedient at home 23. Disobedient at .school | _ 53.Overeating<br>_55.Overweight | n n 34 | 44 16<br>43 1" | | 5 <b>'7</b> 46 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| _33. Feels unloved 35. Feels _45. Nel Worthless _ 50. Fearful _ 52. Feelstoo guitty _ 71. Self-conscious | energy<br>_103.Sad<br>_111.Withdrawn<br><i>Tolaf</i> | _56d. Eyeprobs.<br>_56e. Skinprobs.<br>_56f. Stomach<br>_56g. Vomiling<br> | _38. Gels teased<br>_48. Not liked<br>_62. Clumsy<br>_64. Prefers<br>_younger kids | nne _ 60. Sex parts too | _41. Impulsive<br>_61.Poor<br>schoolwork<br>_78. InaHenIIve<br>_80.Stares<br> | 72, Sets fires Sax problems 73. 81. Steals at home 82. Steals outside horn• 90.Swearing 96.Thinks of sax loomuch 99.Uses tobacco | | _56h.Otherphysical<br>problems<br>74.Shows off<br>_77.Sleepsmore<br>93.Talks too much<br>_98.ThumbsuckIng<br>_107. Wets salf (day)<br>_108.Wets thebad | | 34 12-13<br>33 II<br>10 | 8<br>8<br>S<br>4 | |
| _91.Tatksof<br>suicide<br>_112.Worries<br><i>Total</i> | Copyright 2001 T. Act<br>ASEBA, University of<br>1 South Prospect St<br>Web: www.ASEBA.o.<br>UNAUTHORIZED CO | Vermont<br>Bur1ington, VT 05401-<br>rg | | _ 92. Sleeptalks/walks<br>_100.Troublesleeping<br> | | _101.Truant<br>_105.Uses drugs<br>_106.Vandalism<br> | 95.Temper 97.Threatens others 104. oud Total | _109.Whining<br>110.Wishes to be<br>— os)posille sex<br>_113.Other problems<br>Total | 6·1-01 Edition-202 | n | 2<br>1 | JI<br>27<br>26<br>24 |

## Appendix 6: Method for computing height velocity values and z-scores for individual subjects

For each subject, a height velocity value will be assigned to each calendar year according to the following algorithm:

#### **Notations:**

AB = age at baseline height measurement (Months)

A1 = age at measurements assigned to years 1 (months)

HB = height at baseline (cm)

H1 = height at measurements assigned to years 1 (cm)

HV1 = height velocity at measurements assigned to years 1 (cm/year); computed only if the corresponding year was assigned a non-missing height.

Note: HB and AB are required to be non-missing for all subjects included in the height velocity analysis

| Year | Time Interval (months) | Assigned height value (cm) | Assigned height velocity value (cm/year) |
|---|---|---|---|
| 1 | [AB, AB+12<br>) | to the upper limit of the | If H1 is non-missing,<br>HV1=12*(H1-HB)/(A1-AB)<br>If H1 is missing then HV1 is<br>missing |

For each non-missing height velocity value assigned to a year, the z-score will be computed as

| Year | Z-score |
|---|---|
| 1 | If HV1 is non-missing, |
| | Z1 = (HV1 - Mean at mid-point age in years MA1)/Standard deviation at age |
| | MA1), where |
| | the mid-point age in years $MA1 = ((A1+AB)/2)/12 = (A1+AB)/24$ (rounded to |
| | closest first decimal) |
| | and |
| | the mean (same as 50th percentile) and standard deviation (SD) will be read |
| | from the following tables with height velocity normative data for the |
| | corresponding gender and mid-point age in years MA1 |
| | If HV1 is missing then Z1 is missing |

# Height Velocity Normative Data Based on Tanner et al<sup>[6]</sup>

## **Notes:**

The 3<sup>rd</sup>, 50<sup>th</sup> and 97<sup>th</sup> percentiles are interpolated from the height velocity charts from Tanner et

al<sup>[6]</sup> for the average maturing children. These percentiles were provided by Dr. Paul Boepple, who used them in his previous research.

Mean and standard deviation (SD) derived based on the normal (and therefore symmetrical) distribution assumption:

Mean =  $50^{th}$  percentile

 $SD = [(50^{th} \text{ percentile} - 3^{rd} \text{ percentile}) + (97^{th} \text{ percentile} - 50^{th} \text{ percentile})]/2*1.88$ 

The 2.5 years mean and SD is applied for all subjects with age 2 - 2.5 years. For girls, the 15.5 years mean is applied for subjects with age >15.5 years, the 14.5 years SD is applied for subjects age >14.5 years; For boys, the 17.5 years mean and SD is applied for all subjects with age >17.5 years. The values carried forward have been filled up to age 18.5 years for both boys and girls.

## Girls:

| AGE<br>(YEARS) | 50 <sup>th</sup><br>percentile<br>/ Mean | 3 <sup>rd</sup><br>percentile | 97 <sup>th</sup><br>percentile | Derived<br>SD |
|---|---|---|---|---|
| 2.5 | 8.6 | 5.9 | 11.3 | 1.4 |
| 2.6 | 8.5 | 5.8 | 11.2 | 1.4 |
| 2.7 | 8.4 | 5.7 | 11.0 | 1.4 |
| 2.8 | 8.3 | 5.7 | 10.9 | 1.4 |
| 2.9 | 8.2 | 5.6 | 10.7 | 1.4 |
| 3.0 | 8.1 | 5.5 | 10.6 | 1.4 |
| 3.1 | 8.0 | 5.4 | 10.5 | 1.3 |
| 3.2 | 7.9 | 5.4 | 10.3 | 1.3 |
| 3.3 | 7.8 | 5.3 | 10.2 | 1.3 |
| 3.4 | 7.7 | 5.3 | 10.0 | 1.3 |
| 3.5 | 7.6 | 5.2 | 9.9 | 1.3 |
| 3.6 | 7.5 | 5.1 | 9.8 | 1.2 |
| 3.7 | 7.4 | 5.1 | 9.7 | 1.2 |
| 3.8 | 7.4 | 5.0 | 9.5 | 1.2 |
| 3.9 | 7.3 | 5.0 | 9.4 | 1.2 |
| 4.0 | 7.2 | 4.9 | 9.3 | 1.2 |
| 4.1 | 7.1 | 4.9 | 9.2 | 1.2 |
| 4.2 | 7.0 | 4.8 | 9.2 | 1.2 |
| 4.3 | 7.0 | 4.8 | 9.1 | 1.2 |
| 4.4 | 6.9 | 4.7 | 9.1 | 1.1 |
| 4.5 | 6.8 | 4.7 | 9.0 | 1.1 |
| 4.6 | 6.8 | 4.7 | 8.9 | 1.1 |
| 4.7 | 6.7 | 4.7 | 8.8 | 1.1 |
| 4.8 | 6.7 | 4.6 | 8.8 | 1.1 |
| 4.9 | 6.6 | 4.6 | 8.7 | 1.1 |
| 5.0 | 6.6 | 4.6 | 8.6 | 1.1 |
| 5.1 | 6.6 | 4.6 | 8.5 | 1.1 |
| 5.2 | 6.5 | 4.6 | 8.5 | 1.0 |
| 5.3 | 6.5 | 4.5 | 8.4 | 1.0 |
| 5.4 | 6.4 | 4.5 | 8.4 | 1.0 |
| 5.5 | 6.4 | 4.5 | 8.3 | 1.0 |
| 5.6 | 6.4 | 4.5 | 8.2 | 1.0 |
| 5.7 | 6.3 | 4.5 | 8.2 | 1.0 |
| 5.8 | 6.3 | 4.4 | 8.1 | 1.0 |
| 5.9 | 6.2 | 4.4 | 8.1 | 1.0 |
| 6.0 | 6.2 | 4.4 | 8.0 | 1.0 |
| 6.1 | 6.2 | 4.4 | 8.0 | 1.0 |
| 6.2 | 6.2 | 4.4 | 7.9 | 0.9 |
| 6.3 | 6.1 | 4.3 | 7.9 | 0.9 |
| 6.4 | 6.1 | 4.3 | 7.8 | 0.9 |
| 6.5 | 6.1 | 4.3 | 7.8 | 0.9 |

| AGE<br>(YEARS) | 50 <sup>th</sup><br>percentile<br>/ Mean | 3 <sup>rd</sup><br>percentile | 97 <sup>th</sup><br>percentile | Derived<br>SD |
|---|---|---|---|---|
| 6.6 | 6.1 | 4.3 | 7.8 | 0.9 |
| 6.7 | 6.1 | 4.3 | 7.7 | 0.9 |
| 6.8 | 6.0 | 4.3 | 7.7 | 0.9 |
| 6.9 | 6.0 | 4.3 | 7.6 | 0.9 |
| 7.0 | 6.0 | 4.3 | 7.6 | 0.9 |
| 7.1 | 6.0 | 4.3 | 7.6 | 0.9 |
| 7.2 | 6.0 | 4.3 | 7.6 | 0.9 |
| 7.3 | 5.9 | 4.3 | 7.5 | 0.9 |
| 7.4 | 5.9 | 4.3 | 7.5 | 0.9 |
| 7.5 | 5.9 | 4.3 | 7.5 | 0.9 |
| 7.6 | 5.9 | 4.3 | 7.5 | 0.9 |
| 7.7 | 5.9 | 4.3 | 7.5 | 0.9 |
| 7.8 | 5.8 | 4.2 | 7.4 | 0.9 |
| 7.9 | 5.8 | 4.2 | 7.4 | 0.9 |
| 8.0 | 5.8 | 4.2 | 7.4 | 0.9 |
| 8.1 | 5.8 | 4.2 | 7.4 | 0.8 |
| 8.2 | 5.8 | 4.2 | 7.4 | 0.8 |
| 8.3 | 5.7 | 4.2 | 7.3 | 0.8 |
| 8.4 | 5.7 | 4.2 | 7.3 | 0.8 |
| 8.5 | 5.7 | 4.2 | 7.3 | 0.8 |
| 8.6 | 5.7 | 4.2 | 7.3 | 0.8 |
| 8.7 | 5.7 | 4.2 | 7.3 | 0.8 |
| 8.8 | 5.7 | 4.2 | 7.3 | 0.8 |
| 8.9 | 5.7 | 4.2 | 7.3 | 0.8 |
| 9.0 | 5.7 | 4.2 | 7.3 | 0.8 |
| 9.1 | 5.7 | 4.2 | 7.3 | 0.8 |
| 9.2 | 5.7 | 4.2 | 7.3 | 0.8 |
| 9.3 | 5.8 | 4.3 | 7.4 | 0.8 |
| 9.4 | 5.8 | 4.3 | 7.4 | 0.8 |
| 9.5 | 5.8<br>5.9 | 4.3 | 7.4<br>7.5 | 0.8 |
| 9.6 | 6.0 | 4.3 | 7.5 | 0.9 |
| 9.7 | 6.0 | 4.3 | 7.8 | 0.9 |
| 9.9 | 6.1 | 4.4 | 7.9 | 0.9 |
| 10.0 | 6.2 | 4.4 | 8.0 | 1.0 |
| 10.0 | 6.3 | 4.5 | 8.1 | 1.0 |
| 10.1 | 6.4 | 4.5 | 8.3 | 1.0 |
| 10.2 | 6.5 | 4.6 | 8.4 | 1.0 |
| 10.4 | 6.6 | 4.6 | 8.6 | 1.0 |
| 10.5 | 6.7 | 4.7 | 8.7 | 1.1 |
| 10.6 | 6.9 | 4.9 | 8.9 | 1.1 |
| 10.7 | 7.1 | 5.1 | 9.1 | 1.1 |
| 10.8 | 7.4 | 5.3 | 9.3 | 1.1 |
| 10.9 | 7.6 | 5.5 | 9.5 | 1.1 |
| 11.0 | 7.8 | 5.7 | 9.7 | 1.1 |

| | = oth | and | o =th | |
|---|---|---|---|---|
| AGE | 50 <sup>th</sup> | 3 <sup>rd</sup> | 97 <sup>th</sup> | Derived |
| (YEARS) | percentile | percentile | percentile | SD |
| | / Mean | | | |
| 11.1 | 7.9 | 5.8 | 9.8 | 1.1 |
| 11.2 | 8.0 | 5.9 | 10.0 | 1.1 |
| 11.3 | 8.1 | 5.9 | 10.1 | 1.1 |
| 11.4 | 8.2 | 6.0 | 10.3 | 1.1 |
| 11.5 | 8.3 | 6.1 | 10.4 | 1.1 |
| 11.6 | 8.1 | 5.9 | 10.2 | 1.2 |
| 11.7 | 7.9 | 5.7 | 10.1 | 1.2 |
| 11.8 | 7.7 | 5.5 | 9.9 | 1.2 |
| 11.9 | 7.5 | 5.3 | 9.8 | 1.2 |
| 12.0 | 7.3 | 5.1 | 9.6 | 1.2 |
| 12.1 | 7.0 | 4.8 | 9.3 | 1.2 |
| 12.2 | 6.7 | 4.5 | 9.0 | 1.2 |
| 12.3 | 6.5 | 4.2 | 8.6 | 1.2 |
| 12.4 | 6.2 | 3.9 | 8.3 | 1.2 |
| 12.5 | 5.9 | 3.6 | 8.0 | 1.2 |
| 12.6 | 5.6 | 3.3 | 7.7 | 1.1 |
| 12.7 | 5.3 | 3.1 | 7.3 | 1.1 |
| 12.8 | 4.9 | 2.8 | 7.0 | 1.1 |
| 12.9 | 4.6 | 2.6 | 6.6 | 1.1 |
| 13.0 | 4.3 | 2.3 | 6.3 | 1.1 |
| 13.1 | 4.0 | 2.1 | 6.0 | 1.0 |
| 13.2 | 3.8 | 1.9 | 5.7 | 1.0 |
| 13.3 | 3.5 | 1.6 | 5.4 | 1.0 |
| 13.4 | 3.3 | 1.4 | 5.1 | 1.0 |
| 13.5 | 3.0 | 1.2 | 4.8 | 1.0 |
| 13.6 | 2.8 | 1.0 | 4.5 | 0.9 |
| 13.7 | 2.5 | 0.9 | 4.2 | 0.9 |
| 13.8 | 2.3 | 0.7 | 3.8 | 0.8 |
| 13.9<br>14.0 | 2.0<br>1.8 | 0.6<br>0.4 | 3.2 | 0.8 |
| 14.0 | 1.6 | 0.4 | 2.9 | 0.7 |
| 14.1 | 1.4 | | 2.6 | 0.7 |
| 14.3 | 1.3 | | 2.4 | 0.6 |
| 14.4 | 1.1 | | 2.1 | 0.5 |
| 14.5 | 0.9 | | 1.8 | 0.5 |
| 14.6 | 0.8 | | | 0.5 |
| 14.7 | 0.7 | | | 0.5 |
| 14.8 | 0.6 | | | 0.5 |
| 14.9 | 0.5 | | | 0.5 |
| 15.0 | 0.4 | | | 0.5 |
| 15.1 | 0.3 | | | 0.5 |
| 15.2 | 0.3 | | | 0.5 |
| 15.3 | 0.2 | | | 0.5 |
| 15.4 | 0.2 | | | 0.5 |
| 15.5 | 0.1 | | | 0.5 |

| AGE<br>(YEARS) | 50 <sup>th</sup> percentile / Mean | 3 <sup>rd</sup> percentile | 97 <sup>th</sup><br>percentile | Derived<br>SD |
|---|---|---|---|---|
| 15.6 | 0.1 | | | 0.5 |
| 15.7 | 0.1 | | | 0.5 |
| 15.8 | 0.1 | | | 0.5 |
| 15.9 | 0.1 | | | 0.5 |
| 16.0 | 0.1 | | | 0.5 |
| 16.1 | 0.1 | | | 0.5 |
| 16.2 | 0.1 | | | 0.5 |
| 16.3 | 0.1 | | | 0.5 |
| 16.4 | 0.1 | | | 0.5 |
| 16.5 | 0.1 | | | 0.5 |
| 16.6 | 0.1 | | | 0.5 |
| 16.7 | 0.1 | | | 0.5 |
| 16.8 | 0.1 | | | 0.5 |
| 16.9 | 0.1 | | | 0.5 |
| 17.0 | 0.1 | | | 0.5 |
| 17.1 | 0.1 | | | 0.5 |
| 17.2 | 0.1 | | | 0.5 |
| 17.3 | 0.1 | | | 0.5 |
| 17.4 | 0.1 | | | 0.5 |
| 17.5 | 0.1 | | | 0.5 |
| 17.6 | 0.1 | | | 0.5 |
| 17.7 | 0.1 | | | 0.5 |
| 17.8 | 0.1 | | | 0.5 |
| 17.9 | 0.1 | | | 0.5 |
| 18.0 | 0.1 | | | 0.5 |
| 18.1 | 0.1 | | | 0.5 |
| 18.2 | 0.1 | | | 0.5 |
| 18.3 | 0.1 | | | 0.5 |
| 18.4 | 0.1 | | | 0.5 |
| 18.5 | 0.1 | | | 0.5 |

# **Boys:**

| AGE<br>(YEARS) | 50 <sup>th</sup><br>percentile<br>/ Mean | 3 <sup>rd</sup><br>percentile | 97 <sup>th</sup><br>percentile | Derived<br>SD |
|---|---|---|---|---|
| (ILAKS) | / ivican | percentife | percentific | SD |
| 2.5 | 8.3 | 5.7 | 10.9 | 1.4 |
| , | | - | _ | |

| AGE<br>(YEARS) | 50 <sup>th</sup><br>percentile<br>/ Mean | 3 <sup>rd</sup><br>percentile | 97 <sup>th</sup><br>percentile | Derived<br>SD |
|---|---|---|---|---|
| 2.8 | 8.0 | 5.5 | 10.5 | 1.3 |
| 2.9 | 7.9 | 5.5 | 10.3 | 1.3 |
| 3.0 | 7.8 | 5.4 | 10.2 | 1.3 |
| 3.1 | 7.7 | 5.3 | 10.1 | 1.3 |
| 3.2 | 7.6 | 5.3 | 10.0 | 1.2 |
| 3.3 | 7.6 | 5.2 | 9.8 | 1.2 |
| 3.4 | 7.5 | 5.2 | 9.7 | 1.2 |
| 3.5 | 7.4 | 5.1 | 9.6 | 1.2 |
| 3.6 | 7.3 | 5.1 | 9.5 | 1.2 |
| 3.7 | 7.3 | 5.0 | 9.4 | 1.2 |
| 3.8 | 7.2 | 5.0 | 9.4 | 1.2 |
| 3.9 | 7.2 | 4.9 | 9.3 | 1.2 |
| 4.0 | 7.1 | 4.9 | 9.2 | 1.1 |
| 4.1 | 7.0 | 4.9 | 9.1 | 1.1 |
| 4.2 | 7.0 | 4.8 | 9.0 | 1.1 |
| 4.3 | 6.9 | 4.8 | 9.0 | 1.1 |
| 4.4 | 6.9 | 4.7 | 8.9 | 1.1 |
| 4.5 | 6.8 | 4.7 | 8.8 | 1.1 |
| 4.6 | 6.8 | 4.7 | 8.8 | 1.1 |
| 4.7 | 6.7 | 4.7 | 8.7 | 1.1 |
| 4.8 | 6.7 | 4.6 | 8.7 | 1.1 |
| 4.9 | 6.6 | 4.6 | 8.6 | 1.1 |
| 5.0 | 6.6 | 4.6 | 8.6 | 1.1 |
| 5.1 | 6.6 | 4.6 | 8.5 | 1.1 |
| 5.2 | 6.5 | 4.6 | 8.5 | 1.0 |
| 5.3 | 6.5 | 4.5 | 8.4 | 1.0 |
| 5.4<br>5.5 | 6.4<br>6.4 | 4.5<br>4.5 | 8.4<br>8.3 | 1.0 |
| 5.6 | 6.4 | 4.5 | 8.3 | 1.0 |
| 5.7 | 6.3 | | | 1.0 |
| 5.8 | 6.3 | 4.4 | 8.2<br>8.2 | 1.0 |
| 5.9 | 6.2 | 4.4 | 8.1 | 1.0 |
| 6.0 | 6.2 | 4.3 | 8.1 | 1.0 |
| 6.1 | 6.2 | 4.3 | 8.0 | 1.0 |
| 6.2 | 6.1 | 4.3 | 8.0 | 1.0 |
| 6.3 | 6.1 | 4.2 | 7.9 | 1.0 |
| 6.4 | 6.0 | 4.2 | 7.9 | 1.0 |
| 6.5 | 6.0 | 4.2 | 7.8 | 1.0 |
| 6.6 | 6.0 | 4.2 | 7.8 | 1.0 |
| 6.7 | 6.0 | 4.2 | 7.8 | 0.9 |
| 6.8 | 5.9 | 4.2 | 7.7 | 0.9 |
| 6.9 | 5.9 | 4.2 | 7.7 | 0.9 |
| 7.0 | 5.9 | 4.2 | 7.7 | 0.9 |
| 7.1 | 5.9 | 4.2 | 7.7 | 0.9 |
| 7.2 | 5.9 | 4.2 | 7.6 | 0.9 |

| AGE<br>(YEARS) | 50 <sup>th</sup><br>percentile<br>/ Mean | 3 <sup>rd</sup><br>percentile | 97 <sup>th</sup><br>percentile | Derived<br>SD |
|---|---|---|---|---|
| 7.3 | 5.8 | 4.1 | 7.6 | 0.9 |
| 7.4 | 5.8 | 4.1 | 7.5 | 0.9 |
| 7.5 | 5.8 | 4.1 | 7.5 | 0.9 |
| 7.6 | 5.8 | 4.1 | 7.4 | 0.9 |
| 7.7 | 5.7 | 4.0 | 7.4 | 0.9 |
| 7.8 | 5.7 | 4.0 | 7.3 | 0.9 |
| 7.9 | 5.6 | 3.9 | 7.3 | 0.9 |
| 8.0 | 5.6 | 3.9 | 7.2 | 0.9 |
| 8.1 | 5.6 | 3.9 | 7.2 | 0.9 |
| 8.2 | 5.5 | 3.9 | 7.1 | 0.9 |
| 8.3 | 5.5 | 3.8 | 7.1 | 0.9 |
| 8.4 | 5.4 | 3.8 | 7.0 | 0.9 |
| 8.5 | 5.4 | 3.8 | 7.0 | 0.9 |
| 8.6 | 5.4 | 3.8 | 7.0 | 0.8 |
| 8.7 | 5.4 | 3.8 | 6.9 | 0.8 |
| 8.8 | 5.3 | 3.8 | 6.9 | 0.8 |
| 8.9 | 5.3 | 3.8 | 6.8 | 0.8 |
| 9.0 | 5.3 | 3.8 | 6.8 | 0.8 |
| 9.1 | 5.3 | 3.8 | 6.8 | 0.8 |
| 9.2 | 5.3 | 3.8 | 6.8 | 0.8 |
| 9.3 | 5.2 | 3.7 | 6.7 | 0.8 |
| 9.4 | 5.2 | 3.7 | 6.7 | 0.8 |
| 9.5 | 5.2 | 3.7 | 6.7 | 0.8 |
| 9.6 | 5.2 | 3.7 | 6.7 | 0.8 |
| 9.7 | 5.2 | 3.7 | 6.6 | 8.0 |
| 9.8 | 5.1 | 3.7 | 6.6 | 8.0 |
| 9.9 | 5.1 | 3.7 | 6.5 | 0.8 |
| 10.0 | 5.1 | 3.7 | 6.5 | 0.7 |
| 10.1 | 5.1 | 3.7 | 6.5 | 0.7 |
| 10.2 | 5.1 | 3.7 | 6.5 | 0.7 |
| 10.3 | 5.1 | 3.7 | 6.5 | 0.7 |
| 10.4 | 5.1 | 3.7 | 6.5 | 0.7 |
| 10.5 | 5.1 | 3.7 | 6.5 | 0.7 |
| 10.6 | 5.1 | 3.7 | 6.5 | 0.8 |
| 10.7 | 5.1 | 3.7 | 6.5 | 8.0 |
| 10.8 | 5.2 | 3.7 | 6.6 | 0.8 |
| 10.9 | 5.2 | 3.7 | 6.6 | 0.8 |
| 11.0 | 5.2 | 3.7 | 6.6 | 0.8 |
| 11.1 | 5.2 | 3.7 | 6.6 | 0.8 |
| 11.2 | 5.2 | 3.7 | 6.6 | 8.0 |
| 11.3 | 5.3 | 3.8 | 6.7 | 0.8 |
| 11.4 | 5.3 | 3.8 | 6.7 | 0.8 |
| 11.5 | 5.3 | 3.8 | 6.7 | 0.8 |
| 11.6 | 5.4 | 3.8 | 6.8 | 0.8 |
| 11.7 | 5.5 | 3.9 | 6.9 | 8.0 |

| AGE<br>(YEARS) | 50 <sup>th</sup><br>percentile<br>/ Mean | 3 <sup>rd</sup><br>percentile | 97 <sup>th</sup><br>percentile | Derived<br>SD |
|---|---|---|---|---|
| 11.8 | 5.5 | 3.9 | 7.1 | 0.8 |
| 11.9 | 5.6 | 4.0 | 7.2 | 0.9 |
| 12.0 | 5.7 | 4.0 | 7.3 | 0.9 |
| 12.1 | 5.9 | 4.2 | 7.6 | 0.9 |
| 12.2 | 6.1 | 4.3 | 8.0 | 1.0 |
| 12.3 | 6.4 | 4.5 | 8.3 | 1.0 |
| 12.4 | 6.6 | 4.6 | 8.7 | 1.1 |
| 12.5 | 6.8 | 4.8 | 9.0 | 1.1 |
| 12.6 | 7.2 | 5.1 | 9.4 | 1.2 |
| 12.7 | 7.6 | 5.3 | 9.9 | 1.2 |
| 12.8 | 7.9 | 5.6 | 10.3 | 1.3 |
| 12.9 | 8.3 | 5.8 | 10.8 | 1.3 |
| 13.0 | 8.7 | 6.1 | 11.2 | 1.4 |
| 13.1 | 8.9 | 6.3 | 11.3 | 1.3 |
| 13.2 | 9.0 | 6.5 | 11.5 | 1.3 |
| 13.3 | 9.2 | 6.7 | 11.6 | 1.3 |
| 13.4 | 9.3 | 6.9 | 11.8 | 1.3 |
| 13.5 | 9.5 | 7.1 | 11.9 | 1.3 |
| 13.6 | 9.3 | 6.9 | 11.7 | 1.3 |
| 13.7 | 9.0 | 6.7 | 11.5 | 1.3 |
| 13.8 | 8.8 | 6.4 | 11.2 | 1.3 |
| 13.9 | 8.5 | 6.2 | 11.0 | 1.3 |
| 14.0 | 8.3 | 6.0 | 10.8 | 1.3 |
| 14.1 | 7.9 | 5.6 | 10.4 | 1.3 |
| 14.2 | 7.6 | 5.2 | 10.0 | 1.3 |
| 14.3 | 7.2 | 4.9 | 9.6 | 1.3 |
| 14.4 | 6.9 | 4.5 | 9.2 | 1.3 |
| 14.5 | 6.5 | 4.1 | 8.8 | 1.3 |
| 14.6 | 6.1 | 3.7 | 8.4 | 1.3 |
| 14.7 | 5.8 | 3.4 | 8.1 | 1.3 |
| 14.8 | 5.4 | 3.0 | 7.7 | 1.3 |
| 14.9 | 5.1 | 2.7 | 7.4 | 1.3 |
| 15.0 | 4.7 | 2.3 | 7.0 | 1.3 |
| 15.1 | 4.4 | 2.1 | 6.7 | 1.2 |
| 15.2 | 4.1 | 1.9 | 6.4 | 1.2 |
| 15.3 | 3.9 | 1.6 | 6.1 | 1.2 |
| 15.4 | 3.6 | 1.4 | 5.8 | 1.2 |
| 15.5 | 3.3 | 1.2 | 5.5 | 1.1 |
| 15.6 | 3.1 | 1.0 | 5.2 | 1.1 |
| 15.7 | 2.9 | 0.9 | 4.9 | 1.1 |
| 15.8 | 2.6 | 0.7 | 4.7 | 1.0 |
| 15.9 | 2.4 | 0.6 | 4.4 | 1.0 |
| 16.0 | 2.2 | 0.4 | 4.1 | 1.0 |
| 16.1 | 2.1 | | 3.9 | 1.0 |
| 16.2 | 1.9 | | 3.7 | 0.9 |

| AGE<br>(YEARS) | 50 <sup>th</sup> percentile / Mean | 3 <sup>rd</sup> percentile | 97 <sup>th</sup><br>percentile | Derived<br>SD |
|---|---|---|---|---|
| 16.3 | 1.8 | | 3.4 | 0.9 |
| 16.4 | 1.6 | | 3.2 | 0.8 |
| 16.5 | 1.5 | | 3.0 | 0.8 |
| 16.6 | 1.4 | | 2.8 | 0.8 |
| 16.7 | 1.3 | | 2.7 | 0.8 |
| 16.8 | 1.1 | | 2.5 | 0.7 |
| 16.9 | 1.0 | | 2.4 | 0.7 |
| 17.0 | 0.9 | | 2.2 | 0.7 |
| 17.1 | 0.8 | | 2.1 | 0.7 |
| 17.2 | 0.7 | | 2.0 | 0.6 |
| 17.3 | 0.7 | | 1.8 | 0.6 |
| 17.4 | 0.6 | | 1.7 | 0.6 |
| 17.5 | 0.5 | | 1.6 | 0.6 |
| 17.6 | 0.5 | | | 0.6 |
| 17.7 | 0.5 | | | 0.6 |
| 17.8 | 0.5 | | | 0.6 |
| 17.9 | 0.5 | | | 0.6 |
| 18.0 | 0.5 | | | 0.6 |
| 18.1 | 0.5 | | | 0.6 |
| 18.2 | 0.5 | | | 0.6 |
| 18.3 | 0.5 | | | 0.6 |
| 18.4 | 0.5 | | | 0.6 |
| 18.5 | 0.5 | _ | | 0.6 |

## Appendix 7: List of generic and brand names of AED medications

## **Generic names**

Acetazolamide

Cannabidiol

Carbamazepine

Clobazam

Clonazepam

Diazepam

Eslicarbazepine

acetate Ethosuximide

Gabapentin

Lacosamide

Lamotrigine

Levetiracetam

Nitrazepam

Oxcarbazepine

Perampanel

Piracetam

Phenobarbital

Phenytoin

Pregabalin

Primidone

Retigabine

Rufinamide

Sodium

valproate

Stiripentol

Tiagabine

Topiramate

Valproic acid

Vigabatrin

Zonisamide

## Brand names (available as):

Carbogen modified release

Convulex

Desitrend

Diacomit

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| D | iaı | n | O> | ۲S | R |
|---|-----|----|----|----|---|
| _ | | ٠. | • | | |

Emeside

**Epanutin** 

**Epidiolex** 

**Epilim** 

**Epilim Chrono** 

**Epilim Chronosphere** 

Episenta (prolonged

release) Epival

Frisium

Fycompa

Gabitril

Inovelon

Keppra

Lamictal

Lyrica

Neurontin

Nootropil

Phenytoin Sodium Flynn

Rivotril

Sabril

Tapclob

Tegretol

**Tegretol Prolonged Release** 

**Topamax** 

Trileptal

Trobalt

Valium

Vimpat

Zarontin

Zebinix

Zonegran